CLINICAL TRIAL: NCT03158285
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of Guselkumab Administered Subcutaneously in Subjects With Active Psoriatic Arthritis
Brief Title: A Study Evaluating the Efficacy and Safety of Guselkumab Administered Subcutaneously in Participants With Active Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108219; CNTO1959PSA3002 (Other: Janssen Research & Development, LLC); 2016-001224-63 (EudraCT Number)
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Results first posted 2020-11-05 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Guselkumab (Experimental): Participants will receive subcutaneous (SC) guselkumab 100 milligram (mg) once every 4 weeks (q4w) from Week 0 through Week 100.
  Interventions: Drug: Guselkumab
- Group 2: Guselkumab and Placebo (Experimental): Participants will receive SC guselkumab 100 mg at Weeks 0 and 4 then once every 8 weeks (q8w) (Weeks 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, and 100) and placebo injections at other visits (Weeks 8, 16, 24, 32, 40, 48, 56, 64, 72, 80, 88, and 96) to maintain the blind.
  Interventions: Drug: Guselkumab; Drug: Placebo
- Group 3: Placebo Followed by Guselkumab (Experimental): Participants will receive SC placebo q4w from Week 0 to Week 20 and will cross over at Week 24 to receive SC guselkumab 100 mg q4w from Week 24 through Week 100.
  Interventions: Drug: Guselkumab; Drug: Placebo

INTERVENTIONS:
Drug: Guselkumab — Participants will receive 100 mg of guselkumab as a sterile liquid for SC injection.
  Other Names: CNTO 1959
Drug: Placebo — Participants will receive matching placebo as SC injection.
  Arms: Group 2: Guselkumab and Placebo; Group 3: Placebo Followed by Guselkumab

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of guselkumab treatment in participants with active psoriatic arthritis (PsA) by assessing the reduction in signs and symptoms of PsA.

DETAILED DESCRIPTION:
This is a study of guselkumab in participants with active PsA who are biologically naive and have had inadequate response to standard therapies. It will evaluate the clinical efficacy of guselkumab in the reduction of signs and symptoms, structural damage inhibition and the safety profile of guselkumab in the treatment of PsA. The study will consist of a screening phase (up to 6 weeks), a blinded treatment phase (approximately 100 weeks) including a placebo controlled period from Week 0 to Week 24 and an active treatment period from Week 24 to Week 100 and a safety follow-up phase of 12 weeks after the last administration of study agent. Efficacy, health economics, safety, pharmacokinetics, immunogenicity, biomarker and pharmacogenomics evaluations will be performed in the study at defined schedule.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Psoriatic Arthritis (PsA) for at least 6 months before the first administration of study agent and meet Classification criteria for Psoriatic Arthritis (CASPAR) at screening
* Have active PsA as defined by: at least 5 swollen joints and at least 5 tender joints at screening and at baseline, and CRP greater than or equal to (>=) 0.6 milligram per deciLitre (mg/dL) at screening from the central laboratory
* Have at least 1 of the PsA subsets: distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis (confirmation of sacroiliitis should be performed at the screening visit by a locally performed pelvic x-ray [single anterior-posterior view] unless a pelvic or SI joint x-ray or pelvic magnetic resonance imaging (MRI) has been previously performed. Results must be documented)
* Have active plaque psoriasis, with at least one psoriatic plaque of >= 2 centimeter (cm) diameter or nail changes consistent with psoriasis or documented history of plaque psoriasis
* Have active PsA despite previous non-biologic disease-modifying antirheumatic drug (DMARD), apremilast, and/or nonsteroidal anti-inflammatory drug (NSAID) therapy

Exclusion Criteria:

* Has other inflammatory diseases that might confound the evaluations or benefit of guselkumab therapy, including but not limited to rheumatoid arthritis (RA), axial spondyloarthritis (this does not include a primary diagnosis of PsA with spondylitis), systemic lupus erythematosus, or Lyme disease
* Has previously received any biologic treatment
* Has ever received tofacitinib, baricitinib, filgotinib, peficitinib (ASP015K), decernotinib (VX-509), or any other Janus kinase (JAK) inhibitor
* Has received any systemic immunosuppressants (eg, azathioprine, cyclosporine, 6 thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, tacrolimus) within 4 weeks of the first administration of study agent
* Is currently receiving 2 or more non-biologic DMARDs (other than methotrexate [MTX], sulfasalazine [SSZ], Hydroxychloroquine [HCQ], leflunomide [LEF]) including, but not limited to chloroquine, gold preparations, and penicillamine within 4 weeks before the first administration of study agent
* Has received apremilast within 4 weeks prior to the first administration of study agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2020-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (138):
- United States (8):
  - Rheumatology Associates, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Associates PC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - Clinical Research Center of Connecticut, Danbury, Connecticut
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - University of Michigan, Ann Arbor, Michigan
  - Arthritis Consultants, St Louis, Missouri
  - Austin Regional Clinic, Austin, Texas
- Bulgaria (7):
  - Multiprofile Hospital for Active Treatment - Plovdiv, Plovdiv
  - Multiprofile Hosptal for Active Treatment Eurohospital Plovdiv, Plovdiv
  - Medical Center Teodora, Rousse
  - Diagnostic Consulting Center No 17, Sofia
  - Military Medical Academy, Sofia
  - Medical Centre Synexus, Sofia
  - MHAT-Targovishte, AD, Targovishte
- Czechia (7):
  - Revmaclinic, Brno
  - Revmacentrum MUDr. Mostera, s.r.o., Brno-Židenice
  - MUDr. Rosypalova, s.r.o, Ostrava
  - Revmatologicky institut, Prague
  - Revmatologicka ambulance, Prague
  - Medical Plus S.R.O., Uherské Hradiště
  - PV-Medical S.R.O, Zlín
- Estonia (4):
  - Parnu Hospital, Pärnu
  - OU Innomedica, Tallinn
  - East Tallinn Central Hospital, Tallinn
  - Clinical Research Centre, Tartu
- Latvia (4):
  - Daugavpils Regional Hospital, Daugavpils
  - Derma Clinic Riga, Riga
  - J Kisis Ltd, Riga
  - Orto Clinic Ltd, Riga
- Lithuania (4):
  - Vakk, Jsc, Kaunas
  - Siauliai Republican Hospital, Public Institution, Šiauliai
  - Central Outpatient Clinic, Vilnius
  - National Osteoporosis Centre, Vilnius
- Malaysia (6):
  - Hospital Selayang, Batu Caves
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Sarawak General Hospital, Kuching
  - Hospital Melaka, Malacca
  - Hospital Putrajaya, Putrajaya
  - Hospital Tuanku Jaafar, Seremban
- Poland (16):
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Bydgoszcz
  - NSZOZ Unica CR, Dąbrówka
  - Centrum Kliniczno Badawcze, Elblag
  - Centrum Badań Klinicznych PI-House sp. z o.o., Gdansk
  - Centrum Badawcze Wspolczesnej Terapii, Lodz
  - Centrum Medyczne AMED oddzial w Lodzi, Lodz
  - NZOZ Lecznica MAK-MED. S.C., Nadarzyn
  - Etyka Osrodek Badan Klinicznych, Olsztyn
  - Centrum Medyczne Hetmańska, Poznan
  - Lubelskie Centrum Diagnostyczne, Świdnik
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - Medycyna Kliniczna, Warsaw
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. prof. dr hab. med. Eleonory Reicher, Warsaw
  - Centrum Medyczne AMED Warszawa Targowek, Warsaw
  - Wromedica, Wroclaw
  - Biogenes Sp. z o. o., Wroclaw
- Russia (25):
  - Chelyabinsk Regional Clinical Dermatovenerological Dispensary, Chelyabinsk
  - Medical and Sanitary Unit ''Severstal'', Cherepovets
  - Regional Clinical Hospital for War Veterans, Kemerovo
  - Medical Centre Maximum Health, Kemerovo
  - Family polyclinic #4, Korolyov
  - Krasnodar Clinical Dermatovenerologic Dispensary, Krasnodar
  - Krasnoyarsk State Medical University, Krasnoyarsk
  - Lipetsk Regional Dermatovenerological Dispensary, Lipetsk
  - Moscow State Medical and Stomatological University, Moscow
  - Clinical Diagnostic Center 'Ultramed', Omsk
  - Orenburg State Medical University, Orenburg
  - Republican Hospital n.a.V.A.Baranov, Petrozavodsk
  - Rostov Regional Clinical Dermatovenerological Dispensary, Rostov
  - Ryazan Regional Clinical Dermatovenerological Dispensary, Ryazan
  - City Clinic №25 - City Rheumatology Centre, Saint Petersburg
  - Leningrad region clinical hospital, Saint Petersburg
  - Saratov Regional Clinical Hospital, Saratov
  - Smolensk regional hospital on Smolensk railway station, Smolensk
  - Tula Regional Clinical Dermatovenerological Dispensary, Tula
  - Regional Clinical Hospital, Tver'
  - Republican Clinical Hospital - G.G. Kuvatov, Ufa
  - Clinical Emergency Hospital n.a. N.V. Solovyev, Yaroslavl
  - Clinical Hospital #3, Yaroslavl
  - Clinical Hospital #10, Yaroslavl
  - Research Institute of Dermatovenerology, Immunology, Yekaterinburg
- Spain (15):
  - Hosp. Univ. A Coruña, A Coruña
  - Hosp. Univ. de Cruces, Barakaldo
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp. Reina Sofia, Córdoba
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Regional. Carlos Haya, Málaga
  - Hosp. de Merida, Mérida
  - H.U. Infanta Sofía, San Sebastián de los Reyes
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Infanta Luisa, Seville
  - Hosp. Unv. de Valme, Seville
  - Hosp. Univ. Dr. Peset, Valencia
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. Do Meixoeiro, Vigo
- Taiwan (5):
  - Hualien Tzu Chi Hospital, Hualien City
  - Chang Gung Memorial Hospital Kaohsiung Branch, Kaohsiung City
  - National Cheng Kung University Medical Center, Tainan
  - Chang Kung Memorial Hospital, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- Turkey (Türkiye) (9):
  - Ankara Bilkent City Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Uludag University Medical Faculty, Bursa
  - Osmangazi University Medical Faculty, Eskişehir
  - Bakirkoy Training and Research Hospital, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Izmir Katip Celebi University Medical Faculty Ataturk Training and Research Hospital, Izmir
- Ukraine (28):
  - Communal Noncommercial Enterprise Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - Municipal health care institution Chernihiv Regional Hospital, Chernihiv
  - Ivano-Frankivsk National Medical University, Ivano-Frankivsk City Clinical Hospital, Ivano-Frankivsk
  - Communal Institution of Health Kharkiv City multifield hospital №18, Kharkiv
  - Kharkiv Railway Clinical Hospital N1 Of Brance 'Health Center', Kharkiv
  - State Institution Institute of therapy named after L.T.Malaya AMS Ukraine, Kharkiv
  - Municipal Institution Regional hospital-center of emergency care and disasters medicine, Kharkiv
  - Mi 'Kherson City Clinical Hospital Of E.E. Karabelesh', Kherson
  - Khmelnitckiy regional hospital, Khmelnytsky
  - City Clinical Hospital No. 2, Kryvyi Rih
  - Kyiv City Clinical Hospital #3, Kyiv
  - Medical Center 'Consylium Medical', Kyiv
  - Kyiv Regional Clinical Hospital, Kyiv
  - Kyiv Railway Station Clinical Hospital #2, Kyiv
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - Danylo Halytsky Lviv National Medical University, Lviv
  - Lviv Communcal City Clinical Hospital #4, Lviv
  - Municipal Non-profit Enterprise 'Odesa Regional Clinical Hospital' Odesa Regional Council, Odesa
  - Multidisciplinary Medical Center of Odessa National Medical University, Odesa
  - Poltava Regional Clinical Hospital HSEI of Ukraine Ukrainian Medical Stomatological Academy, Poltava
  - Sumy State University, Sumy
  - Municipal institution of Tepnopil Regional Council 'Ternopil University Hospital', Ternopil
  - Municipal Non-commercial Enterprise Ternopil University Hospital of Ternopil Regional Council, Ternopil
  - MNCE Zakarpatska Regional Clinical Hospital named after A Novak of Zakarpatska Regional Council, Uzhhorod
  - Medical Center LTD Health Clinic Department of Cardiology and Rheumatology, Vinnytsia
  - VNMUn.af.Pyrogova,CNE Vinnytsia Regional Clinical Hospital n.af.Pyrogova Vinnytsia Regional Council, Vinnytsia
  - Zaporizhzhya Regional Clinical Hospital, Zaporizhzhya
  - Municipal institution Central Clinical Hospital #1 Zhytomir, Zhytomyr

REFERENCES:
- [Derived] Gladman DD, Eder L, Selmi C, Mease PJ, Ogdie A, Lozenski K, Adamson E, Sharaf M, Rampakakis E, Pina Vegas L, Coates LC. Influence of Biological Sex on Participant Characteristics, Guselkumab Efficacy and Radiographic Progression in Active Psoriatic Arthritis: Post Hoc Analysis of Three Randomized Trials. Rheumatol Ther. 2025 Dec 15. doi: 10.1007/s40744-025-00812-3. Online ahead of print. PMID 41396391
- [Derived] Crauwels H, Ringold S, Howard S, Van Hartingsveldt B, Smith V, Jett M, Baguet T, Adamson E, Chakravarty SD, Leu JH. Extrapolating Guselkumab Efficacy to Juvenile Psoriatic Arthritis from Adult Psoriatic Arthritis and Adult and Pediatric Psoriasis Data. Paediatr Drugs. 2025 Oct 28. doi: 10.1007/s40272-025-00725-2. Online ahead of print. PMID 41152645
- [Derived] Ritchlin CT, Lubrano E, Chimenti MS, Leibowitz E, Sharaf M, Rampakakis E, Nantel F, Lavie F, Deodhar A. Guselkumab Efficacy in Biologic-Naive Participants with Psoriatic Arthritis and Severe Disease Activity: Post Hoc Analysis of a Phase 3 Study. Rheumatol Ther. 2025 Oct;12(5):925-940. doi: 10.1007/s40744-025-00777-3. Epub 2025 Jul 21. PMID 40690163
- [Derived] Siebert S, Schett G, Raychaudhuri SP, Guma M, Chen W, Gao S, Chakravarty SD, Lavie F, Rahman P. Correlation of changes in inflammatory and collagen biomarkers with durable guselkumab efficacy through 2 years in participants with active psoriatic arthritis: results from a phase III randomized controlled trial. Ther Adv Musculoskelet Dis. 2024 Oct 27;16:1759720X241283536. doi: 10.1177/1759720X241283536. eCollection 2024. PMID 39493888
- [Derived] Mease P, Korotaeva T, Shesternya P, Kokhan M, Rukavitsyn A, Vasilchenkov D, Sharaf M, Lavie F, Deodhar A. Guselkumab in Biologic-Naive Patients with Active Psoriatic Arthritis in Russia: A Post Hoc Analysis of the DISCOVER-1 and -2 Randomized Clinical Trials. Rheumatol Ther. 2024 Dec;11(6):1551-1567. doi: 10.1007/s40744-024-00713-x. Epub 2024 Sep 25. PMID 39320583
- [Derived] Curtis JR, Deodhar A, Soriano ER, Rampakakis E, Shawi M, Shiff NJ, Han C, Tillett W, Gladman DD. Early Improvements with Guselkumab Associate with Sustained Control of Psoriatic Arthritis: Post hoc Analyses of Two Phase 3 Trials. Rheumatol Ther. 2024 Dec;11(6):1501-1517. doi: 10.1007/s40744-024-00702-0. Epub 2024 Sep 11. PMID 39261446
- [Derived] Ritchlin CT, Mease PJ, Boehncke WH, Tesser J, Chakravarty SD, Rampakakis E, Shawi M, Schiopu E, Merola JF, McInnes IB, Deodhar A. Durable control of psoriatic arthritis with guselkumab across domains and patient characteristics: post hoc analysis of a phase 3 study. Clin Rheumatol. 2024 Aug;43(8):2551-2563. doi: 10.1007/s10067-024-06991-8. Epub 2024 Jun 7. PMID 38844682
- [Derived] Baraliakos X, Gladman DD, Chakravarty SD, Gong C, Shawi M, Rampakakis E, Kishimoto M, Soriano ER, Mease PJ. BASDAI versus ASDAS in evaluating axial involvement in patients with psoriatic arthritis: a pooled analysis of two phase 3 studies. Rheumatol Adv Pract. 2024 Apr 23;8(2):rkae058. doi: 10.1093/rap/rkae058. eCollection 2024. PMID 38765190
- [Derived] Warren RB, McInnes IB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, Mease PJ. Comparative Effectiveness of Bimekizumab and Guselkumab in Patients with Psoriatic Arthritis at 52 Weeks Assessed Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):829-839. doi: 10.1007/s40744-024-00659-0. Epub 2024 Mar 15. PMID 38488975
- [Derived] Rahman P, McInnes IB, Deodhar A, Schett G, Mease PJ, Shawi M, Cua DJ, Sherlock JP, Kollmeier AP, Xu XL, Sheng S, Ritchlin CT, McGonagle D. Association between enthesitis/dactylitis resolution and patient-reported outcomes in guselkumab-treated patients with psoriatic arthritis. Clin Rheumatol. 2024 May;43(5):1591-1604. doi: 10.1007/s10067-024-06921-8. Epub 2024 Mar 12. PMID 38472528
- [Derived] Curtis JR, McInnes IB, Rahman P, Gladman DD, Peterson S, Yang F, Adejoro O, Kollmeier AP, Shiff NJ, Han C, Shawi M, Tillett W, Mease PJ. Work Productivity and General Health Through 2 Years of Guselkumab Treatment in a Phase 3 Randomized Trial of Patients With Active Psoriatic Arthritis. Rheumatol Ther. 2024 Apr;11(2):425-441. doi: 10.1007/s40744-024-00642-9. Epub 2024 Feb 22. PMID 38386178
- [Derived] Coates LC, Rahman P, Mease PJ, Shawi M, Rampakakis E, Kollmeier AP, Xu XL, Chakravarty SD, McInnes IB, Tam LS. Continuous improvement through differential trajectories of individual minimal disease activity criteria with guselkumab in active psoriatic arthritis: post hoc analysis of a phase 3, randomized, double-blind, placebo-controlled study. BMC Rheumatol. 2024 Feb 4;8(1):6. doi: 10.1186/s41927-024-00375-w. PMID 38310261
- [Derived] Strober B, Coates LC, Lebwohl MG, Deodhar A, Leibowitz E, Rowland K, Kollmeier AP, Miller M, Wang Y, Li S, Chakravarty SD, Chan D, Shawi M, Yang YW, Thaҫi D, Rahman P. Long-Term Safety of Guselkumab in Patients with Psoriatic Disease: An Integrated Analysis of Eleven Phase II/III Clinical Studies in Psoriasis and Psoriatic Arthritis. Drug Saf. 2024 Jan;47(1):39-57. doi: 10.1007/s40264-023-01361-w. Epub 2023 Oct 31. PMID 37906417
- [Derived] Mease PJ, Gladman DD, Poddubnyy D, Chakravarty SD, Shawi M, Kollmeier AP, Xu XL, Xu S, Deodhar A, Baraliakos X. Efficacy of Guselkumab on Axial-Related Symptoms Through up to 2 Years in Adults with Active Psoriatic Arthritis in the Phase 3, Randomized, Placebo-Controlled DISCOVER-2 Study. Rheumatol Ther. 2023 Dec;10(6):1637-1653. doi: 10.1007/s40744-023-00592-8. Epub 2023 Oct 11. PMID 37819505
- [Derived] Gottlieb AB, McInnes IB, Rahman P, Kollmeier AP, Xu XL, Jiang Y, Sheng S, Shawi M, Chakravarty SD, Lavie F, Mease PJ. Low rates of radiographic progression associated with clinical efficacy following up to 2 years of treatment with guselkumab: results from a phase 3, randomised, double-blind, placebo-controlled study of biologic-naive patients with active psoriatic arthritis. RMD Open. 2023 Feb;9(1):e002789. doi: 10.1136/rmdopen-2022-002789. PMID 36828643
- [Derived] Rahman P, Boehncke WH, Mease PJ, Gottlieb AB, McInnes IB, Shawi M, Wang Y, Sheng S, Kollmeier AP, Theander E, Yu J, Leibowitz E, Marrache AM, Coates LC. Safety of Guselkumab With and Without Prior Tumor Necrosis Factor Inhibitor Treatment: Pooled Results Across 4 Studies in Patients With Psoriatic Arthritis. J Rheumatol. 2023 Jun;50(6):769-780. doi: 10.3899/jrheum.220928. Epub 2023 Jan 15. PMID 36642439
- [Derived] Curtis JR, McInnes IB, Rahman P, Gladman DD, Peterson S, Agarwal P, Yang F, Kollmeier AP, Hsia EC, Shiff NJ, Zhou B, Han C, Shawi M, Tillett W, Mease PJ. The Effect of Guselkumab on Work Productivity in Biologic-Naive Patients with Active Psoriatic Arthritis Through Week 52 of the Phase 3, Randomized, Placebo-Controlled DISCOVER-2 Trial. Adv Ther. 2022 Oct;39(10):4613-4631. doi: 10.1007/s12325-022-02270-7. Epub 2022 Aug 10. PMID 35947349
- [Derived] Curtis JR, McInnes IB, Rahman P, Gladman DD, Yang F, Peterson S, Agarwal P, Kollmeier AP, Hsia EC, Han C, Shiff NJ, Shawi M, Tillett W, Mease PJ. The Effect of Guselkumab on General Health State in Biologic-Naive Patients with Active Psoriatic Arthritis Through Week 52 of the Phase 3, Randomized, Placebo-Controlled DISCOVER-2 Trial. Adv Ther. 2022 Oct;39(10):4632-4644. doi: 10.1007/s12325-022-02269-0. Epub 2022 Aug 10. PMID 35947348
- [Derived] Coates LC, Ritchlin CT, Gossec L, Helliwell PS, Rahman P, Kollmeier AP, Xu XL, Shawi M, Karyekar CS, Contre C, Noel W, Sheng S, Wang Y, Xu S, Mease PJ. Guselkumab provides sustained domain-specific and comprehensive efficacy using composite indices in patients with active psoriatic arthritis. Rheumatology (Oxford). 2023 Feb 1;62(2):606-616. doi: 10.1093/rheumatology/keac375. PMID 35766811
- [Derived] Schett G, Loza MJ, Palanichamy A, FitzGerald O, Ritchlin C, Bay-Jensen AC, Nielsen SH, Gao S, Hsia EC, Kollmeier AP, Xu XL, Baribaud F, Sweet K. Collagen Turnover Biomarkers Associate with Active Psoriatic Arthritis and Decrease with Guselkumab Treatment in a Phase 3 Clinical Trial (DISCOVER-2). Rheumatol Ther. 2022 Aug;9(4):1017-1030. doi: 10.1007/s40744-022-00444-x. Epub 2022 Mar 30. PMID 35352313
- [Derived] Ritchlin CT, Mease PJ, Boehncke WH, Tesser J, Schiopu E, Chakravarty SD, Kollmeier AP, Xu XL, Shawi M, Jiang Y, Sheng S, Wang Y, Xu S, Merola JF, McInnes IB, Deodhar A. Sustained and improved guselkumab response in patients with active psoriatic arthritis regardless of baseline demographic and disease characteristics: pooled results through week 52 of two phase III, randomised, placebo-controlled studies. RMD Open. 2022 Mar;8(1):e002195. doi: 10.1136/rmdopen-2022-002195. PMID 35296534
- [Derived] Rahman P, Mease PJ, Helliwell PS, Deodhar A, Gossec L, Kavanaugh A, Kollmeier AP, Hsia EC, Zhou B, Lin X, Shawi M, Karyekar CS, Han C. Guselkumab demonstrated an independent treatment effect in reducing fatigue after adjustment for clinical response-results from two phase 3 clinical trials of 1120 patients with active psoriatic arthritis. Arthritis Res Ther. 2021 Jul 14;23(1):190. doi: 10.1186/s13075-021-02554-3. PMID 34261541
- [Derived] Sweet K, Song Q, Loza MJ, McInnes IB, Ma K, Leander K, Lakshminarayanan V, Franks C, Cooper P, Siebert S. Guselkumab induces robust reduction in acute phase proteins and type 17 effector cytokines in active psoriatic arthritis: results from phase 3 trials. RMD Open. 2021 May;7(2):e001679. doi: 10.1136/rmdopen-2021-001679. PMID 34011674
- [Derived] Rahman P, Ritchlin CT, Helliwell PS, Boehncke WH, Mease PJ, Gottlieb AB, Kafka S, Kollmeier AP, Hsia EC, Xu XL, Shawi M, Sheng S, Agarwal P, Zhou B, Ramachandran P, Zhuang Y, McInnes IB. Pooled Safety Results Through 1 Year of 2 Phase III Trials of Guselkumab in Patients With Psoriatic Arthritis. J Rheumatol. 2021 Dec;48(12):1815-1823. doi: 10.3899/jrheum.201532. Epub 2021 May 1. PMID 33934076
- [Derived] McGonagle D, McInnes IB, Deodhar A, Schett G, Shawi M, Kafka S, Karyekar CS, Kollmeier AP, Hsia EC, Xu XL, Sheng S, Agarwal P, Zhou B, Ritchlin CT, Rahman P, Mease PJ. Resolution of enthesitis by guselkumab and relationships to disease burden: 1-year results of two phase 3 psoriatic arthritis studies. Rheumatology (Oxford). 2021 Nov 3;60(11):5337-5350. doi: 10.1093/rheumatology/keab285. PMID 33822898
- [Derived] McInnes IB, Rahman P, Gottlieb AB, Hsia EC, Kollmeier AP, Chakravarty SD, Xu XL, Subramanian RA, Agarwal P, Sheng S, Jiang Y, Zhou B, Zhuang Y, van der Heijde D, Mease PJ. Efficacy and Safety of Guselkumab, an Interleukin-23p19-Specific Monoclonal Antibody, Through One Year in Biologic-Naive Patients With Psoriatic Arthritis. Arthritis Rheumatol. 2021 Apr;73(4):604-616. doi: 10.1002/art.41553. Epub 2021 Mar 17. PMID 33043600
- [Derived] Mease PJ, Rahman P, Gottlieb AB, Kollmeier AP, Hsia EC, Xu XL, Sheng S, Agarwal P, Zhou B, Zhuang Y, van der Heijde D, McInnes IB; DISCOVER-2 Study Group. Guselkumab in biologic-naive patients with active psoriatic arthritis (DISCOVER-2): a double-blind, randomised, placebo-controlled phase 3 trial. Lancet. 2020 Apr 4;395(10230):1126-1136. doi: 10.1016/S0140-6736(20)30263-4. Epub 2020 Mar 13. PMID 32178766

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 741 participants were randomized and 739 participants received at least one dose of study drug: 246 in placebo group, 248 in guselkumab 100 mg q8w group, and 245 in guselkumab 100 mg q4w group. Two participants were randomized in error and were never treated. Disposition is presented till active treatment period (Week100).
Groups:
- Placebo to Guselkumab 100 mg q4w: Participants were randomized to receive placebo matched to guselkumab subcutaneous injections every 4 weeks through Week 20 in the placebo controlled period (PCP), then to receive guselkumab 100 milligrams (mg) subcutaneous injection from Week 24 every 4 weeks through Week 100 in the active treatment period.
- Guselkumab 100 mg q8w: Participants were randomized to receive guselkumab 100 mg subcutaneous injections at Weeks 0 and 4, then every 8 weeks (q8w) through Week 100 and placebo matched to guselkumab injections at Week 8 then q8w through Week 100.
- Guselkumab 100 mg q4w: Participants were randomized to receive guselkumab 100 mg subcutaneous injections every 4 weeks (q4w) through Week 100.
Period: Placebo-controlled Period: Week 0 - 24
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Started | 246 | 248 | 245
Pooled Population: Enthesitis Assessment | 255 (Pooled population (255) = 77 (CNTO1959PSA3001[NCT03162796]) + 178 (CNTO1959PSA3002)) | 230 (Pooled population (230)= 72 (CNTO1959PSA3001) + 158 (CNTO1959PSA3002)) | 243 (Pooled population (243)= 73 (CNTO1959PSA3001) + 170 (CNTO1959PSA3002))
Pooled Population: Dactylitis Assessment | 154 (Pooled population (154) = 55 (CNTO1959PSA3001) + 99 (CNTO1959PSA3002)) | 160 (Pooled population (160) = 49 (CNTO1959PSA3001) + 111 (CNTO1959PSA3002)) | 159 (Pooled population (159) = 38 (CNTO1959PSA3001) + 121 (CNTO1959PSA3002))
Completed | 240 | 240 | 236
Not Completed | 6 | 8 | 9
Not completed — Adverse Event | 4 | 2 | 6
Not completed — Lack of Efficacy | 0 | 3 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other | 1 | 1 | 0
Period: Active Treatment Period: Week 24 - 52
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Started | 238 (2 participants did not enter the active treatment.) | 240 | 234 (2 participants did not enter the active treatment.)
Completed | 228 | 234 | 227
Not Completed | 10 | 6 | 7
Not completed — Adverse Event | 3 | 0 | 1
Not completed — Lack of Efficacy | 5 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Other | 1 | 1 | 0
Period: Active Treatment Period: Week 52-100
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Started | 228 | 232 (2 participants did not enter the active treatment.) | 227
Completed | 210 | 223 | 219
Not Completed | 18 | 9 | 8
Not completed — Adverse Event | 7 | 5 | 3
Not completed — Lack of Efficacy | 1 | 1 | 3
Not completed — Withdrawal by Subject | 5 | 2 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Other | 4 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w | Total
Number analyzed (Participants) | 246 | 248 | 245 | 739
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.68) | 44.9 (11.89) | 45.9 (11.47) | 45.7 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 119 | 103 | 351
  Male | 117 | 129 | 142 | 388
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 245 | 247 | 245 | 737
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 8 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 242 | 240 | 242 | 724
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  BULGARIA | 14 | 9 | 6 | 29
  CZECH REPUBLIC | 13 | 5 | 15 | 33
  ESTONIA | 5 | 8 | 5 | 18
  LATVIA | 3 | 3 | 0 | 6
  LITHUANIA | 8 | 8 | 4 | 20
  MALAYSIA | 3 | 6 | 3 | 12
  POLAND | 35 | 27 | 23 | 85
  RUSSIAN FEDERATION | 92 | 77 | 104 | 273
  SPAIN | 3 | 12 | 4 | 19
  TAIWAN | 0 | 1 | 0 | 1
  TURKEY | 2 | 8 | 6 | 16
  UKRAINE | 65 | 83 | 73 | 221
  UNITED STATES | 3 | 1 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20 Response at Week 24
Description: ACR 20 response: >=20% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=20% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of Health Assessment Questionnaire (HAQ-DI; 20-question instrument assessing 8 functional areas; range: 0-3, 0= no difficulty, 3= inability to perform task in that area), and CRP. Treatment Failure (TF) criteria- discontinued study drug, initiated/increased dose of non-biologic disease-modifying antirheumatic drugs (DMARDs) or oral corticosteroids, initiated prohibited psoriatic arthritis treatment.
Time Frame: Week 24
Population: Analysis population is full analysis set 1 (FAS1). Participants who achieved ACR 20 response at Week 24 and did not meet any treatment failure (TF) criteria before Week 24 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants | 32.9 | 64.1 | 63.7
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 31.2, 95% CI 2-sided [22.9 to 39.5]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 30.8, 95% CI 2-sided [22.4 to 39.1]

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24
Description: HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3 where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning. Negative change from baseline indicates improvement of physical function.
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be missing at random (MAR) and imputed using multiple imputation (MI).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale | -0.1300 [-0.1912 to -0.0687] | -0.3672 [-0.4282 to -0.3062] | -0.4004 [-0.4617 to -0.3390]
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, ANCOVA; Least Square (LS) Mean difference = -0.2372, 95% CI 2-sided [-0.3210 to -0.1534]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference = -0.2704, 95% CI 2-sided [-0.3544 to -0.1864]

3. Secondary Outcome: Percentage of Participants Who Achieved an ACR 50 Response at Week 24
Description: ACR 50 response was defined as greater than or equal to (>=)50 percent (%) improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=50% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI; a 20-question instrument assessing 8 functional areas; range: 0-3, 0=no difficulty, 3=inability to perform a task in that area), and C-Reactive Protein (CRP).
Time Frame: Week 24
Population: Analysis population is FAS1. Participants who achieved ACR 50 response at Week 24 and did not meet any TF criteria before Week 24 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants | 14.2 | 31.5 | 33.1
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 17.2, 95% CI [10.0 to 24.4]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 18.8, 95% CI 2-sided [11.5 to 26.1]

4. Secondary Outcome: Percentage of Participants Who Achieved Psoriasis Response With IGA Score of 0 (Cleared) or 1 (Minimal) and >=2 Grade Reduction From Baseline at Week 24 Among Participants With >=3% BSA Psoriatic Involvement and IGA Score of >=2 (Mild) at Baseline
Description: A psoriasis Investigator's Global Assessment (IGA) response was defined as an IGA score of 0 (cleared) or 1 (minimal) and >=2 grade reduction from baseline in the IGA psoriasis score. The IGA documents the investigator's assessment of the patient's psoriasis and lesions are graded for induration, erythema and scaling, each using a 5 point scale: 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe). The IGA score of psoriasis was based upon the average of induration, erythema and scaling scores. The participant's psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: Week 24
Population: FAS1 among participants with >=3% BSA psoriatic involvement and an IGA score >=2 (mild) at baseline. Participants who achieved psoriasis IGA response at Week 24 and did not meet any TF criteria before Week 24 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 183 | 176 | 184
percentage of participants | 19.1 | 70.5 | 68.5
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 50.9, 95% CI 2-sided [42.2 to 59.7]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Difference in percentage = 49.8, 95% CI 2-sided [41.2 to 58.4]

5. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20 Response at Week 16
Description: ACR 20 response was defined as >= 20% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=20% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI; a 20-question instrument assessing 8 functional areas; range: 0-3, 0=no difficulty, 3=inability to perform a task in that area), and CRP.
Time Frame: Week 16
Population: Analysis population is FAS1. Participants who achieved ACR 20 response at Week 16 and did not meet any TF criteria before Week 16 were considered as responders. Participants who met 1 or more TF criteria before Week 16 or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants | 33.7 | 55.2 | 55.9
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 21.5, 95% CI 2-sided [13.1 to 30.0]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 22.2, 95% CI 2-sided [13.7 to 30.7]

6. Secondary Outcome: Change From Baseline in Modified Van Der Heijde-Sharp (vdH-S) Score at Week 24
Description: Modified vdH-S score is the sum of the erosion score (hand, feet) and joint space narrowing (JSN) score (hand, feet). Joint erosion score is the summary of erosion severity in 40 joints of hand scored according to the surface area, from 0 (no erosion) to 5 (complete collapse of bone) and 12 joints of 2 feet (each side of the foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum erosion score of 320. JSN score is the total JSN score in same 52 joints as above, each joint scored according to the subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum JSN score of 208. Total score ranges from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score indicates more joint damage. Positive changes from baseline in the modified vdH-S total, erosion and JSN scores indicate progression of joint damage.
Time Frame: Baseline and Week 24
Population: FAS1 for structural damage (FAS1-SD) included all participants who received at least 1 dose (complete/partial) of study agent according to randomized treatment group regardless of treatment actually received. Observed data were used regardless if 1 or more TF criteria were met. Missing data were assumed to be MAR and imputed using MI.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale | 0.95 [0.61 to 1.29] | 0.52 [0.18 to 0.86] | 0.29 [-0.05 to 0.63]
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.072, ANCOVA; LS Mean difference = -0.43, 95% CI 2-sided [-0.90 to 0.03]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.011, ANCOVA; LS Mean difference = -0.66, 95% CI 2-sided [-1.13 to -0.19]

7. Secondary Outcome: Percentage of Participants With Resolution of Enthesitis at Week 24 Among the Participants With Enthesitis at Baseline
Description: Enthesitis was assessed using the Leeds Enthesitis Index (LEI), a tool developed to assess enthesitis in participants with PsA and evaluates the presence (score of 1) or absence (score of 0) of pain by applying local pressure to the following entheses: left and right lateral epicondyle humerus, left and right medial femoral condyle, and left and right achilles tendon insertion. The enthesitis index score is a total score of the 6 evaluated sites from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). A LEI score of 0 at a post baseline visit indicates resolution of enthesitis when baseline LEI>0. The outcome measure was planned to be reported for pooled population from CNTO1959PSA3001 and CNTO1959PSA3002 studies.
Time Frame: Week 24
Population: FAS1 among participants with enthesitis at baseline pooled from CNTO1959PSA3001 (NCT03162796) and CNTO1959PSA3002 (NCT03158285) studies. Participants with enthesitis resolution at Week 24 and did not meet any TF criteria before Week 24 considered responders. Participants who met 1/more TF criteria or with missing data considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 255 | 230 | 243
percentage of participants | 29.4 | 49.6 | 44.9
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.030, Cochran-Mantel-Haenszel; Difference in response rates = 20.1, 95% CI 2-sided [11.8 to 28.5]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.030, Cochran-Mantel-Haenszel; Difference in response rates = 14.6, 95% CI 2-sided [6.4 to 22.7]

8. Secondary Outcome: Percentage of Participants With Resolution of Dactylitis at Week 24 Among the Participants With Dactylitis at Baseline
Description: The presence and severity of dactylitis was assessed in both hands and feet using a scoring system from 0 to 3 (0-no dactylitis, 1-mild dactylitis, 2-moderate dactylitis, and 3-severe dactylitis) for each digit. The results were summed to produce a final score ranging from 0 to 60. Higher score indicates more severe dactylitis. Resolution of dactylitis was defined as a dactylitis score of 0 with the baseline dactylitis score >0. The outcome measure was planned to be reported for pooled population from CNTO1959PSA3001 and CNTO1959PSA3002 studies.
Time Frame: Week 24
Population: FAS1 among participants with dactylitis at baseline pooled from CNTO1959PSA3001 (NCT03162796) and CNTO1959PSA3002 (NCT03158285) studies. Participants with dactylitis resolution at Week 24 and did not meet any TF criteria before Week 24 considered responders. Participants who met 1/more TF criteria or with missing data considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 154 | 160 | 159
percentage of participants | 42.2 | 59.4 | 63.5
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.030, Cochran-Mantel-Haenszel; Difference in response rates = 18.0, 95% CI 2-sided [7.4 to 28.6]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.011, Cochran-Mantel-Haenszel; Difference in response rates = 21.3, 95% CI 2-sided [10.5 to 32.0]

9. Secondary Outcome: Change From Baseline in Enthesitis Score (Based on LEI) at Week 24 Among the Participants With Enthesitis at Baseline
Description: Enthesitis was assessed using the LEI, a tool developed to assess enthesitis in participants with PsA and evaluates the presence (score of 1) or absence (score of 0) of pain by applying local pressure to the following entheses: left and right lateral epicondyle humerus, left and right medial femoral condyle, and left and right achilles tendon insertion. The enthesitis index score is a total score of the 6 evaluated sites from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). Negative changes from baseline indicate improvement of enthesitis. The outcome measure was planned to be reported for pooled population from CNTO1959PSA3001 and CNTO1959PSA3002 studies.
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1 among participants with enthesitis at baseline pooled from both CNTO1959PSA3001 (NCT03162796) and CNTO1959PSA3002 (NCT03158285) studies. Data after meeting 1 or more TF criteria were imputed as no change from baseline. Missing data were assumed missing at random and imputed using multiple imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 255 | 230 | 243
units on a scale | -1.02 [-1.22 to -0.82] | -1.52 [-1.73 to -1.31] | -1.59 [-1.79 to -1.38]
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, ANCOVA — Nominal; LS Mean Difference = -0.50, 95% CI 2-sided [-0.77 to -0.23]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, ANCOVA — Nominal; LS Mean Difference = -0.57, 95% CI 2-sided [-0.83 to -0.31]

10. Secondary Outcome: Change From Baseline in Dactylitis Scores at Week 24 Among the Participants With Dactylitis at Baseline
Description: The presence and severity of dactylitis was assessed in both hands and feet using a scoring system from 0 to 3 (0-no dactylitis, 1-mild dactylitis, 2-moderate dactylitis, and 3-severe dactylitis) for each digit. The results were summed to produce a final score ranging from 0 to 60. Higher score indicates more severe dactylitis. Negative changes from baseline indicate improvement of dactylitis. The outcome measure was planned to be reported for pooled population from CNTO1959PSA3001 and CNTO1959PSA3002 studies.
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1 among participants with dactylitis at baseline pooled from both from CNTO1959PSA3001 (NCT03162796) and CNTO1959PSA3002 (NCT03158285) studies. Data after meeting 1 or more TF criteria were imputed as no change from baseline. Missing data were assumed missing at random and imputed using multiple imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 154 | 160 | 159
units on a scale | -4.21 [-5.05 to -3.36] | -6.10 [-6.92 to -5.27] | -5.97 [-6.84 to -5.11]
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, ANCOVA — Nominal; LS Mean Difference = -1.89, 95% CI 2-sided [-2.99 to -0.79]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.002, ANCOVA — Nominal; LS Mean Difference = -1.77, 95% CI 2-sided [-2.87 to -0.66]

11. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) Score at Week 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The PCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale | 3.42 [2.53 to 4.32] | 7.39 [6.50 to 8.29] | 7.04 [6.14 to 7.94]
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.011, ANCOVA; LS Mean difference = 3.97, 95% CI 2-sided [2.75 to 5.20]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.011, ANCOVA; LS Mean difference = 3.62, 95% CI 2-sided [2.39 to 4.85]

12. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS28) (C-reactive Protein [CRP]) Score at Week 24
Description: The Disease Activity Index Score (DAS28) based on C-Reactive Protein (CRP) is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. Negative changes from baseline indicate improvement of arthritis.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale | -0.97 [-1.11 to -0.84] | -1.59 [-1.72 to -1.45] | -1.62 [-1.76 to -1.49]
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, ANCOVA — Nominal; LS Mean difference = -0.61, 95% CI 2-sided [-0.80 to -0.43]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, ANCOVA — Nominal; LS Mean difference = -0.65, 95% CI 2-sided [-0.83 to -0.47]

13. Secondary Outcome: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Mental Component Summary (MCS) at Week 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The MCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline and Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale | 2.14 [1.07 to 3.22] | 4.17 [3.10 to 5.23] | 4.22 [3.14 to 5.29]
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p = 0.072, ANCOVA; LS Mean difference = 2.02, 95% CI 2-sided [0.56 to 3.49]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p = 0.072, ANCOVA; LS Mean difference = 2.07, 95% CI 2-sided [0.60 to 3.54]

14. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 50 Response at Week 16
Description: ACR 50 response was defined as >= 50% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=50% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI; a 20-question instrument assessing 8 functional areas; range: 0-3, 0=no difficulty, 3=inability to perform a task in that area), and CRP.
Time Frame: Week 16
Population: Analysis population is FAS1. Participants who achieved ACR 50 response at Week 16 and did not meet any TF criteria before Week 16 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants | 9.3 | 28.6 | 20.8
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 19.3, 95% CI 2-sided [12.6 to 25.9]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 11.5, 95% CI 2-sided [5.2 to 17.7]

15. Secondary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 70 Response at Week 24
Description: ACR 70 response was defined as >= 70% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=70% improvement from baseline in 3 of 5 assessments: patient's assessment of pain using visual analog scale (VAS; 0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI; a 20-question instrument assessing 8 functional areas; range: 0-3, 0=no difficulty, 3=inability to perform a task in that area), and CRP.
Time Frame: Week 24
Population: Analysis population is FAS1. Participants who achieved ACR 70 response at Week 24 and did not meet any TF criteria before Week 24 were considered as responders. Participants who met 1 or more TF criteria or with missing data were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants | 4.1 | 18.5 | 13.1
Statistical Analysis 1: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q8w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 14.5, 95% CI 2-sided [9.1 to 19.9]
Statistical Analysis 2: Comparison: Placebo to Guselkumab 100 mg q4w vs Guselkumab 100 mg q4w; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — Nominal; Difference in percentage = 9.0, 95% CI 2-sided [4.1 to 13.8]

16. Secondary Outcome: Percentage of Participants Who Achieved ACR 20 Response Through Week 24
Description: as for outcome 5
Time Frame: Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved ACR 20 response at a specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Week 2 | 8.1 | 10.1 | 10.6
  Week 4 | 11.8 | 19.8 | 21.6
  Week 8 | 17.5 | 39.1 | 40.0
  Week 12 | 26.4 | 49.6 | 51.0
  Week 16 | 33.7 | 55.2 | 55.9
  Week 20 | 29.7 | 62.9 | 58.8
  Week 24 | 32.9 | 64.1 | 63.7

17. Secondary Outcome: Percentage of Participants Who Achieved ACR 50 Response Through Week 24
Description: as for outcome 14
Time Frame: Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved ACR 50 response at a specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Week 2 | 0.4 | 1.6 | 0.4
  Week 4 | 1.2 | 4.0 | 3.3
  Week 8 | 4.1 | 10.1 | 11.0
  Week 12 | 6.1 | 19.0 | 16.7
  Week 16 | 9.3 | 28.6 | 20.8
  Week 20 | 16.3 | 31.5 | 29.8
  Week 24 | 14.2 | 31.5 | 33.1

18. Secondary Outcome: Percentage of Participants Who Achieved ACR 70 Response Through Week 24
Description: as for outcome 15
Time Frame: Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved ACR 70 response at a specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Week 2 | 0 | 0 | 0
  Week 4 | 0.8 | 0.4 | 0.8
  Week 8 | 0.8 | 3.6 | 2.0
  Week 12 | 0.4 | 8.1 | 4.9
  Week 16 | 0.8 | 13.7 | 8.2
  Week 20 | 3.3 | 15.3 | 13.9
  Week 24 | 4.1 | 18.5 | 13.1

19. Secondary Outcome: Percent Change From Baseline in ACR Components at Weeks 2, 4, 8, 12, 16, 20 and 24
Description: ACR components include swollen joint count (66 joints), tender joint count (68 joints), patient's assessment of pain using visual analog scale (VAS; 0-10 cm, 0=no pain and 10=worst possible pain), patient's global assessment (PtGA) of disease activity (arthritis, VAS; 0-10 cm, 0=excellent and 10= poor), physician's global assessment (PGA) of disease activity (VAS; 0-10 cm, 0=no arthritis activity and 10=extremely active arthritis), patient's assessment of physical function measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI; a 20-question instrument assessing 8 functional areas; range: 0-3, 0=no difficulty, 3=inability to perform a task in that area), and CRP (milligram/deciliter [mg/dL]).
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Here 'n' (number analyzed) signifies number of participants with observed data regardless meeting TF criteria at specified categories.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percent change
  Week 2: Swollen Joint Count: number analyzed (Participants) | 242 | 245 | 239
  Week 2: Swollen Joint Count | -18.9 (32.16) | -18.8 (39.68) | -18.5 (38.38)
  Week 4: Swollen Joint Count: number analyzed (Participants) | 245 | 246 | 240
  Week 4: Swollen Joint Count | -27.1 (37.29) | -30.5 (36.92) | -33.6 (37.57)
  Week 8: Swollen Joint Count: number analyzed (Participants) | 246 | 246 | 243
  Week 8: Swollen Joint Count | -37.4 (39.03) | -46.8 (40.68) | -46.7 (37.69)
  Week 12: Swollen Joint Count: number analyzed (Participants) | 246 | 246 | 242
  Week 12: Swollen Joint Count | -46.1 (41.20) | -57.6 (39.22) | -58.3 (35.42)
  Week 16: Swollen Joint Count: number analyzed (Participants) | 245 | 244 | 240
  Week 16: Swollen Joint Count | -48.6 (43.01) | -64.1 (35.46) | -63.7 (34.42)
  Week 20: Swollen Joint Count: number analyzed (Participants) | 243 | 243 | 236
  Week 20: Swollen Joint Count | -54.2 (41.70) | -69.3 (33.63) | -71.4 (30.42)
  Week 24: Swollen Joint Count: number analyzed (Participants) | 243 | 243 | 240
  Week 24: Swollen Joint Count | -53.9 (45.54) | -71.3 (34.06) | -73.1 (30.67)
  Week 2: Tender Joint Count: number analyzed (Participants) | 242 | 245 | 239
  Week 2: Tender Joint Count | -9.4 (25.99) | -10.4 (40.31) | -14.8 (28.31)
  Week 4: Tender Joint Count: number analyzed (Participants) | 245 | 246 | 240
  Week 4: Tender Joint Count | -14.1 (36.04) | -15.0 (41.57) | -22.6 (32.91)
  Week 8: Tender Joint Count: number analyzed (Participants) | 246 | 246 | 243
  Week 8: Tender Joint Count | -21.9 (37.83) | -31.0 (42.36) | -33.8 (37.58)
  Week 12: Tender Joint Count: number analyzed (Participants) | 246 | 246 | 242
  Week 12: Tender Joint Count | -30.4 (37.57) | -40.9 (42.73) | -43.0 (35.90)
  Week 16: Tender Joint Count: number analyzed (Participants) | 245 | 244 | 240
  Week 16: Tender Joint Count | -30.6 (41.87) | -47.0 (40.96) | -48.1 (37.01)
  Week 20: Tender Joint Count: number analyzed (Participants) | 243 | 243 | 236
  Week 20: Tender Joint Count | -33.9 (44.22) | -53.9 (37.83) | -54.2 (35.43)
  Week 24: Tender Joint Count: number analyzed (Participants) | 243 | 243 | 240
  Week 24: Tender Joint Count | -33.3 (44.87) | -54.2 (37.15) | -57.3 (34.98)
  Week 2: Patient's Assessment of Pain: number analyzed (Participants) | 244 | 246 | 240
  Week 2: Patient's Assessment of Pain | 0.05 (35.794) | -8.92 (32.374) | -4.66 (32.229)
  Week 4: Patient's Assessment of Pain: number analyzed (Participants) | 246 | 247 | 240
  Week 4: Patient's Assessment of Pain | -0.64 (35.849) | -12.58 (33.065) | -7.96 (37.958)
  Week 8: Patient's Assessment of Pain: number analyzed (Participants) | 246 | 245 | 243
  Week 8: Patient's Assessment of Pain | -6.76 (34.213) | -21.61 (36.705) | -17.05 (44.783)
  Week 12: Patient's Assessment of Pain: number analyzed (Participants) | 246 | 246 | 242
  Week 12: Patient's Assessment of Pain | -9.01 (36.061) | -26.26 (40.223) | -25.91 (37.862)
  Week 16: Patient's Assessment of Pain(0-10cm): number analyzed (Participants) | 245 | 244 | 240
  Week 16: Patient's Assessment of Pain(0-10cm) | -9.70 (41.673) | -31.94 (42.882) | -27.85 (38.913)
  Week 20: Patient's Assessment of Pain: number analyzed (Participants) | 244 | 243 | 237
  Week 20: Patient's Assessment of Pain | -10.85 (46.497) | -35.16 (39.471) | -35.35 (39.016)
  Week 24: Patient's Assessment of Pain: number analyzed (Participants) | 243 | 243 | 240
  Week 24: Patient's Assessment of Pain | -11.84 (48.324) | -38.06 (40.565) | -36.52 (38.423)
  Week 2: PtGA of Disease Activity: number analyzed (Participants) | 244 | 246 | 240
  Week 2: PtGA of Disease Activity | -1.12 (35.882) | -10.15 (31.060) | -5.25 (32.658)
  Week 4: PtGA of Disease Activity: number analyzed (Participants) | 246 | 247 | 240
  Week 4: PtGA of Disease Activity | -2.27 (34.291) | -12.71 (34.440) | -11.02 (33.605)
  Week 8: PtGA of Disease Activity: number analyzed (Participants) | 246 | 245 | 243
  Week 8: PtGA of Disease Activity | -6.51 (35.908) | -21.58 (33.697) | -19.13 (40.545)
  Week 12: PtGA of Disease Activity: number analyzed (Participants) | 246 | 246 | 242
  Week 12: PtGA of Disease Activity | -9.30 (37.185) | -27.86 (38.900) | -28.33 (34.058)
  Week 16: PtGA of Disease Activity: number analyzed (Participants) | 245 | 244 | 240
  Week 16: PtGA of Disease Activity | -12.34 (39.207) | -32.25 (40.056) | -28.60 (39.759)
  Week 20: PtGA of Disease Activity: number analyzed (Participants) | 244 | 243 | 237
  Week 20: PtGA of Disease Activity | -12.52 (42.498) | -35.31 (36.205) | -35.11 (37.791)
  Week 24: PtGA of Disease Activity: number analyzed (Participants) | 243 | 243 | 240
  Week 24: PtGA of Disease Activity | -13.87 (45.650) | -37.05 (38.372) | -34.13 (51.445)
  Week 2: PGA of Disease Activity: number analyzed (Participants) | 240 | 241 | 231
  Week 2: PGA of Disease Activity | -9.79 (25.687) | -15.06 (27.150) | -13.85 (23.307)
  Week 4: PGA of Disease Activity: number analyzed (Participants) | 243 | 245 | 239
  Week 4: PGA of Disease Activity | -16.63 (27.573) | -23.72 (27.658) | -22.32 (28.183)
  Week 8: PGA of Disease Activity: number analyzed (Participants) | 244 | 244 | 240
  Week 8: PGA of Disease Activity | -23.29 (28.416) | -36.54 (31.224) | -37.99 (29.970)
  Week 12: PGA of Disease Activity: number analyzed (Participants) | 245 | 243 | 242
  Week 12: PGA of Disease Activity | -27.63 (32.379) | -46.54 (30.489) | -42.84 (31.305)
  Week 16: PGA of Disease Activity: number analyzed (Participants) | 245 | 244 | 240
  Week 16: PGA of Disease Activity | -31.11 (32.023) | -52.02 (31.915) | -49.18 (31.383)
  Week 20: PGA of Disease Activity: number analyzed (Participants) | 240 | 243 | 234
  Week 20: PGA of Disease Activity | -34.13 (36.576) | -54.32 (30.941) | -54.59 (29.336)
  Week 24: PGA of Disease Activity: number analyzed (Participants) | 243 | 242 | 238
  Week 24: PGA of Disease Activity | -36.59 (33.740) | -57.22 (32.480) | -58.70 (28.255)
  Week 2: HAQ-DI Score: number analyzed (Participants) | 240 | 236 | 237
  Week 2: HAQ-DI Score | -0.3191 (36.62364) | -6.3577 (50.81980) | -0.2385 (57.44896)
  Week 4: HAQ-DI Score: number analyzed (Participants) | 242 | 237 | 237
  Week 4: HAQ-DI Score | -2.8744 (46.90795) | -9.1272 (53.41051) | -5.1209 (85.16625)
  Week 8: HAQ-DI Score: number analyzed (Participants) | 242 | 235 | 240
  Week 8: HAQ-DI Score | -5.0965 (39.89566) | -12.7684 (67.23239) | -9.8081 (86.78973)
  Week 12: HAQ-DI Score: number analyzed (Participants) | 242 | 236 | 239
  Week 12: HAQ-DI Score | -8.0811 (46.90093) | -18.0336 (66.96524) | -17.7758 (67.44643)
  Week 16: HAQ-DI Score: number analyzed (Participants) | 241 | 235 | 237
  Week 16: HAQ-DI Score | -7.1776 (48.33253) | -19.3627 (70.83578) | -26.6732 (53.14973)
  Week 20: HAQ-DI Score: number analyzed (Participants) | 240 | 234 | 234
  Week 20: HAQ-DI Score | -10.4296 (50.87958) | -24.9496 (64.86820) | -28.9317 (60.67279)
  Week 24: HAQ-DI Score: number analyzed (Participants) | 239 | 233 | 237
  Week 24: HAQ-DI Score | -6.7995 (54.78602) | -25.2578 (63.15450) | -33.8837 (51.59441)
  Week 2: CRP: number analyzed (Participants) | 246 | 247 | 242
  Week 2: CRP | 86.677 (645.0281) | 0.935 (91.3783) | 10.664 (132.5947)
  Week 4: CRP: number analyzed (Participants) | 242 | 244 | 236
  Week 4: CRP | 28.042 (208.6385) | -16.885 (79.3501) | 1.128 (168.9301)
  Week 8: CRP: number analyzed (Participants) | 240 | 240 | 241
  Week 8: CRP | 45.451 (322.4433) | -11.214 (150.1689) | -17.474 (112.3803)
  Week 12: CRP: number analyzed (Participants) | 241 | 242 | 236
  Week 12: CRP | 47.034 (313.9875) | -25.620 (97.1384) | -22.277 (122.3489)
  Week 16: CRP: number analyzed (Participants) | 241 | 239 | 238
  Week 16: CRP | 28.595 (237.6660) | -19.874 (134.5210) | -26.592 (86.8465)
  Week 20: CRP: number analyzed (Participants) | 241 | 239 | 236
  Week 20: CRP | 42.282 (284.1330) | -13.551 (193.3814) | -28.701 (83.0912)
  Week 24: CRP: number analyzed (Participants) | 240 | 243 | 239
  Week 24: CRP | 19.263 (149.5120) | -27.470 (109.5239) | -28.125 (87.7229)

20. Secondary Outcome: Change From Baseline in HAQ-DI Score at Weeks 2, 4, 8, 12, 16, 20 and 24
Description: HAQ-DI score assess functional status of participant. It is a 20 question instrument that assess the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3 where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning. Negative changes from baseline indicate improvement of physical function.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 2 | -0.0594 [-0.1023 to -0.0165] | -0.1423 [-0.1850 to -0.0997] | -0.0795 [-0.1226 to -0.0364]
  Week 4 | -0.0722 [-0.1196 to -0.0247] | -0.1472 [-0.1944 to -0.1000] | -0.1605 [-0.2081 to -0.1128]
  Week 8 | -0.0942 [-0.1464 to -0.0420] | -0.2294 [-0.2815 to -0.1773] | -0.2336 [-0.2859 to -0.1813]
  Week 12 | -0.1332 [-0.1875 to -0.0790] | -0.2870 [-0.3411 to -0.2330] | -0.3010 [-0.3554 to -0.2466]
  Week 16 | -0.1167 [-0.1753 to -0.0582] | -0.3177 [-0.3760 to -0.2595] | -0.3442 [-0.4029 to -0.2855]
  Week 20 | -0.1565 [-0.2163 to -0.0968] | -0.3536 [-0.4131 to -0.2941] | -0.4019 [-0.4618 to -0.3420]
  Week 24 | -0.1300 [-0.1912 to -0.0687] | -0.3672 [-0.4282 to -0.3062] | -0.4004 [-0.4617 to -0.3390]

21. Secondary Outcome: Percentage of Participants Who Achieved >=0.35 Improvement From Baseline in HAQ-DI Score Through Week 24 Among Participants With HAQ-DI Score >=0.35 at Baseline
Description: HAQ-DI score assess functional status of participant. It is a 20 question instrument that assess the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3, where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning and a decrease of 0.35 from baseline in HAQ-DI score indicates a meaningful improvement.
Time Frame: Weeks 2, 4, 8, 12, 16, 20 and 24
Population: FAS1 among participants with HAQ-DI >=0.35 at baseline. Participants with HAQ-DI >=0.35 improvement from baseline at specific timepoint and did not meet any TF criteria before, were considered responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 236 | 228 | 228
percentage of participants
  Week 2 | 19.9 | 30.7 | 23.2
  Week 4 | 23.7 | 32.0 | 35.1
  Week 8 | 28.0 | 43.4 | 42.5
  Week 12 | 31.8 | 47.4 | 46.9
  Week 16 | 30.9 | 50.0 | 51.8
  Week 20 | 38.6 | 48.7 | 53.1
  Week 24 | 31.4 | 50.0 | 56.1

22. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 (CRP) Response Through Week 24
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. DAS 28 (CRP) response criteria was defined as follows: Good response: <=3.2 at visit and >1.2 improvement; Moderate response: >3.2 at visit and >1.2 improvement or <=5.1 at visit and >0.6-1.2 improvement; No response: <=0.6 improvement, or >5.1 at visit and <=1.2 improvement. The values are 0=best to 10=worst. A DAS28 (CRP) responder is defined as achieving a good or moderate DAS28 response at a specific visit.
Time Frame: Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved a DAS28 (CRP) response at a specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Week 2 | 21.5 | 23.8 | 24.5
  Week 4 | 32.9 | 38.7 | 40.8
  Week 8 | 38.6 | 56.9 | 54.7
  Week 12 | 51.2 | 67.3 | 65.7
  Week 16 | 51.2 | 69.8 | 72.7
  Week 20 | 50.4 | 75.0 | 76.3
  Week 24 | 52.4 | 75.4 | 80.0

23. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 (CRP) Remission Through Week 24
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. DAS 28 (CRP) remission was defined as DAS 28 (CRP) value <2.6 at the analysis visit.
Time Frame: Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved a DAS28 (CRP) remission at a specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Week 2 | 0.8 | 2.4 | 2.4
  Week 4 | 2.0 | 5.2 | 4.9
  Week 8 | 0.8 | 10.5 | 9.0
  Week 12 | 6.1 | 14.1 | 11.8
  Week 16 | 6.5 | 18.5 | 16.3
  Week 20 | 9.8 | 23.0 | 21.2
  Week 24 | 8.5 | 24.6 | 23.3

24. Secondary Outcome: Change From Baseline in DAS28 (CRP) at Weeks 2, 4, 8, 12, 16, 20 and 24
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. Negative changes from baseline indicate improvement of arthritis.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 2 | -0.29 [-0.37 to -0.21] | -0.42 [-0.50 to -0.33] | -0.43 [-0.51 to -0.35]
  Week 4 | -0.44 [-0.53 to -0.35] | -0.62 [-0.71 to -0.53] | -0.65 [-0.74 to -0.55]
  Week 8 | -0.59 [-0.71 to -0.48] | -0.99 [-1.11 to -0.88] | -0.98 [-1.09 to -0.86]
  Week 12 | -0.85 [-0.97 to -0.73] | -1.27 [-1.39 to -1.15] | -1.22 [-1.35 to -1.10]
  Week 16 | -0.88 [-1.01 to -0.75] | -1.39 [-1.52 to -1.26] | -1.37 [-1.50 to -1.24]
  Week 20 | -1.00 [-1.13 to -0.87] | -1.52 [-1.65 to -1.38] | -1.56 [-1.70 to -1.43]
  Week 24 | -0.97 [-1.11 to -0.84] | -1.59 [-1.72 to -1.45] | -1.62 [-1.76 to -1.49]

25. Secondary Outcome: Percentage of Participants Who Achieved a Response Based on Modified Psoriatic Arthritis Responder Criteria (PsARC) Through Week 24
Description: The modified PsARC response was defined as improvement in at least 2 of the four criteria: >=30% decrease in swollen joint count, >=30% decrease in tender joint count, >=20% improvement in patient's Global Assessment of Disease Activity (arthritis) on a VAS (0-100 mm, 0=excellent and 100= poor), >=20% improvement in physician's Global Assessment of Disease Activity using VAS (VAS: 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), and at least one of the 2 joint criteria with no deterioration in the other criteria.
Time Frame: Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Analysis population is FAS1. Participants who achieved a modified PsARC response at a specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Week 2 | 13.0 | 22.2 | 18.0
  Week 4 | 27.2 | 32.7 | 29.8
  Week 8 | 35.8 | 48.8 | 50.2
  Week 12 | 40.7 | 60.9 | 60.8
  Week 16 | 44.7 | 66.5 | 66.5
  Week 20 | 46.7 | 72.2 | 69.0
  Week 24 | 44.7 | 72.6 | 68.6

26. Secondary Outcome: Percentage of Participants With Resolution of Enthesitis Through Week 24 Among the Participants With Enthesitis at Baseline
Description: Enthesitis was assessed using the LEI, a tool developed to assess enthesitis in participants with PsA and evaluates the presence (score of 1) or absence (score of 0) of pain by applying local pressure to the following entheses: left and right lateral epicondyle humerus, left and right medial femoral condyle, and left and right achilles tendon insertion. The enthesitis index score is a total score of the 6 evaluated sites from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). A LEI score of 0 at a post baseline visit indicates resolution of enthesitis when baseline LEI>0.
Time Frame: Weeks 2, 4, 8, 16 and 24
Population: FAS1 among participants with enthesitis at baseline. Participants with enthesitis resolution at specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 178 | 158 | 170
percentage of participants
  Week 2 | 16.3 | 17.7 | 17.1
  Week 4 | 18.0 | 21.5 | 25.3
  Week 8 | 24.7 | 31.0 | 27.6
  Week 16 | 30.9 | 47.5 | 40.6
  Week 24 | 30.3 | 53.8 | 43.5

27. Secondary Outcome: Percentage of Participants With Resolution of Dactylitis Through Week 24 Among the Participants With Dactylitis at Baseline
Description: The presence and severity of dactylitis was assessed in both hands and feet using a scoring system from 0 to 3 (0-no dactylitis, 1-mild dactylitis, 2-moderate dactylitis, and 3-severe dactylitis) for each digit. The results were summed to produce a final score ranging from 0 to 60. Higher score indicates more severe dactylitis. Resolution of dactylitis was defined as a dactylitis score of 0 with the baseline dactylitis score >0.
Time Frame: Weeks 2, 4, 8, 16 and 24
Population: FAS1 among participants with dactylitis at baseline. Participants who achieved dactylitis resolution at specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 99 | 111 | 121
percentage of participants
  Week 2 | 12.1 | 13.5 | 13.2
  Week 4 | 18.2 | 19.8 | 20.7
  Week 8 | 29.3 | 30.6 | 31.4
  Week 16 | 36.4 | 45.0 | 52.1
  Week 24 | 38.4 | 56.8 | 63.6

28. Secondary Outcome: Change From Baseline in Enthesitis Score (Based on LEI) at Weeks 2, 4, 8, 16, and 24 Among the Participants With Enthesitis at Baseline
Description: Enthesitis was assessed using the LEI, a tool developed to assess enthesitis in participants with PsA and evaluates the presence (score of 1) or absence (score of 0) of pain by applying local pressure to the following entheses: left and right lateral epicondyle humerus, left and right medial femoral condyle, and left and right achilles tendon insertion. The enthesitis index score is a total score of the 6 evaluated sites from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness). Negative changes from baseline indicate improvement of enthesitis.
Time Frame: Baseline, Weeks 2, 4, 8, 16 and 24
Population: Analysis population is FAS1 among participants with enthesitis at baseline. Data after meeting 1 or more TF criteria were imputed as no change from baseline. Missing data were assumed missing at random and imputed using multiple imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 178 | 158 | 170
units on a scale
  Week 2 | -0.33 [-0.53 to -0.12] | -0.37 [-0.59 to -0.16] | -0.49 [-0.70 to -0.29]
  Week 4 | -0.46 [-0.68 to -0.24] | -0.56 [-0.79 to -0.33] | -0.69 [-0.92 to -0.47]
  Week 8 | -0.67 [-0.90 to -0.45] | -0.92 [-1.16 to -0.67] | -0.88 [-1.11 to -0.64]
  Week 16 | -0.94 [-1.18 to -0.71] | -1.37 [-1.62 to -1.12] | -1.42 [-1.66 to -1.18]
  Week 24 | -1.03 [-1.25 to -0.81] | -1.60 [-1.84 to -1.37] | -1.52 [-1.75 to -1.29]

29. Secondary Outcome: Change From Baseline in Dactylitis Scores at Weeks 2, 4, 8, 16 and 24 Among the Participants With Dactylitis at Baseline
Description: The presence and severity of dactylitis was assessed in both hands and feet using a scoring system from 0 to 3 (0-no dactylitis, 1-mild dactylitis, 2-moderate dactylitis, and 3-severe dactylitis) for each digit. The results were summed to produce a final score ranging from 0 to 60. Higher score indicates more severe dactylitis. Negative changes from baseline indicate improvement of dactylitis.
Time Frame: Baseline, Weeks 2, 4, 8, 16 and 24
Population: Analysis population is FAS1 among participants with dactylitis at baseline. Data after meeting 1 or more TF criteria were imputed as no change from baseline. Missing data were assumed missing at random and imputed using multiple imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 99 | 111 | 121
units on a scale
  Week 2 | -0.21 [-1.11 to 0.69] | -1.11 [-1.95 to -0.26] | -0.78 [-1.61 to 0.05]
  Week 4 | -1.10 [-2.07 to -0.13] | -2.11 [-3.02 to -1.20] | -1.56 [-2.47 to -0.66]
  Week 8 | -2.17 [-3.19 to -1.16] | -3.17 [-4.12 to -2.22] | -3.11 [-4.05 to -2.17]
  Week 16 | -3.40 [-4.42 to -2.38] | -4.88 [-5.84 to -3.92] | -4.80 [-5.75 to -3.85]
  Week 24 | -4.03 [-4.96 to -3.10] | -5.95 [-6.83 to -5.08] | -5.88 [-6.74 to -5.01]

30. Secondary Outcome: Change From Baseline in the Psoriatic Arthritis Disease Activity Score (PASDAS) at Weeks 8, 16 and 24
Description: PASDAS (score range of 0 to 10, where higher score indicated more severe disease) is a composite score of overall disease activity combining Patient's Global Assessment of Disease Activity (arthritis and psoriasis, using VAS [0-100 mm, 0=excellent and 100= poor), Physician's Global Assessment of Disease Activity (using VAS [0-100 mm, 0=no arthritis activity and 100=extremely active arthritis]), swollen joint count (0-66 joints), tender joint count (0-68 joints), CRP (mg/L), enthesitis based on LEI (0= 0 sites with tenderness to 6= worst possible score; 6 sites with tenderness), tender dactylitis count (scoring each digit from 0-3 [where 0= no tenderness and 3= extreme tenderness] and recoding to 0-1, where any score > 0 equaled 1), and the PCS score with score range 0-100 (higher score-better quality of life) of the SF-36 health survey. The cutoffs for disease activity were 3.2 (low) to 5.4 (high). Negative changes from baseline indicate improvement of overall disease activity.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: Analysis population is FAS1. Data after meeting 1 or more TF criteria were imputed as no change from baseline. Missing data were assumed missing at random. The LS mean is based on Mixed-effect repeated measures (MMRM) model that included data from all visits for all participants included in the model.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 8 | -0.863 [-1.007 to -0.719] | -1.452 [-1.595 to -1.309] | -1.413 [-1.557 to -1.270]
  Week 16 | -1.158 [-1.327 to -0.988] | -2.110 [-2.278 to -1.942] | -1.994 [-2.164 to -1.825]
  Week 24 | -1.336 [-1.516 to -1.156] | -2.403 [-2.582 to -2.225] | -2.399 [-2.579 to -2.219]

31. Secondary Outcome: Change From Baseline in Group for Research and Assessment of Psoriasis and Psoriatic Arthritis (GRAPPA) Composite Score (GRACE) at Weeks 16 and 24
Description: GRACE index is a composite PsA disease activity score converted from Arithmetic Mean of Desirability Function (AMDF), derived from TJC (0-68) and SJC (0-66), HAQ-DI (0-3), patient's global assessment of disease activity on arthritis and psoriasis (0-100 mm, 0=excellent and 100=poor), patient's assessment of skin disease activity (0-100 mm, 0=excellent and 100=poor), patient's global assessment of disease activity on arthritis (0-100 mm, 0=excellent and 100=poor), PASI (0-72), and PsA Quality of Life Index (derived as PsAQOL=25.355 + [2.367*HAQ-DI]-[0.234*SF-PCS]-[0.244*SF-MCS]), where HAQ-DI: HAQ-DI score (0-3, 0=least difficulty and 3=extreme difficulty), SF-PCS (Score ranges from 0-100, higher scores= better quality of life) and SF-MCS (score ranges from 0-100, higher scores= better quality of life). Total score is from 0-10, lower score=better response. Higher score indicates more active disease activity. Negative change from baseline indicates improvement of PsA disease activity.
Time Frame: Baseline, Weeks 16 and 24
Population: Analysis population is FAS1. Data after meeting 1 or more TF criteria were imputed as no change from baseline. Missing data were assumed missing at random. The LS mean is based on MMRM model that included data from all visits for all participants included in the model.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 16 | -1.029 [-1.212 to -0.847] | -2.326 [-2.507 to -2.145] | -2.214 [-2.397 to -2.032]
  Week 24 | -1.198 [-1.395 to -1.001] | -2.593 [-2.789 to -2.397] | -2.589 [-2.786 to -2.392]

32. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Scores (Percent Work Time Missed) at Weeks 16 and 24
Description: Work Productivity and Activity Impairment was assessed using the Work Productivity and Activity Impairment Questionnaire - Specific Health Problem (WPAI-SHP) of PsA (WPAI-PsA). The WPAI-PsA consisted of 6 questions to determine employment status, hours missed from work due to PsA, hours missed from work for other reasons, hours actually worked, the degree to which PsA affected work productivity while at work and the degree to which PsA affected activities outside of work during the past 7 days. WPAI outcomes included percent work time missed due to PsA, percent impairment while working due to PsA, percent overall work impairment due to PsA, and percent activity impairment outside of work due to PsA. These WPAI outcomes were expressed as impairment percentages (0-100, 0=no impairment and 100=100% impaired), with higher numbers indicating greater impairment and less productivity. Negative changes from baseline indicate improvement of work productivity and activity impairment.
Time Frame: Baseline, Weeks 16 and 24
Population: Analysis population is FAS1. Data after meeting 1/more TF criteria imputed as no change from baseline. Missing data assumed MAR. LS mean is based on MMRM model that included data from all visits for all participants included in model. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of work time missed
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 155 | 145 | 145
percentage of work time missed
  Week 16 | -4.553 [-7.199 to -1.906] | -3.451 [-6.199 to -0.703] | -4.717 [-7.449 to -1.985]
  Week 24 | -3.491 [-6.403 to -0.578] | -3.103 [-6.062 to -0.144] | -3.827 [-6.826 to -0.828]

33. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Scores (Percent Impairment While Working) at Weeks 16 and 24
Description: as for outcome 32
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 32
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of impairment
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 131 | 129 | 133
percentage of impairment
  Week 16 | -10.281 [-13.887 to -6.675] | -16.054 [-19.699 to -12.409] | -15.083 [-18.655 to -11.511]
  Week 24 | -10.157 [-13.663 to -6.650] | -19.366 [-22.857 to -15.875] | -19.492 [-22.982 to -16.003]

34. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Scores (Percent Overall Work Impairment) at Weeks 16 and 24
Description: as for outcome 32
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 32
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of overall work impairment
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 131 | 129 | 133
percentage of overall work impairment
  Week 16 | -11.232 [-14.962 to -7.501] | -15.926 [-19.694 to 12.159] | -15.808 [-19.501 to -12.115]
  Week 24 | -10.869 [-14.591 to -7.147] | -19.711 [-23.416 to -16.006] | -20.023 [-23.726 to -16.320]

35. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Scores (Percent Activity Impairment Outside of Work ) at Weeks 16 and 24
Description: as for outcome 32
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 32
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of activity impairment
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 244 | 247 | 245
percentage of activity impairment
  Week 16 | -10.569 [-13.262 to -7.877] | -17.107 [-19.787 to -14.428] | -17.029 [-19.727 to -14.331]
  Week 24 | -10.320 [-13.071 to -7.570] | -21.467 [-24.204 to -18.729] | -20.480 [-23.226 to -17.734]

36. Secondary Outcome: Change From Baseline in Modified Composite Psoriatic Disease Activity Index (mCPDAI) Score at Week 16 and 24
Description: The mCPDAI assessed 4 domains (joints, skin, entheses, and dactylitis). The mCPDAI scores were calculated using the following assessments: joints (66 swollen and 68 tender joint counts), HAQ-DI score, PASI, dactylitis, and enthesitis. Within each domain a score (range 0-3) was assigned, where 0= Not involved, 1= Mild, 2= Moderate and 3= Severe. The scores for each domain were then added together to give a final score range of 0 to 12. A higher score indicates more active disease activity. Negative changes from baseline indicate improvement of PsA disease activity.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 16 | -1.18 [-1.43 to -0.93] | -2.39 [-2.64 to -2.14] | -2.57 [-2.82 to -2.31]
  Week 24 | -1.30 [-1.57 to -1.04] | -2.94 [-3.20 to -2.68] | -3.09 [-3.35 to -2.83]

37. Secondary Outcome: Change From Baseline in Disease Activity Index for Psoriatic Arthritis (DAPSA) at Weeks 2, 4, 8, 12, 16, 20 and 24
Description: DAPSA assessed the joint domain of PsA and was derived from the sum of the following components: tender joint count (0-68), swollen joint count (0-66), CRP level (mg/dL, value <lower limit of quantification [LLOQ] is considered equal to half of the value of LLOQ for numerical calculations), patient assessment of pain (0-10cm VAS, 0=no pain, 10=worst possible pain), and patient's global assessment of disease activity on arthritis (0 to 10cm VAS, 0=excellent and 10=poor). A higher score indicates more active disease activity. Negative changes from baseline indicate improvement of PsA disease activity. The assessment does not have a score range with an upper or lower bound.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 2 | -4.6447 [-5.9287 to -3.3607] | -6.7838 [-8.0642 to -5.5034] | -6.3783 [-7.6664 to -5.0902]
  Week 4 | -7.6695 [-9.2194 to -6.1197] | -9.9687 [-11.5128 to -8.4246] | -10.2484 [-11.8049 to -8.6919]
  Week 8 | -10.4480 [-12.1877 to -8.7084] | -15.3303 [-17.0682 to -13.5924] | -15.8657 [-17.6038 to -14.1277]
  Week 12 | -14.2915 [-16.1107 to -12.4724] | -18.9772 [-20.7912 to -17.1632] | -19.9687 [-21.7915 to -18.1459]
  Week 16 | -14.8556 [-16.8664 to -12.8448] | -21.6939 [-23.6979 to -19.6899] | -21.4722 [-23.4873 to -19.4571]
  Week 20 | -16.1375 [-18.1165 to -14.1586] | -23.3163 [-25.2890 to -21.3436] | -24.6844 [-26.6691 to -22.6997]
  Week 24 | -15.8489 [-17.9229 to -13.7750] | -24.0359 [-26.1019 to -21.9699] | -25.1583 [-27.2341 to -23.0824]

38. Secondary Outcome: Percentage of Participants Who Achieved Minimal Disease Activity (MDA) Criteria Through Week 24
Description: MDA is a measure that defines a satisfactory state of disease activity that includes the 5 domains of PsA (joint symptoms, skin psoriasis, patient's perspective of pain and disease activity, physical function, and enthesitis). A participant was considered as having achieved the PsA MDA at a visit if the participant has fulfilled at least 5 of the following 7 criteria at that visit: Tender joint count (68 joints)<=1, Swollen joint count (66 joints) <=1, Psoriasis activity and severity index <=1, Patient's Assessment of Pain <=15 on a 100-unit VAS, Patient's Global Assessment of Disease Activity (arthritis and psoriasis) <=20 on a 100-unit VAS, HAQ-DI score <=0.5, and Tender entheseal points <= 1 (LEI index score <= 1).
Time Frame: Weeks 16 and 24
Population: Analysis population is FAS1. Participants who achieved MDA at a specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Week 16 | 3.3 | 16.9 | 13.1
  Week 24 | 6.1 | 25.0 | 18.8

39. Secondary Outcome: Percentage of Participants Who Achieved >= 20%, >=50%, >=70%, and >=90% Improvement From Baseline in BASDAI Score Through Week 24 Among the Participants With Spondylitis and Peripheral Arthritis and BASDAI Score >0 at Baseline
Description: Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) is a self-assessment tool that consists of 6 questions relating to the 5 major symptoms of ankylosing spondylitis: fatigue, spinal pain, joint pain, enthesitis, qualitative morning stiffness and quantitative morning stiffness. The first 5 items were scored on a 10 centimeter (cm) VAS ranging from 0=none to 10=very severe. Quantitative morning stiffness was scored on a 10cm VAS ranging from 0=0 hours to 10=2 or more hours. The 2 scores for qualitative and quantitative morning stiffness were averaged, and the total BASDAI score was the average of the 5 scores of each symptom, ranging from 0 (none) to 10 (very severe). Higher scores indicate greater disease severity and an improvement of 50% from baseline is considered clinically meaningful. Only participants with spondylitis and peripheral arthritis as their primary arthritic presentation of PsA completed the BASDAI indicate the degree of their symptoms over the past week.
Time Frame: Weeks 8, 16 and 24
Population: FAS1 with spondylitis and peripheral arthritis and BASDAI score >0 at baseline. Participants with the specified improvement in BASDAI at specific time point and did not meet TF criteria before, considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 92 | 67 | 83
percentage of participants
  Week 8: Participants with >=20% Improvement | 38.0 | 46.3 | 53.0
  Week 16: Participants with >=20% Improvement | 39.1 | 58.2 | 69.9
  Week 24: Participants with >=20% Improvement | 42.4 | 59.7 | 68.7
  Week 8: Participants with >=50% Improvement | 6.5 | 17.9 | 18.1
  Week 16: Participants with >=50% Improvement | 17.4 | 37.3 | 26.5
  Week 24: Participants with >=50% Improvement | 21.7 | 38.8 | 37.3
  Week 8: Participants with >=70% Improvement | 3.3 | 11.9 | 4.8
  Week 16: Participants with >=70% Improvement | 5.4 | 23.9 | 9.6
  Week 24: Participants with >=70% Improvement | 8.7 | 20.9 | 15.7
  Week 8: Participants with >=90% Improvement | 0 | 1.5 | 0
  Week 16: Participants with >=90% Improvement | 1.1 | 0 | 2.4
  Week 24: Participants with >=90% Improvement | 2.2 | 1.5 | 3.6

40. Secondary Outcome: Percentage of Participants Who Achieved PASI 75 Response Through Week 24 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. A PASI 75 response: >=75% improvement in PASI score from baseline.
Time Frame: Weeks 16 and 24
Population: FAS1 among participants with >=3% BSA of psoriasis and IGA score >=2 at baseline. Participants with PASI 75 response at specific time point and did not meet any TF criteria before, were considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 183 | 176 | 184
percentage of participants
  Week 16 | 18.6 | 73.3 | 73.9
  Week 24 | 23.0 | 79.0 | 78.3

41. Secondary Outcome: Percentage of Participants Who Achieved PASI 90 Response Through Week 24 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. A PASI 90 response: >=90% improvement in PASI score from baseline.
Time Frame: Weeks 16 and 24
Population: FAS1 among participants with >=3% BSA of psoriasis and IGA score >=2 at baseline. Participants with PASI 90 response at specific time point and did not meet any TF criteria before, were considered responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 183 | 176 | 184
percentage of participants
  Week 16 | 8.2 | 55.1 | 53.8
  Week 24 | 9.8 | 68.8 | 60.9

42. Secondary Outcome: Percentage of Participants Who Achieved PASI 100 Response Through Week 24 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. A PASI 100 response: 100% improvement in PASI score from baseline.
Time Frame: Weeks 16 and 24
Population: FAS1 among participants with >=3% BSA of psoriasis and IGA score >=2 at baseline. Participants with PASI 100 response at specific time point and did not meet any TF criteria before, were considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 183 | 176 | 184
percentage of participants
  Week 16 | 3.8 | 27.3 | 33.2
  Week 24 | 2.7 | 45.5 | 44.6

43. Secondary Outcome: Percentage of Participants With an IGA Score of 0 (Cleared) Through Week 24 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: A psoriasis IGA response was defined as an IGA score of 0 (cleared) or 1 (minimal) and >=2 grade reduction from baseline in the IGA psoriasis score. The IGA documents the investigator's assessment of the patient's psoriasis and lesions are graded for induration, erythema and scaling, each using a 5 point scale: 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe). The IGA score of psoriasis was based upon the average of induration, erythema and scaling scores. The participant's psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: Weeks 16 and 24
Population: FAS1 among participants with >=3% BSA of psoriasis and IGA score >=2 at baseline. Participants with IGA score of 0(cleared) at specific time point and did not meet TF criteria before, were considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 183 | 176 | 184
percentage of participants
  Week 16 | 6.0 | 38.6 | 40.8
  Week 24 | 7.7 | 50.0 | 51.5

44. Secondary Outcome: Change From Baseline in PASI Score at Weeks 16 and 24 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. Negative change from baseline indicates improvement of psoriasis.
Time Frame: Baseline, Weeks 16 and 24
Population: FAS1 among participants who had >=3% BSA of psoriatic involvement and IGA score >=2 (mild) at baseline. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR. The LS mean is based on MMRM model that included data from all visits for all participants included in the model.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 183 | 176 | 184
units on a scale
  Week 16 | -3.482 [-4.346 to -2.618] | -11.151 [-12.028 to -10.274] | -11.278 [-12.153 to -10.404]
  Week 24 | -3.904 [-4.748 to -3.059] | -11.407 [-12.265 to -10.549] | -11.471 [-12.325 to -10.617]

45. Secondary Outcome: Percentage of Participants Who Achieved a DLQI Score of 0 or 1 Through Week 24 Among the Participants With DLQI Score >1, With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: Dermatology Life Quality Index (DLQI) is a 10-item instrument questionnaire used to assess the patient's perspective of the impact of psoriasis on daily living. Each item was scored on a 4-point scale (0 =not at all /not relevant; 1 =a little; 2 =a lot; 3 =very much), and the total score (0-30) is the sum of the 10 items. The higher the score, the more quality of life is impaired. A DLQI score of 0 or 1 indicates psoriasis had no effect at all on patient's life.
Time Frame: Weeks 8, 16, 24
Population: FAS1 among participants with DLQI >1, >=3% BSA of psoriasis and IGA score >=2 (mild) at baseline. Participants with DLQI score of 0/1 at specific time point and did not meet TF criteria before, considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 170 | 158 | 173
percentage of participants
  Week 8 | 7.6 | 33.5 | 26.6
  Week 16 | 10.0 | 51.3 | 45.1
  Week 24 | 11.8 | 63.9 | 59.0

46. Secondary Outcome: Percentage of Participants Who Achieved >=5-point Improvement From Baseline in DLQI Score Through Week 24 Among the Participants With DLQI Score >=5, >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: Dermatology Life Quality Index (DLQI) is a 10-item instrument questionnaire used to assess the patient's perspective of the impact of psoriasis on daily living. Each item was scored on a 4-point scale (0 =not at all /not relevant; 1 =a little; 2 =a lot; 3 =very much), and the total score (0-30) is the sum of the 10 items. The higher the score, the more quality of life is impaired. An improvement of 5 points was considered clinically meaningful.
Time Frame: Weeks 8, 16, 24
Population: FAS1 with DLQI>=5, >=3% BSA of psoriasis and IGA score >=2 (mild) at baseline. Participants with >=5-point improvement from baseline in DLQI score at specific time point and did not meet TF criteria before, considered responders at that time point. Participants who met 1/more TF criteria before or with missing data considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 143 | 132 | 152
percentage of participants
  Week 8 | 30.1 | 71.2 | 69.7
  Week 16 | 36.4 | 79.5 | 79.6
  Week 24 | 37.8 | 83.3 | 86.8

47. Secondary Outcome: Change From Baseline in DLQI Score at Weeks 8, 16 and 24 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: Dermatology Life Quality Index (DLQI) is a 10-item instrument questionnaire used to assess the patient's perspective of the impact of psoriasis on daily living. Each item was scored on a 4-point scale (0 =not at all /not relevant; 1 =a little; 2 =a lot; 3 =very much), and the total score (0-30) is the sum of the 10 items. The higher the score, the more quality of life is impaired. Negative changes from baseline indicate improvement of life quality impacted by psoriasis.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: Analysis population is FAS1 among participants with >=3% BSA of psoriasis and an IGA score >=2 (mild) at baseline. Data after meeting 1 or more TF criteria were imputed as no change from baseline. Missing data were assumed missing at random. LS mean is based on MMRM model that included data from all visits for all participants included in model.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 183 | 176 | 184
units on a scale
  Week 8 | -1.653 [-2.373 to -0.933] | -6.818 [-7.549 to -6.086] | -6.396 [-7.121 to -5.671]
  Week 16 | -2.410 [-3.109 to -1.710] | -8.545 [-9.255 to -7.835] | -8.147 [-8.853 to -7.441]
  Week 24 | -2.129 [-2.854 to -1.404] | -8.954 [-9.691 to -8.218] | -8.853 [-9.581 to -8.124]

48. Secondary Outcome: Percentage of Participants Who Achieved Both PASI 75 and ACR 20 Responses Through Week 24 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: In PASI, each area (head, trunk, upper and lower extremities) was assessed for % of area involved and translated to numeric score from 0 (no involvement) to 6 (90-100% involvement) and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI produces numeric score from 0 to 72. Higher scores=more severe disease. PASI 75: >=75% improvement in PASI score from baseline. ACR 20: >=20% improvement in swollen joint count (SJC) (66 joints) + tender joint count (TJC) (68 joints) and >=20% improvement in 3 of 5: patient's assessment of pain (VAS; 0-100 mm, 0=no pain to 100=worst possible pain), PtGA of disease activity (VAS; 0-100 mm, 0=excellent to 100=poor), PGA of disease activity (VAS; 0-100 mm, 0=no arthritis to 100=extremely active arthritis), patient's assessment of physical function (HAQ-DI -20-question instrument; range- 0=no difficulty to 3=inability to perform task) and CRP.
Time Frame: Weeks 16 and 24
Population: FAS1 participants with >=3% BSA psoriatic involvement and IGA score >=2 at baseline. Participants with both PASI75 and ACR20 responses at specific timepoint and did not meet TF criteria before, considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 183 | 176 | 184
percentage of participants
  Week 16 | 10.4 | 48.9 | 48.4
  Week 24 | 11.5 | 56.8 | 57.1

49. Secondary Outcome: Percentage of Participants Who Achieved Both PASI 75 and Modified PsARC Response Through Week 24 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: In PASI, each area (head, trunk, upper and lower extremities) was assessed separately for % of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90-100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severtiy. PASI produces numeric score range from 0 to 72. Higher scores=more severe disease. PASI 75 response: >=75% improvement in PASI score from baseline. Modified PsARC response: improvement in at least 2 of 4 criteria: >=30% decrease in SJC and TJC, >=20% improvement in PtGA of Disease Activity (arthritis) on VAS (0-100 mm, 0=excellent and 100=poor), >=20% improvement in PGA of Disease Activity on VAS (VAS: 0-100 mm, 0=no arthritis and 100=extremely active arthritis), and at least 1 of 2 joint criteria with no deterioration in other criteria.
Time Frame: Weeks 16 and 24
Population: FAS1 with >=3% BSA psoriatic involvement and IGA score >=2 at baseline. Participants with both PASI 75 and modified PsARC responses at specific timepoint and did not meet TF criteria before, considered responders at that time point. Participants who met 1/more TF criteria before or with missing data at that time point considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 183 | 176 | 184
percentage of participants
  Week 16 | 13.1 | 56.8 | 54.3
  Week 24 | 15.3 | 65.3 | 60.9

50. Secondary Outcome: Change From Baseline in Modified vdH-S Erosion Score at Week 24
Description: as for outcome 6
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1-SD. Observed data were used regardless if 1 or more TF criteria were met. Missing data were assumed to be missing at random and imputed using multiple imputation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale | 0.58 [0.33 to 0.83] | 0.36 [0.11 to 0.61] | 0.13 [-0.12 to 0.38]

51. Secondary Outcome: Change From Baseline in Modified vdH-S Joint Space Narrowing (JSN) Score at Week 24
Description: The modified vdH-S score is the sum of the erosion score (hand, feet) and joint space narrowing (JSN) score (hand, feet). The JSN score is the total JSN score in 40 joints of the two hands and 12 joints of the 2 feet. Each joint is scored from 0 to 4 with 0 indicating no JSN, and 4 indicating a complete loss of joint space, bony ankylosis, or complete luxation, for a maximum JSN score of 208. Higher score indicates more severe joint space narrowing. A positive change from baseline in the modified vdH-S JSN score indicates progression of joint space narrowing.
Time Frame: Baseline and Week 24
Population: as for outcome 50
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale | 0.37 [0.23 to 0.51] | 0.16 [0.02 to 0.30] | 0.16 [0.02 to 0.30]

52. Secondary Outcome: Change From Baseline in Modified vdH-S Score by Region and Type of Damage (ie, Hand Erosion, Hand JSN, Foot Erosion, Foot JSN Subscores) at Week 24
Description: Modified vdH-S score is the sum of the erosion score (hand, feet) and JSN score (hand, feet). Joint erosion score is the summary of erosion severity in 40 joints of hand (Hand erosion score) scored according to 0 (no erosion) to 5 (complete collapse of bone) for a maximum hand erosion score of 200, and 12 joints of 2 feet (each side of the foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum foot erosion score of 120. Higher scores indicate more joint damage. JSN score is the total JSN score in same 52 joints as above, each joint scored according to the subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum Hand JSN score of 160 and maximum Foot JSN score of 48. Higher scores indicate more joint damage. Hand Score (sum of Hand Erosion Score and Hand JSN Score) scored as 0-360 and Foot score (sum of foot erosion score and foot JSN score) scored as 0-168. Higher scores indicate more joint damage.
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1-SD. Observed data were summarized regardless if 1 or more TF criteria were met. Here, 'n' (number analyzed) signifies the number of participants analyzed for a specified score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Hand Erosion Score: number analyzed (Participants) | 245 | 247 | 240
  Hand Erosion Score | 0.40 (1.555) | 0.18 (1.280) | -0.03 (1.514)
  Hand JSN Score: number analyzed (Participants) | 245 | 247 | 240
  Hand JSN Score | 0.26 (1.106) | 0.10 (0.637) | 0.08 (0.607)
  Hand Score: number analyzed (Participants) | 245 | 247 | 240
  Hand Score | 0.66 (2.441) | 0.28 (1.649) | 0.05 (1.881)
  Foot Erosion Score: number analyzed (Participants) | 245 | 247 | 240
  Foot Erosion Score | 0.14 (0.801) | 0.15 (0.982) | 0.14 (0.894)
  Foot JSN Score: number analyzed (Participants) | 245 | 247 | 240
  Foot JSN Score | 0.10 (0.516) | 0.02 (0.516) | 0.07 (0.632)
  Foot Score: number analyzed (Participants) | 245 | 247 | 240
  Foot Score | 0.24 (1.116) | 0.17 (1.180) | 0.21 (1.210)

53. Secondary Outcome: Percentage of Participants With a Change of <=0 or <=0.5 From Baseline in Modified vdH-S Score at Week 24
Description: as for outcome 6
Time Frame: Week 24
Population: as for outcome 50
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Change of <=0 from Baseline | 64.7 | 63.5 | 67.3
  Change of <=0.5 from Baseline | 72.1 | 74.4 | 78.0

54. Secondary Outcome: Percentage of Participants With a Change of <=0 From Baseline and <=0.5 From Baseline in Modified vdH-S Erosion Score at Week 24
Description: as for outcome 6
Time Frame: Week 24
Population: as for outcome 50
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Change of <=0 from Baseline | 66.8 | 66.3 | 71.4
  Change of <=0.5 from Baseline | 72.9 | 76.8 | 80.2

55. Secondary Outcome: Percentage of Participants With a Change of <=0 From Baseline and <=0.5 From Baseline in Modified vdH-S JSN Score at Week 24
Description: The modified vdH-S score is the sum of the erosion score (hand, feet) and joint space narrowing (JSN) score (hand, feet). The JSN score is the sum of JSN score in 40 joints of the two hands and 12 joints of the 2 feet. Each joint is scored from 0 - 4 with 0 indicating no JSN, and 4 indicating a complete loss of joint space, bony ankylosis, or complete luxation, for a maximum JSN score of 208. Higher score indicates more severe joint space narrowing. Change from baseline in the modified vdH-S JSN score <=0 (assessed by both readers) or <=0.5 (assessed by at least one reader) was considered as no progression of JSN.
Time Frame: Week 24
Population: as for outcome 50
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Change of <=0 from Baseline | 78.6 | 78.8 | 80.1
  Change of <=0.5 from Baseline | 85.5 | 88.1 | 88.3

56. Secondary Outcome: Percentage of Participants Without Radiographic Progression (Based on the Smallest Detectable Change [SDC]) From Baseline at Week 24
Description: Modified vdH-S score is the sum of the erosion score (hand, feet) and JSN score (hand, feet). Joint erosion score is the summary of erosion severity in 40 joints of hand scored according to the surface area, from 0 (no erosion) to 5 (complete collapse of bone) and 12 joints of 2 feet (each side of foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum erosion score of 320. JSN score is the total JSN score in same 52 joints as above, each joint scored according to the subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum JSN score of 208. Total score ranges from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score indicates more joint damage. SDC was defined as the cut-off above which the changes can be detected beyond measurement error. Without radiographic progression was defined as change from baseline in the modified vdH-S score <=SDC of 2.18.
Time Frame: Week 24
Population: as for outcome 50
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants | 86.4 | 87.8 | 89.3

57. Secondary Outcome: Percentage of Participants Without Radiographic Joint Erosion Progression (Based on SDC) From Baseline at Week 24
Description: Modified vdH-S score is sum of erosion score (hand, feet) and JSN score (hand, feet). Joint erosion score is the summary of erosion severity in 40 joints of hand scored according to the surface area, from 0 (no erosion) to 5 (complete collapse of bone) and 12 joints of 2 feet (each side of foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum erosion score of 320. JSN score is the total JSN score in same 52 joints as above, each joint scored according to subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum JSN score of 208. Total score ranges from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score indicates more joint damage. SDC defined as the cut-off above which changes can be detected beyond measurement error. Without radiographic joint erosion progression was defined as change from baseline in modified vdH-S erosion score <=SDC of 1.83.
Time Frame: Week 24
Population: as for outcome 50
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants | 84.0 | 89.0 | 89.9

58. Secondary Outcome: Percentage of Participants Without Radiographic JSN Progression (Based on the SDC) From Baseline at Week 24
Description: The modified vdH-S score is the sum of the erosion score (hand, feet) and joint space narrowing (JSN) score (hand, feet). The JSN score is the sum of JSN score in 40 joints of the two hands and 12 joints of the 2 feet. Each joint is scored from 0 - 4 with 0 indicating no JSN, and 4 indicating a complete loss of joint space, bony ankylosis, or complete luxation, for a maximum JSN score of 208. Higher score indicates more severe joint space narrowing. The smallest detectable change (SDC) was defined as the cut-off above which the changes can be detected beyond measurement error. Without radiographic JSN progression was defined as change from baseline in the modified vdH-S JSN score <=SDC of 1.11.
Time Frame: Week 24
Population: as for outcome 50
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants | 91.3 | 93.5 | 91.7

59. Secondary Outcome: Percentage of Participants With Pencil in Cup or Gross Osteolysis Deformities at Baseline and Week 24
Description: Pencil in Cup or Gross Osteolytis Deformities are radiographic features specific for psoriatic arthritis.
Time Frame: Baseline and Week 24
Population: Analysis population is FAS1-SD. Observed data were summarized regardless if 1 or more TF criteria were met.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Baseline | 4.5 | 3.6 | 3.7
  Week 24: number analyzed (Participants) | 245 | 247 | 240
  Week 24 | 4.9 | 3.6 | 3.8

60. Secondary Outcome: Change From Baseline in SF-36 PCS Score at Weeks 8, 16 and 24
Description: as for outcome 11
Time Frame: Baseline, Weeks 8, 16 and 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 8 | 2.75 [1.98 to 3.52] | 4.83 [4.06 to 5.59] | 4.34 [3.56 to 5.1]
  Week 16 | 3.03 [2.18 to 3.88] | 6.65 [5.80 to 7.49] | 5.93 [5.07 to 6.78]
  Week 24 | 3.42 [2.53 to 4.32] | 7.39 [6.50 to 8.29] | 7.04 [6.14 to 7.94]

61. Secondary Outcome: Change From Baseline in SF-36 MCS Score at Weeks 8, 16 and 24
Description: as for outcome 13
Time Frame: Baseline, Weeks 8, 16 and 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 8 | 1.11 [0.12 to 2.09] | 2.28 [1.30 to 3.27] | 2.87 [1.89 to 3.86]
  Week 16 | 1.96 [0.91 to 3.01] | 4.28 [3.24 to 5.33] | 3.41 [2.36 to 4.47]
  Week 24 | 2.14 [1.07 to 3.22] | 4.17 [3.10 to 5.23] | 4.22 [3.14 to 5.29]

62. Secondary Outcome: Change From Baseline in Norm Based Scores of SF-36 Scales at Weeks 8, 16 and 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales: physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health. The scores 0-100 (where higher scores indicated a better quality of life) from each subscale of SF-36 were normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. Higher score indicates better health status. A positive change indicates improvement while a negative change indicates worsening of health status and quality of life.
Time Frame: Baseline and Weeks 8, 16 and 24
Population: Analysis population is FAS1. Data after meeting one or more TF criteria were imputed as no change from baseline. Missing data were assumed to be MAR. The LS mean is based on MMRM model that included data from all visits for all participants included in the model.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 8: Physical Function Score | 2.095 [1.251 to 2.940] | 3.879 [3.038 to 4.720] | 3.936 [3.090 to 4.782]
  Week 16: Physical Function Score | 2.581 [1.669 to 3.492] | 6.124 [5.218 to 7.030] | 5.618 [4.704 to 6.532]
  Week 24: Physical Function Score | 3.254 [2.310 to 4.197] | 6.703 [5.764 to 7.642] | 6.624 [5.680 to 7.567]
  Week 8: Role-physical Score | 2.619 [1.828 to 3.410] | 3.599 [2.812 to 4.387] | 3.107 [2.315 to 3.899]
  Week 16: Role-physical Score | 2.965 [2.120 to 3.810] | 5.616 [4.776 to 6.455] | 4.942 [4.095 to 5.789]
  Week 24: Role-physical Score | 3.365 [2.477 to 4.253] | 6.549 [5.666 to 7.433] | 6.241 [5.354 to 7.129]
  Week 8: Bodily Pain Score | 2.760 [1.974 to 3.546] | 5.456 [4.674 to 6.239] | 4.901 [4.115 to 5.688]
  Week 16: Bodily Pain Score | 3.086 [2.196 to 3.977] | 7.485 [6.601 to 8.369] | 6.613 [5.721 to 7.505]
  Week 24: Bodily Pain Score | 3.482 [2.556 to 4.408] | 7.811 [6.890 to 8.733] | 7.739 [6.813 to 8.664]
  Week 8: General Health Score | 1.662 [0.906 to 2.418] | 4.111 [3.358 to 4.863] | 4.174 [3.418 to 4.931]
  Week 16: General Health Score | 2.520 [1.681 to 3.358] | 5.719 [4.886 to 6.552] | 4.808 [3.967 to 5.648]
  Week 24: General Health Score | 2.290 [1.415 to 3.165] | 5.794 [4.924 to 6.665] | 5.269 [4.394 to 6.144]
  Week 8: Vitality Score | 2.505 [1.574 to 3.436] | 4.286 [3.358 to 5.213] | 4.669 [3.736 to 5.601]
  Week 16: Vitality Score | 3.554 [2.559 to 4.548] | 6.967 [5.980 to 7.955] | 5.901 [4.904 to 6.898]
  Week 24: Vitality Score | 3.835 [2.755 to 4.914] | 7.373 [6.299 to 8.447] | 7.009 [5.929 to 8.088]
  Week 8: Social Function Score | 1.929 [0.976 to 2.882] | 3.337 [2.387 to 4.286] | 4.306 [3.352 to 5.260]
  Week 16: Social Function Score | 2.884 [1.853 to 3.915] | 5.584 [4.560 to 6.609] | 5.022 [3.989 to 6.055]
  Week 24: Social Function Score | 2.978 [1.964 to 3.992] | 5.806 [4.796 to 6.816] | 5.922 [4.909 to 6.936]
  Week 8: Role-emotional Score | 1.108 [0.095 to 2.121] | 2.459 [1.451 to 3.468] | 2.294 [1.280 to 3.307]
  Week 16: Role-emotional Score | 1.530 [0.499 to 2.562] | 4.497 [3.472 to 5.522] | 3.596 [2.563 to 4.630]
  Week 24: Role-emotional Score | 1.813 [0.793 to 2.834] | 4.382 [3.367 to 5.398] | 4.255 [3.235 to 5.275]
  Week 8: Mental Health Score | 1.081 [0.137 to 2.025] | 2.380 [1.440 to 3.320] | 3.048 [2.104 to 3.992]
  Week 16: Mental Health Score | 2.195 [1.204 to 3.185] | 4.529 [3.546 to 5.513] | 3.896 [2.905 to 4.888]
  Week 24: Mental Health Score | 2.335 [1.314 to 3.356] | 4.490 [3.474 to 5.506] | 4.767 [3.747 to 5.788]

63. Secondary Outcome: Percentage of Participants Who Achieved >=5-point Improvement From Baseline in SF-36 MCS Score Through Week 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The MCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. Higher score indicates better outcome, with an increase of 5 points considered to be clinically meaningful.
Time Frame: Week 8, 16 and 24
Population: Analysis population is FAS1. Participants who achieved >=5-point improvement from baseline in SF-36 MCS score at specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Week 8 | 26.4 | 33.1 | 27.3
  Week 16 | 31.7 | 42.3 | 31.8
  Week 24 | 30.9 | 37.5 | 34.3

64. Secondary Outcome: Percentage of Participants Who Achieved >=5-point Improvement From Baseline in SF-36 PCS Score Through Week 24
Description: SF-36 is a multi-domain instrument with 36 items to evaluate the health status and quality of life. It included 8 subscales (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health), which yielded a Physical Component Summary (PCS) with score range 0-100 (higher score-better quality of life) and a Mental Component Summary (MCS) with score range 0-100 (higher score-better quality of life) in addition to subscale scores. The PCS scores are normalized to a mean of 50 and standard deviations of 10, based upon general US population norms. Higher score indicates better outcome, with an increase of 5 points considered to be clinically meaningful.
Time Frame: Week 8, 16 and 24
Population: Analysis population is FAS1. Participants who achieved >=5-point improvement from baseline in SF-36 PCS score at specific time point and did not meet any TF criteria before, were considered as responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered as non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Week 8 | 37.8 | 45.2 | 41.2
  Week 16 | 35.8 | 59.3 | 51.0
  Week 24 | 40.2 | 60.1 | 55.9

65. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Weeks 8, 16, and 24
Description: The FACIT-Fatigue is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. The subscale consists 13-item instrument to measure fatigue. Each of the 13 items has a set of five response categories: Not at all (=0), A little bit (=1), Somewhat (=2), Quite a bit (=3) and Very much (=4). A total FACIT-Fatigue subscale score was calculated as the sum of the 13 item scores (reserved scores [4 - score]) and ranges from 0 to 52, with a higher score indicating less fatigue. Positive changes from baseline indicate improvement of fatigue. Items were reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue.
Time Frame: Baseline, Weeks 8, 16 and 24
Population: Analysis population is FAS1. Data after meeting 1 or more TF criteria were imputed as no change from baseline. Missing data were assumed MAR. The LS mean is based on MMRM model that included data from all visits for all participants included in the model.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 8 | 2.451 [1.508 to 3.395] | 5.031 [4.092 to 5.970] | 4.850 [3.905 to 5.795]
  Week 16 | 3.696 [2.675 to 4.717] | 6.977 [5.963 to 7.992] | 6.598 [5.574 to 7.622]
  Week 24 | 3.559 [2.500 to 4.619] | 7.550 [6.496 to 8.603] | 7.111 [6.051 to 8.171]

66. Secondary Outcome: Percentage of Participants Who Achieved >=4-point Improvement From Baseline in FACIT-Fatigue Score Improvement Through Week 24
Description: The FACIT-Fatigue is a questionnaire that assesses self-reported tiredness, weakness, and difficulty conducting usual activities due to fatigue. The subscale consists 13-item instrument to measure fatigue. Each of the 13 items has a set of five response categories: Not at all (=0), A little bit (=1), Somewhat (=2), Quite a bit (=3) and Very much (=4). A total FACIT-Fatigue subscale score was calculated as the sum of the 13 item scores (reserved scores [4 - score]) and ranges from 0 to 52, with a higher score indicating less fatigue. Items were reverse scored when appropriate to provide a scale in which higher scores represent better functioning or less fatigue.
Time Frame: Weeks 8, 16 and 24
Population: Analysis population is FAS1. Participants who achieved >=4-point improvement from baseline in FACIT-fatigue score at specific time point and did not meet any TF criteria before, were considered responders at that time point. Participants who met 1 or more TF criteria before or with missing data at that time point were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
percentage of participants
  Week 8 | 45.9 | 56.0 | 51.8
  Week 16 | 50.4 | 60.9 | 56.7
  Week 24 | 45.5 | 60.5 | 59.6

67. Secondary Outcome: Change From Baseline in EuroQol-5 Dimension-5 Level (EQ-5D-5L) at Weeks 16 and 24: EQ-VAS
Description: EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. The EQ VAS self-rating records the respondent's own assessment of his or her overall health status at the time of completion, on a vertical line VAS with scale of 0 (the worst health you can imagine) to 100 (the best health you can imagine). A higher score indicates better health and positive changes from baseline indicate improvement of health status
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 16 | 6.477 [4.013 to 8.941] | 17.496 [15.049 to 19.943] | 14.646 [12.179 to 17.112]
  Week 24 | 6.796 [4.298 to 9.294] | 18.371 [15.890 to 20.852] | 18.089 [15.596 to 20.581]

68. Secondary Outcome: Change From Baseline in EQ-5D-5L at Weeks 16 and 24: EQ-5D Index
Description: EQ-5D-5L is a 2-part instrument for use as a measure of health outcome, designed for self-completion by respondents. It consists of EQ-5D-5L descriptive system and EQ VAS. EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a weighted summary index (EQ-5D index), which ranges from 0 (dead) to 1.00 (full health). A higher score indicates better health and positive changes from baseline indicate improvement of health.
Time Frame: Baseline, Weeks 16 and 24
Population: as for outcome 31
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 246 | 248 | 245
units on a scale
  Week 16 | 0.058 [0.043 to 0.074] | 0.112 [0.097 to 0.127] | 0.101 [0.086 to 0.116]
  Week 24 | 0.053 [0.037 to 0.069] | 0.115 [0.099 to 0.131] | 0.116 [0.100 to 0.132]

69. Secondary Outcome: Percentage of Participants Who Achieved ACR 20 Response at Weeks 24, 28, 36, 44 and 52
Description: ACR 20 response was defined as >=20% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=20% improvement from baseline in 3 of the 5 assessments: patient's assessment of pain using VAS (0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas; range: 0-3, 0=indicating no difficulty, 3=indicating inability to perform a task in that area), and CRP.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: Full analysis set 2 (FAS2) included all randomized participants who were still on study treatment at Week 24. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 238 | 238 | 234
  Week 24 | 34.0 | 66.8 | 66.2
  Week 28: number analyzed (Participants) | 238 | 236 | 232
  Week 28 | 48.3 | 71.2 | 72.0
  Week 36: number analyzed (Participants) | 231 | 238 | 230
  Week 36 | 68.8 | 77.7 | 78.7
  Week 44: number analyzed (Participants) | 234 | 232 | 223
  Week 44 | 69.7 | 79.7 | 76.7
  Week 52: number analyzed (Participants) | 230 | 234 | 228
  Week 52 | 68.7 | 79.1 | 75.9

70. Secondary Outcome: Percentage of Participants Who Achieved ACR 50 Response at Weeks 24, 28, 36, 44 and 52
Description: ACR 50 response was defined as >=50% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=50% improvement from baseline in 3 of the 5 assessments: patient's assessment of pain using VAS (0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas; range: 0-3, 0=indicating no difficulty, 3=indicating inability to perform a task in that area), and CRP.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: Analysis population is FAS2. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 237 | 238 | 233
  Week 24 | 15.2 | 32.8 | 34.3
  Week 28: number analyzed (Participants) | 238 | 237 | 232
  Week 28 | 22.7 | 41.4 | 40.5
  Week 36: number analyzed (Participants) | 234 | 238 | 230
  Week 36 | 39.3 | 44.1 | 45.7
  Week 44: number analyzed (Participants) | 235 | 234 | 224
  Week 44 | 43.8 | 48.3 | 48.7
  Week 52: number analyzed (Participants) | 231 | 234 | 228
  Week 52 | 43.7 | 51.3 | 49.1

71. Secondary Outcome: Percentage of Participants Who Achieved ACR 70 Response at Weeks 24, 28, 36, 44 and 52
Description: ACR 70 response was defined as >=70% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=70% improvement from baseline in 3 of the 5 assessments: patient's assessment of pain using VAS (0-100 mm, 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas; range: 0-3, 0=indicating no difficulty, 3=indicating inability to perform a task in that area), and CRP.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 238 | 238 | 233
  Week 24 | 4.6 | 19.3 | 13.7
  Week 28: number analyzed (Participants) | 237 | 237 | 232
  Week 28 | 7.6 | 21.1 | 21.1
  Week 36: number analyzed (Participants) | 234 | 238 | 231
  Week 36 | 15.4 | 27.3 | 24.7
  Week 44: number analyzed (Participants) | 235 | 234 | 225
  Week 44 | 20.9 | 29.9 | 24.4
  Week 52: number analyzed (Participants) | 229 | 234 | 228
  Week 52 | 19.2 | 29.5 | 28.1

72. Secondary Outcome: ACR Components at Weeks 24, 28, 36, 44 and 52
Description: ACR components include swollen joint count (66 joints), tender joint count (68 joints), patient's assessment of pain using visual analog scale (VAS; 0-10 cm, 0=no pain and 10=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-10 cm, 0=excellent and 10= poor), physician's global assessment of disease activity (VAS; 0-10 cm, 0=no arthritis activity and 10=extremely active arthritis), patient's assessment of physical function measured by Disability Index of the Health Assessment Questionnaire (HAQ-DI; a 20-question instrument assessing 8 functional areas; range: 0-3, 0=no difficulty, 3=inability to perform a task in that area), and CRP (mg/dL).
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: Swollen Joint Count: number analyzed (Participants) | 238 | 238 | 234
  Week 24: Swollen Joint Count | 5.8 (6.99) | 3.4 (5.19) | 4.1 (5.77)
  Week 28: Swollen Joint Count: number analyzed (Participants) | 238 | 238 | 232
  Week 28: Swollen Joint Count | 4.1 (5.17) | 2.9 (4.95) | 3.2 (5.53)
  Week 36: Swollen Joint Count: number analyzed (Participants) | 233 | 238 | 230
  Week 36: Swollen Joint Count | 2.5 (3.77) | 2.4 (4.58) | 2.7 (4.67)
  Week 44: Swollen Joint Count: number analyzed (Participants) | 234 | 234 | 224
  Week 44: Swollen Joint Count | 2.1 (3.19) | 2.3 (4.42) | 2.8 (5.65)
  Week 52: Swollen Joint Count: number analyzed (Participants) | 231 | 234 | 228
  Week 52: Swollen Joint Count | 2.1 (3.59) | 2.1 (4.16) | 2.5 (4.83)
  Week 24: Tender Joint Count: number analyzed (Participants) | 238 | 238 | 234
  Week 24: Tender Joint Count | 14.4 (13.16) | 9.1 (9.94) | 10.5 (11.82)
  Week 28: Tender Joint Count: number analyzed (Participants) | 238 | 238 | 232
  Week 28: Tender Joint Count | 11.7 (11.87) | 7.9 (9.02) | 8.6 (10.03)
  Week 36: Tender Joint Count: number analyzed (Participants) | 233 | 238 | 230
  Week 36: Tender Joint Count | 8.5 (10.00) | 7.0 (8.72) | 7.5 (9.25)
  Week 44: Tender Joint Count: number analyzed (Participants) | 234 | 234 | 224
  Week 44: Tender Joint Count | 7.5 (9.42) | 6.3 (8.45) | 7.0 (9.42)
  Week 52: Tender Joint Count: number analyzed (Participants) | 231 | 234 | 228
  Week 52: Tender Joint Count | 7.4 (10.24) | 6.2 (8.18) | 7.3 (9.46)
  Week 24: Patient's Assessment of Pain: number analyzed (Participants) | 238 | 238 | 234
  Week 24: Patient's Assessment of Pain | 5.21 (2.368) | 3.77 (2.457) | 3.70 (2.193)
  Week 28: Patient's Assessment of Pain: number analyzed (Participants) | 238 | 237 | 232
  Week 28: Patient's Assessment of Pain | 4.66 (2.341) | 3.50 (2.311) | 3.45 (2.259)
  Week 36: Patient's Assessment of Pain: number analyzed (Participants) | 234 | 239 | 231
  Week 36: Patient's Assessment of Pain | 3.78 (2.297) | 3.28 (2.336) | 3.20 (2.242)
  Week 44: Patient's Assessment of Pain: number analyzed (Participants) | 235 | 233 | 225
  Week 44: Patient's Assessment of Pain | 3.67 (2.312) | 3.22 (2.370) | 3.24 (2.277)
  Week 52: Patient's Assessment of Pain: number analyzed (Participants) | 231 | 234 | 229
  Week 52: Patient's Assessment of Pain | 3.53 (2.253) | 3.10 (2.333) | 3.21 (2.371)
  Week 24: PtGA of Disease Activity: number analyzed (Participants) | 238 | 238 | 234
  Week 24: PtGA of Disease Activity | 5.29 (2.367) | 4.01 (2.516) | 3.93 (2.276)
  Week 28: PtGA of Disease Activity: number analyzed (Participants) | 238 | 237 | 232
  Week 28: PtGA of Disease Activity | 4.75 (2.338) | 3.76 (2.348) | 3.62 (2.275)
  Week 36: PtGA of Disease Activity: number analyzed (Participants) | 234 | 239 | 231
  Week 36: PtGA of Disease Activity | 3.84 (2.295) | 3.52 (2.390) | 3.30 (2.318)
  Week 44: PtGA of Disease Activity: number analyzed (Participants) | 235 | 233 | 226
  Week 44: PtGA of Disease Activity | 3.78 (2.378) | 3.36 (2.447) | 3.50 (2.323)
  Week 52: PtGA of Disease Activity: number analyzed (Participants) | 231 | 234 | 229
  Week 52: PtGA of Disease Activity | 3.68 (2.318) | 3.23 (2.383) | 3.28 (2.354)
  Week 24: PGA of Disease Activity: number analyzed (Participants) | 238 | 237 | 232
  Week 24: PGA of Disease Activity | 4.22 (2.342) | 2.74 (2.113) | 2.66 (1.906)
  Week 28: PGA of Disease Activity: number analyzed (Participants) | 236 | 236 | 231
  Week 28: PGA of Disease Activity | 3.27 (1.930) | 2.44 (1.941) | 2.33 (1.668)
  Week 36: PGA of Disease Activity: number analyzed (Participants) | 230 | 235 | 229
  Week 36: PGA of Disease Activity | 2.28 (1.594) | 2.10 (1.777) | 2.06 (1.716)
  Week 44: PGA of Disease Activity: number analyzed (Participants) | 232 | 231 | 224
  Week 44: PGA of Disease Activity | 2.06 (1.649) | 1.97 (1.842) | 1.93 (1.631)
  Week 52: PGA of Disease Activity: number analyzed (Participants) | 229 | 234 | 228
  Week 52: PGA of Disease Activity | 1.90 (1.654) | 1.77 (1.645) | 1.77 (1.616)
  Week 24: HAQ-DI score: number analyzed (Participants) | 238 | 238 | 234
  Week 24: HAQ-DI score | 1.1350 (0.61984) | 0.8766 (0.59893) | 0.8194 (0.57287)
  Week 28: HAQ-DI score: number analyzed (Participants) | 238 | 237 | 232
  Week 28: HAQ-DI score | 1.0457 (0.59051) | 0.8497 (0.61863) | 0.7985 (0.56677)
  Week 36: HAQ-DI score: number analyzed (Participants) | 234 | 239 | 231
  Week 36: HAQ-DI score | 0.9621 (0.60695) | 0.8091 (0.61588) | 0.7376 (0.56257)
  Week 44: HAQ-DI score: number analyzed (Participants) | 235 | 234 | 226
  Week 44: HAQ-DI score | 0.9117 (0.63353) | 0.7927 (0.59979) | 0.7804 (0.57721)
  Week 52: HAQ-DI score: number analyzed (Participants) | 231 | 234 | 229
  Week 52: HAQ-DI score | 0.9069 (0.63695) | 0.7917 (0.59527) | 0.7364 (0.58655)
  Week 24: CRP: number analyzed (Participants) | 236 | 238 | 234
  Week 24: CRP | 1.543 (2.1572) | 0.961 (1.2868) | 0.790 (0.8390)
  Week 28: CRP: number analyzed (Participants) | 235 | 236 | 229
  Week 28: CRP | 1.120 (1.5140) | 0.956 (1.3749) | 0.885 (1.0299)
  Week 36: CRP: number analyzed (Participants) | 231 | 237 | 231
  Week 36: CRP | 0.920 (1.4674) | 0.892 (1.3109) | 0.837 (1.0730)
  Week 44: CRP: number analyzed (Participants) | 234 | 234 | 228
  Week 44: CRP | 0.858 (1.0558) | 0.812 (1.0139) | 0.992 (1.9875)
  Week 52: CRP: number analyzed (Participants) | 228 | 234 | 229
  Week 52: CRP | 0.907 (1.5985) | 0.937 (1.2422) | 0.910 (1.2756)

73. Secondary Outcome: Change From Baseline in ACR Components at Weeks 24, 28, 36, 44 and 52
Description: as for outcome 72
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: Swollen Joint Count: number analyzed (Participants) | 238 | 238 | 234
  Week 24: Swollen Joint Count | -6.4 (7.25) | -8.2 (6.09) | -8.8 (5.50)
  Week 28: Swollen Joint Count: number analyzed (Participants) | 238 | 238 | 232
  Week 28: Swollen Joint Count | -8.1 (6.99) | -8.8 (5.98) | -9.6 (6.65)
  Week 36: Swollen Joint Count: number analyzed (Participants) | 233 | 238 | 230
  Week 36: Swollen Joint Count | -9.9 (6.47) | -9.2 (5.81) | -10.2 (6.76)
  Week 44: Swollen Joint Count: number analyzed (Participants) | 234 | 234 | 224
  Week 44: Swollen Joint Count | -10.1 (6.77) | -9.3 (6.24) | -10.2 (6.28)
  Week 52: Swollen Joint Count: number analyzed (Participants) | 231 | 234 | 228
  Week 52: Swollen Joint Count | -10.2 (6.79) | -9.6 (6.28) | -10.4 (6.17)
  Week 24: Tender Joint Count: number analyzed (Participants) | 238 | 238 | 234
  Week 24: Tender Joint Count | -7.0 (10.91) | -10.4 (9.51) | -11.9 (9.98)
  Week 28: Tender Joint Count: number analyzed (Participants) | 238 | 238 | 232
  Week 28: Tender Joint Count | -9.7 (10.78) | -11.7 (9.24) | -13.7 (10.53)
  Week 36: Tender Joint Count: number analyzed (Participants) | 233 | 238 | 230
  Week 36: Tender Joint Count | -13.2 (10.78) | -12.5 (9.68) | -14.6 (10.31)
  Week 44: Tender Joint Count: number analyzed (Participants) | 234 | 234 | 224
  Week 44: Tender Joint Count | -14.0 (11.02) | -13.3 (9.56) | -15.2 (10.25)
  Week 52: Tender Joint Count: number analyzed (Participants) | 231 | 234 | 228
  Week 52: Tender Joint Count | -14.1 (11.39) | -13.4 (10.03) | -15.0 (10.51)
  Week 24: Patient's Assessment of Pain: number analyzed (Participants) | 238 | 238 | 234
  Week 24: Patient's Assessment of Pain | -1.08 (2.441) | -2.55 (2.477) | -2.41 (2.335)
  Week 28: Patient's Assessment of Pain: number analyzed (Participants) | 238 | 237 | 232
  Week 28: Patient's Assessment of Pain | -1.63 (2.420) | -2.83 (2.519) | -2.66 (2.416)
  Week 36: Patient's Assessment of Pain: number analyzed (Participants) | 234 | 239 | 231
  Week 36: Patient's Assessment of Pain | -2.51 (2.588) | -3.02 (2.534) | -2.89 (2.540)
  Week 44: Patient's Assessment of Pain: number analyzed (Participants) | 235 | 233 | 225
  Week 44: Patient's Assessment of Pain | -2.62 (2.640) | -3.07 (2.644) | -2.87 (2.601)
  Week 52: Patient's Assessment of Pain: number analyzed (Participants) | 231 | 234 | 229
  Week 52: Patient's Assessment of Pain | -2.75 (2.659) | -3.20 (2.555) | -2.89 (2.681)
  Week 24: PtGA of Disease Activity: number analyzed (Participants) | 238 | 238 | 234
  Week 24: PtGA of Disease Activity | -1.25 (2.601) | -2.52 (2.490) | -2.40 (2.383)
  Week 28: PtGA of Disease Activity: number analyzed (Participants) | 238 | 237 | 232
  Week 28: PtGA of Disease Activity | -1.79 (2.543) | -2.79 (2.560) | -2.70 (2.382)
  Week 36: PtGA of Disease Activity: number analyzed (Participants) | 234 | 239 | 231
  Week 36: PtGA of Disease Activity | -2.70 (2.555) | -2.99 (2.569) | -3.01 (2.445)
  Week 44: PtGA of Disease Activity: number analyzed (Participants) | 235 | 233 | 226
  Week 44: PtGA of Disease Activity | -2.76 (2.741) | -3.15 (2.650) | -2.86 (2.559)
  Week 52: PtGA of Disease Activity: number analyzed (Participants) | 231 | 234 | 229
  Week 52: PtGA of Disease Activity | -2.85 (2.757) | -3.29 (2.558) | -3.06 (2.527)
  Week 24: PGA of Disease Activity: number analyzed (Participants) | 238 | 237 | 232
  Week 24: PGA of Disease Activity | -2.45 (2.248) | -3.84 (2.316) | -3.93 (2.227)
  Week 28: PGA of Disease Activity: number analyzed (Participants) | 236 | 236 | 231
  Week 28: PGA of Disease Activity | -3.42 (2.189) | -4.16 (2.175) | -4.28 (2.054)
  Week 36: PGA of Disease Activity: number analyzed (Participants) | 230 | 235 | 229
  Week 36: PGA of Disease Activity | -4.39 (2.052) | -4.49 (2.116) | -4.53 (2.173)
  Week 44: PGA of Disease Activity: number analyzed (Participants) | 232 | 231 | 224
  Week 44: PGA of Disease Activity | -4.61 (2.043) | -4.55 (2.139) | -4.70 (2.084)
  Week 52: PGA of Disease Activity: number analyzed (Participants) | 229 | 234 | 228
  Week 52: PGA of Disease Activity | -4.77 (2.007) | -4.78 (1.996) | -4.81 (2.120)
  Week 24: HAQ-DI score: number analyzed (Participants) | 237 | 238 | 234
  Week 24: HAQ-DI score | -0.1646 (0.53253) | -0.4044 (0.54194) | -0.4257 (0.50337)
  Week 28: HAQ-DI score: number analyzed (Participants) | 237 | 237 | 232
  Week 28: HAQ-DI score | -0.2547 (0.50426) | -0.4383 (0.55648) | -0.4429 (0.51556)
  Week 36: HAQ-DI score: number analyzed (Participants) | 233 | 239 | 231
  Week 36: HAQ-DI score | -0.3423 (0.52951) | -0.4702 (0.55698) | -0.5000 (0.55438)
  Week 44: HAQ-DI score: number analyzed (Participants) | 234 | 234 | 226
  Week 44: HAQ-DI score | -0.3868 (0.57065) | -0.4824 (0.57091) | -0.4652 (0.56121)
  Week 52: HAQ-DI score: number analyzed (Participants) | 230 | 234 | 229
  Week 52: HAQ-DI score | -0.3848 (0.58049) | -0.4824 (0.56167) | -0.5082 (0.58255)
  Week 24: CRP: number analyzed (Participants) | 236 | 238 | 234
  Week 24: CRP | -0.547 (2.5657) | -1.038 (2.0932) | -1.052 (2.1295)
  Week 28: CRP: number analyzed (Participants) | 235 | 236 | 229
  Week 28: CRP | -0.993 (2.3669) | -1.028 (2.0476) | -0.976 (2.1663)
  Week 36: CRP: number analyzed (Participants) | 231 | 237 | 231
  Week 36: CRP | -1.202 (2.3234) | -1.098 (2.1102) | -1.020 (2.1985)
  Week 44: CRP: number analyzed (Participants) | 234 | 234 | 228
  Week 44: CRP | -1.262 (2.5377) | -1.145 (2.1378) | -0.861 (2.8133)
  Week 52: CRP: number analyzed (Participants) | 228 | 234 | 229
  Week 52: CRP | -1.237 (2.8242) | -1.021 (2.2289) | -0.937 (2.4116)

74. Secondary Outcome: Percent Change From Baseline in ACR Components at Weeks 24, 28, 36, 44 and 52
Description: as for outcome 72
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percent change
  Week 24: Swollen Joint Count: number analyzed (Participants) | 238 | 238 | 234
  Week 24: Swollen Joint Count | -53.44 (45.655) | -72.06 (33.971) | -73.17 (30.614)
  Week 28: Swollen Joint Count: number analyzed (Participants) | 238 | 238 | 232
  Week 28: Swollen Joint Count | -66.15 (37.305) | -78.02 (30.197) | -78.85 (28.109)
  Week 36: Swollen Joint Count: number analyzed (Participants) | 233 | 238 | 230
  Week 36: Swollen Joint Count | -80.38 (28.144) | -82.82 (26.054) | -81.49 (27.338)
  Week 44: Swollen Joint Count: number analyzed (Participants) | 234 | 234 | 224
  Week 44: Swollen Joint Count | -81.85 (26.328) | -82.10 (27.742) | -83.32 (24.289)
  Week 52: Swollen Joint Count: number analyzed (Participants) | 231 | 234 | 228
  Week 52: Swollen Joint Count | -82.34 (30.494) | -83.18 (30.121) | -84.07 (24.070)
  Week 24: Tender Joint Count: number analyzed (Participants) | 238 | 238 | 234
  Week 24: Tender Joint Count | -32.53 (44.850) | -54.81 (37.134) | -57.11 (35.073)
  Week 28: Tender Joint Count: number analyzed (Participants) | 238 | 238 | 232
  Week 28: Tender Joint Count | -45.52 (41.132) | -62.48 (32.820) | -64.31 (31.767)
  Week 36: Tender Joint Count: number analyzed (Participants) | 233 | 238 | 230
  Week 36: Tender Joint Count | -62.21 (34.292) | -66.12 (32.829) | -68.50 (30.000)
  Week 44: Tender Joint Count: number analyzed (Participants) | 234 | 234 | 224
  Week 44: Tender Joint Count | -65.88 (33.344) | -70.90 (29.688) | -72.10 (27.670)
  Week 52: Tender Joint Count: number analyzed (Participants) | 231 | 234 | 228
  Week 52: Tender Joint Count | -67.29 (35.583) | -70.29 (31.985) | -69.82 (32.122)
  Week 24: Patient's Assessment of Pain: number analyzed (Participants) | 238 | 238 | 234
  Week 24: Patient's Assessment of Pain | -11.52 (48.647) | -38.44 (40.734) | -36.64 (38.086)
  Week 28: Patient's Assessment of Pain: number analyzed (Participants) | 238 | 237 | 232
  Week 28: Patient's Assessment of Pain | -22.20 (42.404) | -42.17 (41.660) | -41.02 (39.624)
  Week 36: Patient's Assessment of Pain: number analyzed (Participants) | 234 | 239 | 231
  Week 36: Patient's Assessment of Pain | -35.65 (43.207) | -45.89 (40.125) | -43.29 (44.442)
  Week 44: Patient's Assessment of Pain: number analyzed (Participants) | 235 | 233 | 225
  Week 44: Patient's Assessment of Pain | -37.45 (43.534) | -46.48 (41.725) | -43.60 (42.560)
  Week 52: Patient's Assessment of Pain: number analyzed (Participants) | 231 | 234 | 229
  Week 52: Patient's Assessment of Pain | -38.23 (47.430) | -49.00 (39.082) | -43.51 (45.742)
  Week 24: PtGA of Disease Activity: number analyzed (Participants) | 238 | 238 | 234
  Week 24: PtGA of Disease Activity | -13.78 (45.943) | -37.18 (38.628) | -33.90 (51.672)
  Week 28: PtGA of Disease Activity: number analyzed (Participants) | 238 | 237 | 232
  Week 28: PtGA of Disease Activity | -23.78 (40.895) | -39.92 (40.228) | -40.70 (36.587)
  Week 36: PtGA of Disease Activity: number analyzed (Participants) | 234 | 239 | 231
  Week 36: PtGA of Disease Activity | -38.82 (37.114) | -44.21 (36.982) | -45.52 (38.659)
  Week 44: PtGA of Disease Activity: number analyzed (Participants) | 235 | 233 | 226
  Week 44: PtGA of Disease Activity | -38.45 (43.993) | -46.64 (38.228) | -42.45 (39.243)
  Week 52: PtGA of Disease Activity: number analyzed (Participants) | 231 | 234 | 229
  Week 52: PtGA of Disease Activity | -39.34 (44.933) | -48.73 (38.925) | -45.50 (40.653)
  Week 24: PGA of Disease Activity: number analyzed (Participants) | 238 | 237 | 232
  Week 24: PGA of Disease Activity | -36.13 (33.383) | -57.60 (32.634) | -59.06 (28.137)
  Week 28: PGA of Disease Activity: number analyzed (Participants) | 236 | 236 | 231
  Week 28: PGA of Disease Activity | -49.72 (30.129) | -62.89 (28.027) | -64.14 (25.784)
  Week 36: PGA of Disease Activity: number analyzed (Participants) | 230 | 235 | 229
  Week 36: PGA of Disease Activity | -64.57 (25.695) | -67.98 (25.989) | -67.74 (28.029)
  Week 44: PGA of Disease Activity: number analyzed (Participants) | 232 | 231 | 224
  Week 44: PGA of Disease Activity | -68.32 (25.560) | -69.79 (26.949) | -70.27 (24.516)
  Week 52: PGA of Disease Activity: number analyzed (Participants) | 229 | 234 | 228
  Week 52: PGA of Disease Activity | -71.05 (25.056) | -73.09 (24.133) | -72.46 (24.485)
  Week 24: HAQ-DI score: number analyzed (Participants) | 234 | 229 | 231
  Week 24: HAQ-DI score | -6.86 (54.753) | -25.47 (63.639) | -33.72 (51.766)
  Week 28: HAQ-DI score: number analyzed (Participants) | 234 | 229 | 229
  Week 28: HAQ-DI score | -15.66 (49.522) | -28.82 (73.930) | -33.91 (59.310)
  Week 36: HAQ-DI score: number analyzed (Participants) | 230 | 230 | 228
  Week 36: HAQ-DI score | -23.34 (46.393) | -31.95 (78.348) | -37.74 (56.329)
  Week 44: HAQ-DI score: number analyzed (Participants) | 231 | 225 | 223
  Week 44: HAQ-DI score | -27.01 (49.683) | -33.84 (60.164) | -32.45 (72.337)
  Week 52: HAQ-DI score: number analyzed (Participants) | 227 | 225 | 226
  Week 52: HAQ-DI score | -26.83 (54.380) | -33.49 (63.823) | -35.02 (65.765)
  Week 24: CRP: number analyzed (Participants) | 236 | 238 | 234
  Week 24: CRP | 19.81 (150.274) | -26.90 (110.466) | -28.35 (88.038)
  Week 28: CRP: number analyzed (Participants) | 235 | 236 | 229
  Week 28: CRP | -0.80 (155.637) | -21.09 (144.287) | 15.69 (468.613)
  Week 36: CRP: number analyzed (Participants) | 231 | 237 | 231
  Week 36: CRP | -6.70 (183.299) | -25.47 (157.839) | -23.97 (104.641)
  Week 44: CRP: number analyzed (Participants) | 234 | 234 | 228
  Week 44: CRP | -8.33 (143.843) | -37.54 (76.302) | -17.44 (127.594)
  Week 52: CRP: number analyzed (Participants) | 228 | 234 | 229
  Week 52: CRP | -0.25 (208.267) | -23.15 (104.461) | -0.99 (193.429)

75. Secondary Outcome: Percentage of Participants Who Maintained an ACR 20 Response at Week 52 Among Participants Who Achieved an ACR 20 Response at Week 24
Description: as for outcome 69
Time Frame: Week 52
Population: FAS2 among participants achieved ACR20 response at Week 24. Here, N (number of participants analyzed) signifies number of participants analyzed for this OM. OM was planned to assess maintenance of guselkumab effect only through Week 52, hence data is reported for guselkumab 100mg q8w and guselkumab 100mg q4w arms only and not for placebo arm.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 156 | 151
percentage of participants | 91.7 | 86.8

76. Secondary Outcome: Percentage of Participants Who Maintained an ACR 50 Response at Week 52 Among Participants Who Achieved an ACR 50 Response at Week 24
Description: as for outcome 70
Time Frame: Week 52
Population: FAS2 among participants achieved ACR50 response at Week 24. Here, N (number of participants analyzed) signifies number of participants analyzed for this OM. The OM was planned to assess maintenance of guselkumab effect only through Week 52, hence data is reported for guselkumab 100 mg q8w and guselkumab 100 mg q4w arms only and not for placebo arm.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 78 | 77
percentage of participants | 87.2 | 79.2

77. Secondary Outcome: Percentage of Participants Who Maintained an ACR 70 Response at Week 52 Among Participants Who Achieved an ACR 70 Response at Week 24
Description: ACR 70 response was defined as >=70% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints), and >=70% improvement from baseline in 3 of the 5 assessments: patient's assessment of pain using VAS (0-100 millimeters [mm], 0=no pain and 100=worst possible pain), patient's global assessment of disease activity (arthritis, VAS; 0-100 mm, 0=excellent and 100= poor), physician's global assessment of disease activity (VAS; 0-100 mm, 0=no arthritis activity and 100=extremely active arthritis), patient's assessment of physical function measured by HAQ-DI (defined as a 20-question instrument assessing 8 functional areas; range: 0-3, 0=indicating no difficulty, 3=indicating inability to perform a task in that area), and CRP.
Time Frame: Week 52
Population: Analysis population is FAS2 among participants who achieved ACR 70 response at Week 24. The outcome measure was planned to assess the maintenance of guselkumab effect only through Week 52, hence the data in this outcome measure is reported for guselkumab 100 mg q8w and guselkumab 100 mg q4w arms only and not for placebo arm.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 46 | 32
percentage of participants | 82.6 | 75.0

78. Secondary Outcome: Change From Baseline in HAQ-DI Score at Weeks 24, 28, 36, 44 and 52
Description: as for outcome 2
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 237 | 238 | 234
  Week 24 | -0.1646 (0.53253) | -0.4044 (0.54194) | -0.4257 (0.50337)
  Week 28: number analyzed (Participants) | 237 | 237 | 232
  Week 28 | -0.2547 (0.50426) | -0.4383 (0.55648) | -0.4429 (0.51556)
  Week 36: number analyzed (Participants) | 233 | 239 | 231
  Week 36 | -0.3423 (0.52951) | -0.4702 (0.55698) | -0.5000 (0.55438)
  Week 44: number analyzed (Participants) | 234 | 234 | 226
  Week 44 | -0.3868 (0.57065) | -0.4824 (0.57091) | -0.4652 (0.56121)
  Week 52: number analyzed (Participants) | 230 | 234 | 229
  Week 52 | -0.3848 (0.58049) | -0.4824 (0.56167) | -0.5082 (0.58255)

79. Secondary Outcome: Percentage of Participants Who Achieved a Clinically Meaningful Improvement (>=0.35 Improvement From Baseline) in HAQ-DI Score at Weeks 24, 28, 36, 44 and 52 Among Participants With HAQ-DI Score >=0.35 at Baseline
Description: HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3 where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning and a decrease of 0.35 from baseline in HAQ-DI score indicates a meaningful improvement.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: Analysis population is FAS2 among participants with HAQ-DI score >=0.35 at baseline and who achieved a HAQ-DI response at Week 52. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 229 | 221 | 218
percentage of participants
  Week 24: number analyzed (Participants) | 229 | 219 | 218
  Week 24 | 34.1 | 52.5 | 58.3
  Week 28: number analyzed (Participants) | 229 | 219 | 216
  Week 28 | 42.4 | 58.4 | 63.4
  Week 36: number analyzed (Participants) | 225 | 220 | 215
  Week 36 | 48.4 | 58.2 | 61.9
  Week 44: number analyzed (Participants) | 226 | 215 | 210
  Week 44 | 50.9 | 60.0 | 61.4
  Week 52: number analyzed (Participants) | 222 | 215 | 213
  Week 52 | 50.5 | 60.9 | 62.9

80. Secondary Outcome: Percentage of Participants Who Maintained a HAQ-DI Response (>=0.35 Improvement From Baseline in HAQ-DI Score) at Week 52 Among Participants Who Achieved a HAQ-DI Response at Week 24
Description: as for outcome 79
Time Frame: Week 52
Population: Analysis population is FAS2 among participants who achieved a HAQ-DI response at Week 24. The OM was planned to assess the maintenance of guselkumab effect only through Week 52, hence the data in this outcome measure is reported for guselkumab 100 mg q8w and guselkumab 100 mg q4w arms only and not for placebo arm.
Measure: Number; unit: percentage of participants
Arm/Group | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 112 | 123
percentage of participants | 92.0 | 88.6

81. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 (CRP) Response at Weeks 24, 28, 36, 44 and 52
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. DAS28 (CRP) response criteria was defined as follows: Good response: <=3.2 at visit and >1.2 improvement; Moderate response: >3.2 at visit and >1.2 improvement or <=5.1 at visit and >0.6-1.2 improvement; No response: <=0.6 improvement, or >5.1 at visit and <=1.2 improvement. The values are 0=best to 10=worst. A DAS28 (CRP) responder was defined as achieving a good or moderate DAS28 response at a specific visit.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 236 | 238 | 234
  Week 24 | 55.5 | 79.0 | 83.8
  Week 28: number analyzed (Participants) | 235 | 233 | 227
  Week 28 | 72.3 | 85.0 | 85.9
  Week 36: number analyzed (Participants) | 230 | 236 | 228
  Week 36 | 86.5 | 86.9 | 92.5
  Week 44: number analyzed (Participants) | 233 | 232 | 221
  Week 44 | 91.0 | 91.8 | 91.9
  Week 52: number analyzed (Participants) | 228 | 234 | 227
  Week 52 | 89.0 | 89.7 | 89.4

82. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 (CRP) Remission at Weeks 24, 28, 36, 44 and 52
Description: DAS28 based on CRP is an index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. DAS28 (CRP) remission was defined as DAS28 (CRP) value <2.6 at the analysis visit.
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 236 | 238 | 234
  Week 24 | 9.3 | 25.6 | 24.4
  Week 28: number analyzed (Participants) | 235 | 233 | 227
  Week 28 | 13.2 | 27.5 | 30.4
  Week 36: number analyzed (Participants) | 230 | 236 | 228
  Week 36 | 25.7 | 36.0 | 39.5
  Week 44: number analyzed (Participants) | 233 | 232 | 221
  Week 44 | 30.0 | 38.4 | 38.0
  Week 52: number analyzed (Participants) | 228 | 234 | 227
  Week 52 | 34.2 | 39.7 | 39.6

83. Secondary Outcome: Change From Baseline in DAS28 (CRP) Score at Weeks 24, 28, 36, 44 and 52
Description: as for outcome 24
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 236 | 238 | 234
  Week 24 | -1.02 (1.101) | -1.63 (1.051) | -1.68 (0.976)
  Week 28: number analyzed (Participants) | 235 | 233 | 227
  Week 28 | -1.38 (1.099) | -1.78 (1.038) | -1.86 (1.066)
  Week 36: number analyzed (Participants) | 230 | 236 | 228
  Week 36 | -1.92 (1.086) | -1.97 (1.114) | -2.08 (1.088)
  Week 44: number analyzed (Participants) | 233 | 232 | 221
  Week 44 | -2.04 (1.098) | -2.09 (1.107) | -2.08 (1.063)
  Week 52: number analyzed (Participants) | 228 | 234 | 227
  Week 52 | -2.14 (1.142) | -2.08 (1.121) | -2.11 (1.128)

84. Secondary Outcome: Percentage of Participants Who Achieved a Response Based on Modified Psoriatic Arthritis Responder Criteria (PsARC) at Weeks 24, 28, 36, 44 and 52
Description: as for outcome 25
Time Frame: Weeks 24, 28, 36, 44 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 238 | 237 | 232
  Week 24 | 46.6 | 76.4 | 72.8
  Week 28: number analyzed (Participants) | 237 | 237 | 231
  Week 28 | 64.6 | 79.3 | 83.1
  Week 36: number analyzed (Participants) | 230 | 237 | 230
  Week 36 | 78.7 | 82.3 | 84.3
  Week 44: number analyzed (Participants) | 232 | 233 | 225
  Week 44 | 77.6 | 83.7 | 82.2
  Week 52: number analyzed (Participants) | 229 | 234 | 228
  Week 52 | 81.2 | 86.3 | 82.9

85. Secondary Outcome: Percentage of Participants With Resolution of Enthesitis at Weeks 24 and 52 Among the Participants With Enthesitis at Baseline
Description: as for outcome 26
Time Frame: Weeks 24 and 52
Population: Analysis population is FAS2 among the participants with enthesitis (LEI) at baseline. Here, n (number analyzed) signifies the number of participants evaluable for enthesitis resolution at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 152 | 165
percentage of participants
  Week 24: number analyzed (Participants) | 172 | 151 | 165
  Week 24 | 32.6 | 57.6 | 45.5
  Week 52: number analyzed (Participants) | 168 | 148 | 160
  Week 52 | 67.3 | 65.5 | 60.0

86. Secondary Outcome: Change From Baseline in Enthesitis Score (Based on LEI) at Weeks 24 and 52 Among the Participants With Enthesitis at Baseline
Description: as for outcome 28
Time Frame: Baseline, Weeks 24 and 52
Population: Analysis population is FAS2 among the participants with enthesitis (LEI) at baseline. Here n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 152 | 165
units on a scale
  Week 24: number analyzed (Participants) | 170 | 150 | 161
  Week 24 | -1.1 (1.66) | -1.6 (1.75) | -1.6 (1.63)
  Week 52: number analyzed (Participants) | 166 | 147 | 156
  Week 52 | -2.1 (1.61) | -1.9 (1.65) | -2.0 (1.78)

87. Secondary Outcome: Percentage of Participants With Resolution of Dactylitis at Weeks 24 and 52 Among Participants With Dactylitis at Baseline
Description: as for outcome 27
Time Frame: Weeks 24 and 52
Population: Analysis population is FAS2 among the participants with dactylitis at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 95 | 108 | 116
percentage of participants
  Week 24: number analyzed (Participants) | 95 | 107 | 116
  Week 24 | 41.1 | 60.7 | 68.1
  Week 52: number analyzed (Participants) | 93 | 105 | 111
  Week 52 | 78.5 | 81.9 | 81.1

88. Secondary Outcome: Change From Baseline in Dactylitis Score at Weeks 24 and 52 Among the Participants With Dactylitis at Baseline
Description: The presence and severity of dactylitis was assessed in both hands and feet using a scoring system from 0 to 3 (0-no dactylitis, 1-mild dactylitis, 2-moderate dactylitis, and 3-severe dactylitis) for each digit. The results were summed to produce a final score ranging from 0 to 60. A higher score indicates more severe dactylitis. Negative changes from baseline indicate improvement in dactylitis.
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 87
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 95 | 108 | 116
units on a scale
  Week 24: number analyzed (Participants) | 95 | 107 | 116
  Week 24 | -4.6 (7.88) | -6.1 (7.83) | -6.6 (7.84)
  Week 52: number analyzed (Participants) | 93 | 105 | 111
  Week 52 | -7.4 (9.18) | -7.3 (9.74) | -7.4 (8.59)

89. Secondary Outcome: Change From Baseline in Psoriatic Arthritis Disease Activity (PASDAS) Score at Weeks 24 and 52
Description: as for outcome 30
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 232 | 235 | 228
  Week 24 | -1.399 (1.3169) | -2.496 (1.5024) | -2.506 (1.2578)
  Week 52: number analyzed (Participants) | 223 | 232 | 223
  Week 52 | -3.041 (1.4979) | -3.197 (1.5212) | -3.161 (1.4646)

90. Secondary Outcome: Percentage of Participants With Low or Very Low Disease Activity Based on Psoriatic Arthritis Disease Activity Score (PASDAS) at Weeks 24 and 52
Description: as for outcome 30
Time Frame: Weeks 24 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 236 | 237 | 232
  Week 24 | 8.1 | 31.6 | 24.6
  Week 52: number analyzed (Participants) | 226 | 234 | 227
  Week 52 | 38.5 | 45.3 | 46.3

91. Secondary Outcome: Change From Baseline in Group of Research and Assessment of Psoriasis and Psoriatic Arthritis Composite (GRACE) Score Index at Weeks 24 and 52
Description: GRACE index is a composite PsA disease activity score converted from AMDF, which was derived from TJC (0-68) and SJC (0-66), HAQ-DI (0-3), patient's global assessment of disease activity on arthritis and psoriasis (0-100 mm, 0=excellent and 100= poor), patient's assessment of skin disease activity (0-100 mm, 0=excellent and 100=poor), patient's global assessment of disease activity on arthritis (0-100 mm, 0=excellent and 100=poor), PASI (0-72), and PsA Quality of Life Index (derived as PsAQOL =25.355 + [2.367*HAQ-DI] - [0.234*SF-PCS] - [0.244*SF-MCS]), where HAQ-DI: HAQ-DI score (0-3, 0=least difficulty and 3=extreme difficulty), SF-PCS (Score ranges from 0 to 100, higher scores= better quality of life) and SF-MCS (score ranges from 0 to 100, higher scores= better quality of life). The total score is from 0-10, where lower score indicates better response. Higher score indicates more active disease activity. Negative change from baseline indicates improvement of PsA disease activity.
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 237 | 237 | 232
  Week 24 | -1.260 (1.4909) | -2.658 (1.6770) | -2.672 (1.4589)
  Week 52: number analyzed (Participants) | 228 | 234 | 228
  Week 52 | -3.085 (1.6277) | -3.271 (1.6453) | -3.267 (1.5646)

92. Secondary Outcome: Percentage of Participants With Low Disease Activity Based on Group of Research and Assessment of Psoriasis and Psoriatic Arthritis Composite (GRACE) Score Index at Weeks 24 and 52
Description: GRACE index is a composite PsA disease activity score converted from Arithmetic Mean of Desirability Function (AMDF), derived from TJC (0-68) and SJC (0-66), HAQ-DI (0-3), PtGA of disease activity on arthritis and psoriasis (0-100 mm, 0=excellent and 100=poor), patient's assessment of skin disease activity (0-100 mm, 0=excellent and 100=poor), PtGA of disease activity on arthritis (0-100 mm, 0=excellent and 100=poor), PASI (0-72), and PsA Quality of Life Index (derived as PsAQOL=25.355 + [2.367*HAQ-DI]-[0.234*SF-PCS]-[0.244*SF-MCS]), where HAQ-DI: HAQ-DI score (0-3, 0=least difficulty and 3=extreme difficulty), SF-PCS (Score range= 0-100, higher scores= better quality of life) and SF-MCS (score range=0-100, higher scores= better quality of life). Total score is 0-10, lower score=better response. Higher score= more active disease activity. Negative change from baseline indicates improvement of PsA disease activity. GRACE low disease activity is GRACE score <=2.3 at the analysis visit.
Time Frame: Weeks 24 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 238 | 237 | 232
  Week 24 | 7.6 | 29.5 | 27.6
  Week 52: number analyzed (Participants) | 229 | 234 | 228
  Week 52 | 34.9 | 43.2 | 43.0

93. Secondary Outcome: Change From Baseline in the Disease Activity Index for Psoriatic Arthritis (DAPSA) Score at Weeks 24, 28, 36, 44 and 52
Description: DAPSA assessed the joint domain of PsA and was derived from the sum of the following components: tender joint count (0-68), swollen joint count (0-66), CRP level (mg/dL), patient assessment of pain (0-10cm VAS, 0=no pain, 10=worst possible pain), and patient's global assessment of disease activity on arthritis (0 to 10cm VAS, 0=excellent and 10=poor). A higher score indicates more active disease activity. Negative changes from baseline indicate improvement of PsA disease activity. The assessment does not have a score range with an upper or lower bound.
Time Frame: Baseline, Weeks 24, 28, 36, 44 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 236 | 238 | 234
  Week 24 | -16.377 (19.1814) | -24.718 (16.7967) | -26.578 (15.3393)
  Week 28: number analyzed (Participants) | 235 | 233 | 227
  Week 28 | -22.199 (17.9394) | -26.573 (15.5254) | -29.613 (17.6129)
  Week 36: number analyzed (Participants) | 230 | 236 | 228
  Week 36 | -29.251 (18.1137) | -28.889 (16.4372) | -31.782 (16.7698)
  Week 44: number analyzed (Participants) | 233 | 232 | 221
  Week 44 | -30.754 (18.5016) | -30.108 (16.6013) | -32.126 (15.7605)
  Week 52: number analyzed (Participants) | 228 | 234 | 227
  Week 52 | -31.209 (18.9981) | -30.512 (17.5074) | -32.282 (16.6320)

94. Secondary Outcome: Change From Baseline in Modified Composite Psoriatic Disease Activity Index (mCPDAI) Score at Weeks 24 and 52
Description: as for outcome 36
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 234 | 235 | 228
  Week 24 | -1.34 (2.144) | -2.97 (2.382) | -3.32 (2.098)
  Week 52: number analyzed (Participants) | 226 | 232 | 224
  Week 52 | -3.75 (2.391) | -3.84 (2.449) | -4.10 (2.387)

95. Secondary Outcome: Percentage of Participants With Low Disease Activity Based on Modified Composite Psoriatic Disease Activity Index (mCPDAI) Score at Weeks 24 and 52
Description: The mCPDAI assessed 4 domains (joints, skin, entheses, and dactylitis). The mCPDAI scores were calculated using the following assessments: joints (66 swollen and 68 tender joint counts), HAQ-DI score, PASI, dactylitis, and enthesitis. Within each domain a score (range 0-3) was assigned, where 0= Not involved, 1= Mild, 2= Moderate and 3= Severe. The scores for each domain were then added together to give a final score range of 0 to 12. A higher score indicates more active disease activity. Negative changes from baseline indicate improvement of PsA disease activity. mCPDAI low disease activity is defined as mCPDAI score <=3.2 at the analysis visit.
Time Frame: Weeks 24 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 238 | 237 | 232
  Week 24 | 15.1 | 48.9 | 43.5
  Week 52: number analyzed (Participants) | 229 | 234 | 228
  Week 52 | 56.3 | 61.1 | 60.1

96. Secondary Outcome: Percentage of Participants Who Achieved Minimal Disease Activity (MDA) at Weeks 24 and 52
Description: as for outcome 38
Time Frame: Weeks 24 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 238 | 238 | 234
  Week 24 | 6.3 | 26.5 | 19.7
  Week 52: number analyzed (Participants) | 231 | 234 | 228
  Week 52 | 31.6 | 32.9 | 36.8

97. Secondary Outcome: Percentage of Participants With Very Low Disease Activity (VLDA) at Weeks 24 and 52
Description: A measurement that defines a satisfactory state of disease activity that includes the 5 domains of PsA (joint symptoms, skin psoriasis, patient's perspective of pain and disease activity, physical function, and enthesitis). A participant was considered as having achieved VLDA at a visit if the participant fulfilled all 7 criteria (tender joint count <=1; swollen joint count <=1; PASI <=1; patient pain VAS score of <=15; patient global disease activity VAS [arthritis and psoriasis] score of <=20; Health Assessment Questionnaire (HAQ) score <=0.5; and tender entheseal points <=1) at that visit.
Time Frame: Weeks 24 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 238 | 237 | 234
  Week 24 | 1.3 | 4.6 | 5.1
  Week 52: number analyzed (Participants) | 231 | 234 | 229
  Week 52 | 6.9 | 17.1 | 12.2

98. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Score at Weeks 24 and 52 Among Participants With Spondylitis and Peripheral Arthritis at Baseline
Description: as for outcome 39
Time Frame: Baseline, Weeks 24 and 52
Population: Analysis population is FAS2 among the participants with spondylitis and peripheral arthritis and BASDAI score >0 at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 91 | 66 | 79
units on a scale
  Week 24: number analyzed (Participants) | 91 | 64 | 78
  Week 24 | -1.374 (2.4269) | -2.652 (2.3825) | -2.674 (1.9941)
  Week 52: number analyzed (Participants) | 88 | 64 | 79
  Week 52 | -2.986 (2.4945) | -2.883 (2.5193) | -3.084 (2.1843)

99. Secondary Outcome: Percentage of Participants Who Achieved >= 20%, >=50%, >=70%, and >=90% Improvement From Baseline in BASDAI Score at Weeks 24 and 52 Among the Participants With Spondylitis and Peripheral Arthritis and BASDAI Score >0 at Baseline
Description: as for outcome 39
Time Frame: Weeks 24 and 52
Population: as for outcome 98
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 91 | 66 | 79
percentage of participants
  Week 24: Participants with >=20% Improvement: number analyzed (Participants) | 91 | 64 | 78
  Week 24: Participants with >=20% Improvement | 44.0 | 62.5 | 73.1
  Week 52: Participants with >=20% Improvement: number analyzed (Participants) | 88 | 64 | 79
  Week 52: Participants with >=20% Improvement | 71.6 | 70.3 | 79.7
  Week 24: Participants with >=50% Improvement: number analyzed (Participants) | 91 | 64 | 78
  Week 24: Participants with >=50% Improvement | 22.0 | 40.6 | 39.7
  Week 52: Participants with >=50% Improvement: number analyzed (Participants) | 88 | 64 | 79
  Week 52: Participants with >=50% Improvement | 50.0 | 42.2 | 50.6
  Week 24: Participants with >=70% Improvement: number analyzed (Participants) | 91 | 64 | 78
  Week 24: Participants with >=70% Improvement | 8.8 | 21.9 | 16.7
  Week 52: Participants with >=70% Improvement: number analyzed (Participants) | 88 | 64 | 79
  Week 52: Participants with >=70% Improvement | 23.9 | 26.6 | 30.4
  Week 24: Participants with >=90% Improvement: number analyzed (Participants) | 91 | 64 | 78
  Week 24: Participants with >=90% Improvement | 2.2 | 1.6 | 3.8
  Week 52: Participants with >=90% Improvement: number analyzed (Participants) | 88 | 64 | 79
  Week 52: Participants with >=90% Improvement | 6.8 | 10.9 | 8.9

100. Secondary Outcome: Change From Baseline in PASI Score at Weeks 24 and 52 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 44
Time Frame: Baseline, Weeks 24 and 52
Population: Analysis population is FAS2 among the participants who had >=3% BSA of psoriatic involvement and an IGA score >=2 (mild) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 176 | 173 | 177
units on a scale
  Week 24: number analyzed (Participants) | 176 | 172 | 176
  Week 24 | -2.989 (6.1515) | -11.685 (12.3496) | -12.574 (11.8391)
  Week 52: number analyzed (Participants) | 172 | 170 | 173
  Week 52 | -11.016 (9.9801) | -11.977 (12.0847) | -12.857 (11.3052)

101. Secondary Outcome: Percentage of Participants Who Achieved PASI 50 Response at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severity. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. PASI 50 response: >=50% improvement in PASI score from baseline.
Time Frame: Weeks 24 and 52
Population: as for outcome 100
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 176 | 173 | 177
percentage of participants
  Week 24: number analyzed (Participants) | 176 | 172 | 176
  Week 24 | 39.8 | 94.8 | 93.8
  Week 52: number analyzed (Participants) | 172 | 170 | 173
  Week 52 | 95.9 | 97.1 | 98.3

102. Secondary Outcome: Percentage of Participants Who Achieved PASI 75 Response at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severity. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. PASI 75 response: >=75% improvement in PASI score from baseline.
Time Frame: Weeks 24 and 52
Population: as for outcome 100
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 176 | 173 | 177
percentage of participants
  Week 24: number analyzed (Participants) | 176 | 172 | 176
  Week 24 | 23.3 | 80.8 | 81.8
  Week 52: number analyzed (Participants) | 172 | 170 | 173
  Week 52 | 88.4 | 88.8 | 91.9

103. Secondary Outcome: Percentage of Participants Who Achieved PASI 90 Response at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severity. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. PASI 90 response: >=90% improvement in PASI score from baseline.
Time Frame: Weeks 24 and 52
Population: as for outcome 100
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 176 | 173 | 177
percentage of participants
  Week 24: number analyzed (Participants) | 176 | 172 | 176
  Week 24 | 10.2 | 70.3 | 63.6
  Week 52: number analyzed (Participants) | 172 | 170 | 173
  Week 52 | 76.7 | 77.1 | 81.5

104. Secondary Outcome: Percentage of Participants Who Achieved PASI 100 Response at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: PASI is a tool to assess and grade severity of psoriasis and response to therapy. In PASI, body is divided into 4 areas: head, trunk, upper extremities, lower extremities. Each area was assessed separately for percentage of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4 that is none to maximum severity. PASI numeric score range from 0 (no psoriasis) to 72. Higher scores indicate more severe disease. PASI 100 response: 100% improvement in PASI score from baseline.
Time Frame: Weeks 24 and 52
Population: as for outcome 100
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 176 | 173 | 177
percentage of participants
  Week 24: number analyzed (Participants) | 176 | 172 | 176
  Week 24 | 2.8 | 46.5 | 46.6
  Week 52: number analyzed (Participants) | 172 | 170 | 173
  Week 52 | 55.2 | 54.7 | 61.3

105. Secondary Outcome: Percentage of Participants Who Achieved Both PASI 75 and ACR 20 Responses at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: In PASI, each area (head, trunk, upper and lower extremities) was assessed for % of area involved and translated to numeric score from 0 (no involvement) to 6 (90-100% involvement) and for erythema, induration, and scaling, each rated on scale of 0 to 4. PASI produces numeric score from 0 to 72. Higher scores=more severe disease. PASI 75: >=75% improvement in PASI score from baseline. ACR 20: >=20% improvement in SJC (66 joints)+TJC (68 joints) and >=20% improvement in 3 of 5: patient's assessment of pain (VAS; 0-100 mm, 0=no pain to 100=worst possible pain), PtGA of disease activity (VAS; 0-100 mm, 0=excellent to 100=poor), PGA of disease activity (VAS; 0-100 mm, 0=no arthritis to 100=extremely active arthritis), patient's assessment of physical function (HAQ-DI -20-question instrument; range- 0=no difficulty to 3=inability to perform task) and CRP.
Time Frame: Weeks 24 and 52
Population: as for outcome 100
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 176 | 173 | 177
percentage of participants
  Week 24: number analyzed (Participants) | 176 | 172 | 176
  Week 24 | 11.4 | 58.1 | 59.7
  Week 52: number analyzed (Participants) | 171 | 170 | 173
  Week 52 | 59.6 | 73.5 | 69.9

106. Secondary Outcome: Percentage of Participants Who Achieved Both PASI 75 and Modified PsARC Response at Weeks 24 and 52 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: In PASI, each area (head, trunk, upper and lower extremities) was assessed separately for % of area involved and translated to numeric score ranging from 0 (no involvement) to 6 (90-100% involvement), and for erythema, induration, and scaling, each rated on scale of 0 to 4. PASI produces numeric score range from 0 to 72. Higher scores=more severe disease. PASI75 response: >=75% improvement in PASI score from baseline. Modified PsARC response: improvement in at least 2 of 4 criteria: >=30% decrease in SJC and TJC, >=20% improvement in PtGA of Disease Activity (arthritis) on VAS (0-100 mm, 0=excellent and 100=poor), >=20% improvement in PGA of Disease Activity on VAS (VAS: 0-100 mm, 0=no arthritis and 100=extremely active arthritis), and at least 1 of 2 joint criteria with no deterioration in other criteria.
Time Frame: Weeks 24 and 52
Population: as for outcome 100
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 176 | 173 | 177
percentage of participants
  Week 24: number analyzed (Participants) | 176 | 172 | 176
  Week 24 | 15.3 | 66.9 | 63.6
  Week 52: number analyzed (Participants) | 172 | 170 | 173
  Week 52 | 70.9 | 79.4 | 76.3

107. Secondary Outcome: Percentage of Participants Who Achieved an IGA Response at Weeks 24 and 52 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: A psoriasis IGA response was defined as an IGA score of 0 (cleared) or 1 (minimal) and >= 2 grade reduction from baseline in the IGA psoriasis score. The IGA documents the investigator's assessment of the patient's psoriasis and lesions are graded for induration, erythema and scaling, each using a 5 point scale: 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe). The IGA score of psoriasis was based upon the average of induration, erythema and scaling scores. The participant's psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Time Frame: Weeks 24 and 52
Population: Analysis population is FAS2 among the participants who had >=3% BSA of psoriatic involvement and an IGA score >=2 (mild) at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 176 | 173 | 177
percentage of participants
  Week 24: number analyzed (Participants) | 176 | 172 | 176
  Week 24 | 19.9 | 72.1 | 71.0
  Week 52: number analyzed (Participants) | 172 | 170 | 173
  Week 52 | 84.3 | 77.1 | 84.4

108. Secondary Outcome: Percentage of Participants Who Achieved an IGA Score of 0 (Cleared) at Weeks 24 and 52 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 107
Time Frame: Weeks 24 and 52
Population: as for outcome 107
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 176 | 173 | 177
percentage of participants
  Week 24: number analyzed (Participants) | 176 | 172 | 176
  Week 24 | 8.0 | 51.2 | 52.8
  Week 52: number analyzed (Participants) | 172 | 170 | 173
  Week 52 | 66.9 | 60.0 | 66.5

109. Secondary Outcome: Percentage of Participants Who Achieved a DLQI Score of 0 or 1 at Weeks 24 and 52 Among the Participants With DLQI Score >1, With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 45
Time Frame: Weeks 24 and 52
Population: Analysis population is FAS2 among the participants with DLQI Score >1, with >=3% BSA psoriatic involvement and an IGA score of >=2 (mild) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 165 | 155 | 166
percentage of participants
  Week 24: number analyzed (Participants) | 165 | 154 | 166
  Week 24 | 12.1 | 65.6 | 61.4
  Week 52: number analyzed (Participants) | 162 | 153 | 163
  Week 52 | 56.8 | 68.6 | 68.7

110. Secondary Outcome: Percentage of Participants Who Achieved >=5-point Improvement From Baseline in DLQI Score at Weeks 24 and 52 Among the Participants With DLQI Score >=5, >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 46
Time Frame: Weeks 24 and 52
Population: Analysis population is FAS2 among the participants with DLQI score >=5, >=3% BSA psoriatic involvement and an IGA score of >=2 (mild) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 140 | 131 | 145
percentage of participants
  Week 24: number analyzed (Participants) | 140 | 130 | 145
  Week 24 | 40.7 | 85.4 | 90.3
  Week 52: number analyzed (Participants) | 138 | 129 | 142
  Week 52 | 84.8 | 92.2 | 89.4

111. Secondary Outcome: Change From Baseline in DLQI Score at Weeks 24 and 52 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 47
Time Frame: Baseline, Weeks 24 and 52
Population: Analysis population is FAS2 among the participants with >=3% BSA psoriatic involvement and an IGA Score of >=2 (mild) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 176 | 173 | 177
units on a scale
  Week 24: number analyzed (Participants) | 176 | 172 | 177
  Week 24 | -2.142 (6.4593) | -8.901 (7.3657) | -9.249 (7.0988)
  Week 52: number analyzed (Participants) | 173 | 170 | 174
  Week 52 | -8.815 (7.2714) | -9.235 (7.3840) | -9.839 (6.8777)

112. Secondary Outcome: Change From Baseline in Modified vdH-S Score at Week 52
Description: as for outcome 6
Time Frame: Baseline and Week 52
Population: FAS2 for structural damage (FAS2-SD) among all randomized participants who were continuing study treatment at Week 24. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 230 | 235 | 229
units on a scale | 1.25 (3.508) | 0.97 (3.623) | 1.07 (3.843)

113. Secondary Outcome: Change in Total Modified vdH-S Score From Week 24 to Week 52
Description: Modified vdH-S score is the sum of the erosion score (hand, feet) and joint space narrowing (JSN) score (hand, feet). Joint erosion score is the summary of erosion severity in 40 joints of hand scored according to the surface area, from 0 (no erosion) to 5 (complete collapse of bone) and 12 joints of 2 feet (each side of the foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum erosion score of 320. JSN score is the total JSN score in same 52 joints as above, each joint scored according to the subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum JSN score of 208. Total score ranges from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score indicates more joint damage.
Time Frame: From Week 24 to Week 52
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 230 | 235 | 229
units on a scale | 0.25 (1.635) | 0.23 (1.808) | 0.62 (2.530)

114. Secondary Outcome: Change From Baseline in Modified vdH-S Erosion Score at Week 52
Description: as for outcome 6
Time Frame: Baseline and Week 52
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 230 | 235 | 229
units on a scale | 0.92 (2.497) | 0.67 (2.707) | 0.70 (2.631)

115. Secondary Outcome: Change in Modified vdH-S Erosion Score From Week 24 to Week 52
Description: as for outcome 113
Time Frame: From Week 24 to Week 52
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 230 | 235 | 229
units on a scale | 0.17 (1.277) | 0.10 (1.422) | 0.39 (1.725)

116. Secondary Outcome: Change From Baseline in Modified vdH-S JSN Score at Week 52
Description: as for outcome 6
Time Frame: Baseline and Week 52
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 230 | 235 | 229
units on a scale | 0.33 (1.356) | 0.29 (1.272) | 0.38 (1.633)

117. Secondary Outcome: Change in Modified vdH-S JSN Score From Week 24 to Week 52
Description: as for outcome 113
Time Frame: From Week 24 to Week 52
Population: as for outcome 112
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 230 | 235 | 229
units on a scale | 0.07 (0.635) | 0.13 (0.705) | 0.23 (1.088)

118. Secondary Outcome: Change From Baseline in Modified vdH-S Score by Region and Type of Damage (ie, Hand Erosion, Hand JSN, Foot Erosion, Foot JSN Subscores) at Week 52
Description: as for outcome 52
Time Frame: Baseline and Week 52
Population: FAS2 for structural damage (FAS2-SD) among all randomized participants who were continuing study treatment at Week 24. Here, 'n' (number analyzed) signifies the number of participants analyzed for a specified score.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Hand Erosion Score: number analyzed (Participants) | 230 | 235 | 229
  Hand Erosion Score | 0.66 (1.815) | 0.37 (1.969) | 0.35 (1.830)
  Hand JSN Score: number analyzed (Participants) | 230 | 235 | 229
  Hand JSN Score | 0.29 (1.181) | 0.19 (0.913) | 0.22 (1.235)
  Hand Score: number analyzed (Participants) | 230 | 235 | 229
  Hand Score | 0.95 (2.706) | 0.56 (2.589) | 0.57 (2.759)
  Foot Erosion Score: number analyzed (Participants) | 230 | 235 | 229
  Foot Erosion Score | 0.26 (1.014) | 0.30 (1.339) | 0.34 (1.413)
  Foot JSN Score: number analyzed (Participants) | 230 | 235 | 229
  Foot JSN Score | 0.04 (0.353) | 0.10 (0.660) | 0.16 (0.864)
  Foot Score: number analyzed (Participants) | 230 | 235 | 229
  Foot Score | 0.30 (1.220) | 0.40 (1.687) | 0.50 (1.939)

119. Secondary Outcome: Percentage of Participants With a Change of <=0 or <=0.5 From Baseline in Modified vdH-S Score at Week 52
Description: as for outcome 6
Time Frame: Week 52
Population: FAS2 for structural damage (FAS2-SD) among all randomized participants who were continuing study treatment at Week 24. Here, n (number analyzed) signifies the number of participants analyzed at specified category.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Change of <=0 from Baseline: number analyzed (Participants) | 230 | 235 | 229
  Change of <=0 from Baseline | 57.4 | 55.7 | 56.8
  Change of <=0.5 from Baseline: number analyzed (Participants) | 230 | 235 | 229
  Change of <=0.5 from Baseline | 67.4 | 67.2 | 72.1

120. Secondary Outcome: Percentage of Participants With a Change of <=0 or <=0.5 From Baseline in Modified vdH-S Erosion Score at Week 52
Description: as for outcome 6
Time Frame: Week 52
Population: as for outcome 119
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Change of <=0 from Baseline: number analyzed (Participants) | 230 | 235 | 229
  Change of <=0 from Baseline | 58.3 | 59.6 | 60.3
  Change of <=0.5 from Baseline: number analyzed (Participants) | 230 | 235 | 229
  Change of <=0.5 from Baseline | 70.4 | 71.1 | 72.1

121. Secondary Outcome: Percentage of Participants With a Change of <=0 or <=0.5 From Baseline in Modified vdH-S JSN Score at Week 52
Description: as for outcome 6
Time Frame: Week 52
Population: as for outcome 119
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Change of <=0 from Baseline: number analyzed (Participants) | 230 | 235 | 229
  Change of <=0 from Baseline | 78.7 | 75.3 | 79.5
  Change of <=0.5 from Baseline: number analyzed (Participants) | 230 | 235 | 229
  Change of <=0.5 from Baseline | 88.3 | 86.0 | 86.5

122. Secondary Outcome: Percentage of Participants Without Radiographic Progression Based on the (SDC) From Baseline at Week 52
Description: Modified vdH-S score is the sum of the erosion score (hand, feet) and JSN score (hand, feet). Joint erosion score is the summary of erosion severity in 40 joints of hand scored according to the surface area, from 0 (no erosion) to 5 (complete collapse of bone) and 12 joints of 2 feet (each side of foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum erosion score of 320. JSN score is the total JSN score in same 52 joints as above, each joint scored according to the subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum JSN score of 208. Total score ranges from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score indicates more joint damage. SDC was defined as the cut-off above which the changes can be detected beyond measurement error. Without radiographic progression was defined as change from baseline in the modified vdH-S score <=SDC of 2.39.
Time Frame: Week 52
Population: as for outcome 112
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 230 | 235 | 229
percentage of participants | 80.4 | 82.6 | 85.2

123. Secondary Outcome: Percentage of Participants Without Radiographic Joint Erosion Progression Based on (SDC) From Baseline at Week 52
Description: Modified vdH-S score is sum of the erosion score (hand, feet) and JSN score (hand, feet). Joint erosion score is summary of erosion severity in 40 joints of hand scored according to surface area, from 0 (no erosion) to 5 (complete collapse of bone) and 12 joints of 2 feet (each side of foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum erosion score of 320. JSN score is total JSN score in same 52 joints as above, each joint scored according to subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum JSN score of 208. Total score ranges from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score indicates more joint damage. SDC was defined as the cut-off above which the changes can be detected beyond measurement error. Without radiographic joint erosion progression was defined as change from baseline in modified vdH-S erosion score <=SDC of 2.22.
Time Frame: Week 52
Population: as for outcome 112
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 230 | 235 | 229
percentage of participants | 82.2 | 84.3 | 87.3

124. Secondary Outcome: Percentage of Participants Without Radiographic JSN Progression Based on (SDC) From Baseline at Week 52
Description: Modified vdH-S score is sum of erosion score (hand, feet) and JSN score (hand, feet). Joint erosion score is summary of erosion severity in 40 joints of hand scored according to surface area, from 0 (no erosion) to 5 (complete collapse of bone) and 12 joints of 2 feet (each side of foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum erosion score of 320. JSN score is total JSN score in same 52 joints as above, each joint scored according to subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum JSN score of 208. Total score ranges from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score indicates more joint damage. SDC was defined as cut-off above which changes can be detected beyond measurement error. Without radiographic JSN progression was defined as change from baseline in modified vdH-S JSN score <=SDC of 1.02.
Time Frame: Week 52
Population: as for outcome 112
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 230 | 235 | 229
percentage of participants | 91.3 | 91.5 | 90.4

125. Secondary Outcome: Percentage of Participants With Pencil in Cup or Gross Osteolysis Deformities at Baseline and Week 52
Description: Percentage of Participants with Pencil in cup or Gross Osteolysis Deformities were reported. Pencil in Cup or Gross Osteolytis Deformities are radiographic features specific for psoriatic arthritis.
Time Frame: Baseline and Week 52
Population: FAS2 for structural damage (FAS2-SD) among all randomized participants who were continuing study treatment at Week 24. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Baseline: number analyzed (Participants) | 231 | 238 | 232
  Baseline | 6.9 | 4.6 | 6.9
  Week 52: number analyzed (Participants) | 230 | 235 | 229
  Week 52 | 7.8 | 5.1 | 7.0

126. Secondary Outcome: Change From Baseline in SF-36 PCS Score at Weeks 24 and 52
Description: as for outcome 11
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 237 | 238 | 234
  Week 24 | 3.782 (7.1776) | 7.838 (8.0335) | 7.183 (6.9793)
  Week 52: number analyzed (Participants) | 230 | 234 | 229
  Week 52 | 8.124 (8.2192) | 9.511 (8.3176) | 8.960 (8.5891)

127. Secondary Outcome: Change From Baseline in SF-36 MCS Score at Weeks 24 and 52
Description: as for outcome 13
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 237 | 238 | 234
  Week 24 | 2.211 (10.1368) | 4.452 (9.9560) | 4.128 (9.1814)
  Week 52: number analyzed (Participants) | 230 | 234 | 229
  Week 52 | 4.297 (10.8960) | 4.465 (9.7780) | 4.076 (9.1101)

128. Secondary Outcome: Change From Baseline in Norm Based Scores of SF-36 Scales at Weeks 24 and 52
Description: as for outcome 62
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: Physical Function Score: number analyzed (Participants) | 237 | 238 | 234
  Week 24: Physical Function Score | 3.602 (7.7388) | 7.052 (8.5020) | 6.772 (7.5920)
  Week 52: Physical Function Score: number analyzed (Participants) | 230 | 234 | 229
  Week 52: Physical Function Score | 7.722 (8.9480) | 8.489 (8.8599) | 8.374 (8.7884)
  Week 24: Role-physical Score: number analyzed (Participants) | 237 | 238 | 234
  Week 24: Role-physical Score | 3.695 (7.5950) | 6.897 (7.7240) | 6.381 (7.2203)
  Week 52: Role-physical Score: number analyzed (Participants) | 230 | 234 | 229
  Week 52: Role-physical Score | 6.560 (8.5399) | 7.677 (8.2995) | 7.344 (7.7145)
  Week 24: Bodily Pain Score: number analyzed (Participants) | 237 | 238 | 234
  Week 24: Bodily Pain Score | 3.882 (8.3009) | 8.333 (8.3852) | 7.833 (7.3390)
  Week 52: Bodily Pain Score: number analyzed (Participants) | 230 | 234 | 229
  Week 52: Bodily Pain Score | 8.460 (8.4659) | 10.238 (8.7185) | 9.457 (9.7977)
  Week 24: General Health Score: number analyzed (Participants) | 237 | 238 | 234
  Week 24: General Health Score | 2.255 (7.2176) | 5.963 (7.8794) | 5.067 (7.4182)
  Week 52: General Health Score: number analyzed (Participants) | 230 | 234 | 229
  Week 52: General Health Score | 6.396 (8.5589) | 7.173 (7.2703) | 6.366 (8.4199)
  Week 24: Vitality Score: number analyzed (Participants) | 237 | 238 | 234
  Week 24: Vitality Score | 4.224 (9.0878) | 7.914 (9.4638) | 6.970 (9.4889)
  Week 52: Vitality Score: number analyzed (Participants) | 230 | 234 | 229
  Week 52: Vitality Score | 7.879 (9.4160) | 8.646 (9.5131) | 7.654 (9.3905)
  Week 24: Social Function Score: number analyzed (Participants) | 237 | 238 | 234
  Week 24: Social Function Score | 3.088 (10.4330) | 6.551 (9.7076) | 5.892 (8.5510)
  Week 52: Social Function Score: number analyzed (Participants) | 230 | 234 | 229
  Week 52: Social Function Score | 6.278 (10.9444) | 7.199 (10.1315) | 6.787 (9.5326)
  Week 24: Role-emotional Score: number analyzed (Participants) | 237 | 238 | 234
  Week 24: Role-emotional Score | 1.910 (10.0772) | 4.535 (10.1304) | 4.107 (8.9473)
  Week 52: Role-emotional Score: number analyzed (Participants) | 230 | 234 | 229
  Week 52: Role-emotional Score | 4.057 (10.8795) | 4.970 (10.1685) | 4.607 (8.7627)
  Week 24: Mental Health Score: number analyzed (Participants) | 237 | 238 | 234
  Week 24: Mental Health Score | 2.583 (9.2222) | 4.605 (9.7905) | 4.752 (8.9336)
  Week 52: Mental Health Score: number analyzed (Participants) | 230 | 234 | 229
  Week 52: Mental Health Score | 5.153 (10.0724) | 4.829 (9.3665) | 4.741 (9.3825)

129. Secondary Outcome: Percentage of Participants Who Achieved >=5-point Improvement From Baseline in SF-36 PCS Score at Weeks 24 and 52
Description: as for outcome 64
Time Frame: Weeks 24 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 237 | 238 | 234
  Week 24 | 42.2 | 63.4 | 58.5
  Week 52: number analyzed (Participants) | 230 | 234 | 229
  Week 52 | 63.0 | 67.1 | 65.5

130. Secondary Outcome: Percentage of Participants Who Achieved >=5-point Improvement From Baseline in SF-36 MCS Score at Weeks 24 and 52
Description: as for outcome 63
Time Frame: Weeks 24 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 237 | 238 | 234
  Week 24 | 32.5 | 40.3 | 36.8
  Week 52: number analyzed (Participants) | 230 | 234 | 229
  Week 52 | 41.7 | 44.9 | 38.9

131. Secondary Outcome: Change From Baseline in FACIT-Fatigue Score at Weeks 24 and 52
Description: as for outcome 65
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 237 | 238 | 234
  Week 24 | 3.844 (9.0440) | 8.034 (9.8888) | 6.970 (8.6274)
  Week 52: number analyzed (Participants) | 230 | 234 | 229
  Week 52 | 7.548 (9.3745) | 8.927 (9.4646) | 7.686 (9.0833)

132. Secondary Outcome: Percentage of Participants Who Achieved >=4-point Improvement From Baseline in FACIT-Fatigue Score Improvement at Weeks 24 and 52
Description: as for outcome 66
Time Frame: Weeks 24 and 52
Population: as for outcome 70
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
percentage of participants
  Week 24: number analyzed (Participants) | 237 | 238 | 234
  Week 24 | 49.4 | 63.9 | 62.8
  Week 52: number analyzed (Participants) | 230 | 234 | 229
  Week 52 | 68.3 | 69.7 | 68.6

133. Secondary Outcome: Change From Baseline in EQ-5D-5L at Weeks 24 and 52: EQ-VAS
Description: as for outcome 67
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 237 | 238 | 234
  Week 24 | 8.456 (25.7204) | 19.282 (23.5220) | 17.500 (22.6981)
  Week 52: number analyzed (Participants) | 230 | 234 | 229
  Week 52 | 21.474 (25.5974) | 23.295 (23.6270) | 19.983 (24.7643)

134. Secondary Outcome: Change From Baseline in EQ-5D-5L at Weeks 24 and 52: EQ-5D Index
Description: as for outcome 68
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 70
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 238 | 240 | 234
units on a scale
  Week 24: number analyzed (Participants) | 237 | 238 | 234
  Week 24 | 0.060 (0.1558) | 0.124 (0.1476) | 0.117 (0.1307)
  Week 52: number analyzed (Participants) | 230 | 234 | 229
  Week 52 | 0.137 (0.1605) | 0.146 (0.1587) | 0.135 (0.1469)

135. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire Scores (Percent Work Time Missed) at Weeks 24 and 52
Description: as for outcome 32
Time Frame: Baseline, Weeks 24 and 52
Population: Analysis population is FAS2. Here, N (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 148 | 141 | 136
units on a scale
  Week 24 | -5.64 (28.355) | -3.77 (28.029) | -1.20 (17.127)
  Week 52: number analyzed (Participants) | 138 | 131 | 132
  Week 52 | -5.37 (25.365) | -4.47 (20.454) | -1.74 (17.084)

136. Secondary Outcome: Change From Baseline in WPAI Scores (Percent Impairment While Working) at Weeks 24 and 52
Description: as for outcome 32
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 135
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 125 | 124
units on a scale
  Week 24: number analyzed (Participants) | 126 | 125 | 123
  Week 24 | -12.14 (29.027) | -21.28 (25.621) | -20.08 (22.084)
  Week 52: number analyzed (Participants) | 118 | 121 | 124
  Week 52 | -21.27 (31.502) | -27.93 (25.263) | -22.10 (26.172)

137. Secondary Outcome: Change From Baseline in WPAI Scores (Percent Overall Work Impairment) at Weeks 24 and 52
Description: as for outcome 32
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 135
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 126 | 125 | 124
units on a scale
  Week 24: number analyzed (Participants) | 126 | 125 | 123
  Week 24 | -13.42 (29.916) | -21.68 (27.065) | -20.90 (22.814)
  Week 52: number analyzed (Participants) | 118 | 121 | 124
  Week 52 | -22.06 (32.092) | -28.19 (25.536) | -22.24 (26.920)

138. Secondary Outcome: Change From Baseline in WPAI Scores (Percent Activity Impairment Outside of Work) at Weeks 24 and 52
Description: as for outcome 32
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 135
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 237 | 238 | 234
units on a scale
  Week 24 | -10.80 (26.131) | -23.03 (25.559) | -21.07 (21.493)
  Week 52: number analyzed (Participants) | 230 | 234 | 229
  Week 52 | -24.13 (27.436) | -27.14 (25.657) | -26.11 (25.361)

139. Secondary Outcome: Percentage of Participants Who Achieved ACR 20 Response at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 69
Time Frame: Weeks 52, 68, 76, 84 and 100
Population: Analysis population is full analysis set 3 (FAS3) which included all participants still on treatment at Week 52. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | 68.7 | 78.9 | 77.0
  Week 68: number analyzed (Participants) | 222 | 229 | 218
  Week 68 | 77.0 | 85.2 | 80.7
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | 75.6 | 83.1 | 82.5
  Week 84: number analyzed (Participants) | 216 | 221 | 217
  Week 84 | 80.1 | 85.1 | 80.6
  Week 100: number analyzed (Participants) | 212 | 223 | 219
  Week 100 | 79.2 | 82.1 | 84.9

140. Secondary Outcome: Percentage of Participants Who Achieved ACR 50 Response at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 70
Time Frame: Weeks 52, 68, 76, 84 and 100
Population: Analysis population is FAS3 which included all participants still on treatment at Week 52. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 228 | 232 | 226
  Week 52 | 44.3 | 50.9 | 49.6
  Week 68: number analyzed (Participants) | 222 | 227 | 220
  Week 68 | 49.5 | 60.8 | 58.6
  Week 76: number analyzed (Participants) | 222 | 225 | 223
  Week 76 | 50.9 | 56.0 | 58.3
  Week 84: number analyzed (Participants) | 215 | 221 | 218
  Week 84 | 56.3 | 63.8 | 57.8
  Week 100: number analyzed (Participants) | 212 | 224 | 220
  Week 100 | 55.2 | 60.7 | 62.3

141. Secondary Outcome: Percentage of Participants Who Achieved ACR 70 Response at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 71
Time Frame: Weeks 52, 68, 76, 84 and 100
Population: as for outcome 140
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 226 | 232 | 226
  Week 52 | 19.5 | 29.7 | 28.3
  Week 68: number analyzed (Participants) | 223 | 228 | 219
  Week 68 | 27.8 | 35.5 | 36.1
  Week 76: number analyzed (Participants) | 222 | 225 | 223
  Week 76 | 27.9 | 36.4 | 32.7
  Week 84: number analyzed (Participants) | 216 | 222 | 218
  Week 84 | 29.6 | 42.8 | 39.4
  Week 100: number analyzed (Participants) | 213 | 224 | 220
  Week 100 | 34.3 | 39.3 | 38.6

142. Secondary Outcome: ACR Components at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 72
Time Frame: Weeks 52, 68, 76, 84 and 100
Population: Analysis population is FAS3 which included all participants still on treatment at Week 52. Here, n (number analyzed) signifies the number of participants analyzed for specified categories at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: Swollen Joint Count: number analyzed (Participants) | 228 | 232 | 226
  Week 52: Swollen Joint Count | 2.1 (3.58) | 2.1 (4.18) | 2.5 (4.83)
  Week 68: Swollen Joint Count: number analyzed (Participants) | 223 | 229 | 220
  Week 68: Swollen Joint Count | 1.6 (3.10) | 1.7 (3.87) | 2.0 (3.79)
  Week 76: Swollen Joint Count: number analyzed (Participants) | 222 | 225 | 223
  Week 76: Swollen Joint Count | 1.6 (3.17) | 1.8 (3.72) | 2.3 (4.59)
  Week 84: Swollen Joint Count: number analyzed (Participants) | 215 | 220 | 216
  Week 84: Swollen Joint Count | 1.6 (3.02) | 1.6 (3.82) | 2.0 (5.01)
  Week 100: Swollen Joint Count: number analyzed (Participants) | 213 | 224 | 220
  Week 100: Swollen Joint Count | 1.8 (3.75) | 1.6 (3.99) | 2.0 (4.11)
  Week 52: Tender Joint Count: number analyzed (Participants) | 228 | 232 | 226
  Week 52: Tender Joint Count | 7.4 (10.30) | 6.3 (8.20) | 7.2 (9.49)
  Week 68: Tender Joint Count: number analyzed (Participants) | 223 | 229 | 220
  Week 68: Tender Joint Count | 6.0 (8.83) | 5.0 (6.83) | 6.3 (9.27)
  Week 76: Tender Joint Count: number analyzed (Participants) | 222 | 225 | 223
  Week 76: Tender Joint Count | 5.7 (8.31) | 5.2 (7.18) | 6.2 (8.90)
  Week 84: Tender Joint Count: number analyzed (Participants) | 215 | 220 | 216
  Week 84: Tender Joint Count | 5.1 (7.32) | 4.7 (7.20) | 5.9 (9.22)
  Week 100: Tender Joint Count: number analyzed (Participants) | 213 | 224 | 220
  Week 100: Tender Joint Count | 5.5 (8.44) | 4.7 (6.80) | 6.0 (8.90)
  Week 52: Patient's Assessment of Pain: number analyzed (Participants) | 228 | 232 | 226
  Week 52: Patient's Assessment of Pain | 3.53 (2.267) | 3.12 (2.335) | 3.17 (2.343)
  Week 68: Patient's Assessment of Pain: number analyzed (Participants) | 223 | 230 | 222
  Week 68: Patient's Assessment of Pain | 3.26 (2.313) | 2.68 (2.240) | 2.64 (2.105)
  Week 76: Patient's Assessment of Pain: number analyzed (Participants) | 222 | 225 | 223
  Week 76: Patient's Assessment of Pain | 3.17 (2.271) | 2.73 (2.217) | 2.70 (2.115)
  Week 84: Patient's Assessment of Pain: number analyzed (Participants) | 217 | 222 | 219
  Week 84: Patient's Assessment of Pain | 2.97 (2.150) | 2.67 (2.181) | 2.65 (2.217)
  Week 100: Patient's Assessment of Pain: number analyzed (Participants) | 215 | 224 | 220
  Week 100: Patient's Assessment of Pain | 2.90 (2.221) | 2.59 (2.290) | 2.57 (2.138)
  Week 52: PtGA of Disease Activity: number analyzed (Participants) | 228 | 232 | 226
  Week 52: PtGA of Disease Activity | 3.68 (2.331) | 3.25 (2.380) | 3.24 (2.322)
  Week 68: PtGA of Disease Activity: number analyzed (Participants) | 223 | 230 | 222
  Week 68: PtGA of Disease Activity | 3.50 (2.355) | 2.95 (2.282) | 2.85 (2.213)
  Week 76: PtGA of Disease Activity: number analyzed (Participants) | 222 | 225 | 223
  Week 76: PtGA of Disease Activity | 3.25 (2.356) | 2.90 (2.273) | 2.95 (2.222)
  Week 84: PtGA of Disease Activity: number analyzed (Participants) | 217 | 222 | 219
  Week 84: PtGA of Disease Activity | 3.09 (2.273) | 2.88 (2.252) | 2.83 (2.222)
  Week 100: PtGA of Disease Activity: number analyzed (Participants) | 215 | 224 | 220
  Week 100: PtGA of Disease Activity | 3.15 (2.395) | 2.85 (2.378) | 2.60 (2.165)
  Week 52: PGA of Disease Activity: number analyzed (Participants) | 226 | 232 | 226
  Week 52: PGA of Disease Activity | 1.89 (1.654) | 1.78 (1.647) | 1.77 (1.617)
  Week 68: PGA of Disease Activity: number analyzed (Participants) | 223 | 227 | 217
  Week 68: PGA of Disease Activity | 1.63 (1.514) | 1.56 (1.538) | 1.61 (1.466)
  Week 76: PGA of Disease Activity: number analyzed (Participants) | 221 | 223 | 223
  Week 76: PGA of Disease Activity | 1.45 (1.469) | 1.67 (1.660) | 1.57 (1.524)
  Week 84: PGA of Disease Activity: number analyzed (Participants) | 213 | 220 | 216
  Week 84: PGA of Disease Activity | 1.55 (1.492) | 1.51 (1.619) | 1.50 (1.558)
  Week 100: PGA of Disease Activity: number analyzed (Participants) | 212 | 224 | 220
  Week 100: PGA of Disease Activity | 1.39 (1.510) | 1.49 (1.581) | 1.41 (1.405)
  Week 52: HAQ-DI score: number analyzed (Participants) | 228 | 232 | 226
  Week 52: HAQ-DI score | 0.9073 (0.63812) | 0.7942 (0.59711) | 0.7317 (0.58430)
  Week 68: HAQ-DI score: number analyzed (Participants) | 223 | 230 | 222
  Week 68: HAQ-DI score | 0.8425 (0.61757) | 0.7625 (0.59524) | 0.6836 (0.56049)
  Week 76: HAQ-DI score: number analyzed (Participants) | 222 | 225 | 223
  Week 76: HAQ-DI score | 0.8311 (0.62101) | 0.6978 (0.56588) | 0.6996 (0.55988)
  Week 84: HAQ-DI score: number analyzed (Participants) | 217 | 222 | 219
  Week 84: HAQ-DI score | 0.8076 (0.62465) | 0.7134 (0.59528) | 0.6775 (0.58870)
  Week 100: HAQ-DI score: number analyzed (Participants) | 215 | 224 | 220
  Week 100: HAQ-DI score | 0.7692 (0.59960) | 0.6747 (0.57213) | 0.6420 (0.56838)
  Week 52: CRP: number analyzed (Participants) | 225 | 232 | 226
  Week 52: CRP | 0.904 (1.6039) | 0.930 (1.2443) | 0.886 (1.2366)
  Week 68: CRP: number analyzed (Participants) | 218 | 228 | 220
  Week 68: CRP | 0.861 (1.1586) | 0.884 (1.3520) | 0.796 (1.1109)
  Week 76: CRP: number analyzed (Participants) | 220 | 224 | 223
  Week 76: CRP | 0.903 (1.4624) | 0.882 (1.2504) | 0.839 (1.1693)
  Week 84: CRP: number analyzed (Participants) | 217 | 222 | 217
  Week 84: CRP | 0.898 (1.3229) | 0.856 (1.1926) | 0.872 (1.3239)
  Week 100: CRP: number analyzed (Participants) | 211 | 223 | 220
  Week 100: CRP | 0.880 (1.3415) | 0.826 (1.2277) | 0.820 (1.1227)

143. Secondary Outcome: Change From Baseline in ACR Components at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 72
Time Frame: Baseline, Weeks 52, 68, 76, 84 and 100
Population: as for outcome 142
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: Swollen Joint Count: number analyzed (Participants) | 228 | 232 | 226
  Week 52: Swollen Joint Count | -10.2 (6.72) | -9.6 (6.30) | -10.4 (6.16)
  Week 68: Swollen Joint Count: number analyzed (Participants) | 223 | 229 | 220
  Week 68: Swollen Joint Count | -10.7 (6.76) | -10.0 (6.50) | -10.9 (7.22)
  Week 76: Swollen Joint Count: number analyzed (Participants) | 222 | 225 | 223
  Week 76: Swollen Joint Count | -10.7 (5.98) | -10.0 (6.33) | -10.7 (6.18)
  Week 84: Swollen Joint Count: number analyzed (Participants) | 215 | 220 | 216
  Week 84: Swollen Joint Count | -10.6 (6.06) | -10.1 (6.34) | -10.7 (7.08)
  Week 100: Swollen Joint Count: number analyzed (Participants) | 213 | 224 | 220
  Week 100: Swollen Joint Count | -10.6 (6.15) | -10.2 (6.88) | -10.8 (6.66)
  Week 52: Tender Joint Count: number analyzed (Participants) | 228 | 232 | 226
  Week 52: Tender Joint Count | -14.1 (11.38) | -13.5 (10.04) | -15.2 (10.45)
  Week 68: Tender Joint Count: number analyzed (Participants) | 223 | 229 | 220
  Week 68: Tender Joint Count | -15.7 (10.94) | -14.8 (10.15) | -16.0 (11.02)
  Week 76: Tender Joint Count: number analyzed (Participants) | 222 | 225 | 223
  Week 76: Tender Joint Count | -16.1 (10.97) | -14.7 (10.22) | -16.1 (10.91)
  Week 84: Tender Joint Count: number analyzed (Participants) | 215 | 220 | 216
  Week 84: Tender Joint Count | -16.6 (11.33) | -15.3 (10.50) | -16.0 (11.22)
  Week 100: Tender Joint Count: number analyzed (Participants) | 213 | 224 | 220
  Week 100: Tender Joint Count | -16.3 (11.27) | -15.3 (11.10) | -16.4 (10.70)
  Week 52: Patient's Assessment of Pain: number analyzed (Participants) | 228 | 232 | 226
  Week 52: Patient's Assessment of Pain | -2.78 (2.645) | -3.20 (2.557) | -2.92 (2.686)
  Week 68: Patient's Assessment of Pain: number analyzed (Participants) | 223 | 230 | 222
  Week 68: Patient's Assessment of Pain | -3.10 (2.707) | -3.62 (2.530) | -3.46 (2.574)
  Week 76: Patient's Assessment of Pain: number analyzed (Participants) | 222 | 225 | 223
  Week 76: Patient's Assessment of Pain | -3.18 (2.724) | -3.57 (2.566) | -3.38 (2.620)
  Week 84: Patient's Assessment of Pain: number analyzed (Participants) | 217 | 222 | 219
  Week 84: Patient's Assessment of Pain | -3.35 (2.595) | -3.64 (2.568) | -3.42 (2.669)
  Week 100: Patient's Assessment of Pain: number analyzed (Participants) | 215 | 224 | 220
  Week 100: Patient's Assessment of Pain | -3.41 (2.578) | -3.69 (2.625) | -3.52 (2.615)
  Week 52: PtGA of Disease Activity: number analyzed (Participants) | 228 | 232 | 226
  Week 52: PtGA of Disease Activity | -2.87 (2.761) | -3.29 (2.553) | -3.09 (2.523)
  Week 68: PtGA of Disease Activity: number analyzed (Participants) | 223 | 230 | 222
  Week 68: PtGA of Disease Activity | -3.08 (2.786) | -3.58 (2.446) | -3.49 (2.500)
  Week 76: PtGA of Disease Activity: number analyzed (Participants) | 222 | 225 | 223
  Week 76: PtGA of Disease Activity | -3.32 (2.860) | -3.63 (2.512) | -3.38 (2.501)
  Week 84: PtGA of Disease Activity: number analyzed (Participants) | 217 | 222 | 219
  Week 84: PtGA of Disease Activity | -3.46 (2.752) | -3.67 (2.572) | -3.50 (2.579)
  Week 100: PtGA of Disease Activity: number analyzed (Participants) | 215 | 224 | 220
  Week 100: PtGA of Disease Activity | -3.40 (2.846) | -3.67 (2.612) | -3.73 (2.493)
  Week 52: PGA of Disease Activity: number analyzed (Participants) | 226 | 232 | 226
  Week 52: PGA of Disease Activity | -4.79 (1.992) | -4.77 (2.001) | -4.82 (2.117)
  Week 68: PGA of Disease Activity: number analyzed (Participants) | 223 | 227 | 217
  Week 68: PGA of Disease Activity | -5.06 (2.037) | -4.98 (1.992) | -5.01 (2.105)
  Week 76: PGA of Disease Activity: number analyzed (Participants) | 221 | 223 | 223
  Week 76: PGA of Disease Activity | -5.23 (1.995) | -4.86 (2.044) | -5.03 (2.078)
  Week 84: PGA of Disease Activity: number analyzed (Participants) | 213 | 220 | 216
  Week 84: PGA of Disease Activity | -5.13 (2.040) | -5.06 (2.074) | -5.09 (2.142)
  Week 100: PGA of Disease Activity: number analyzed (Participants) | 212 | 224 | 220
  Week 100: PGA of Disease Activity | -5.26 (2.098) | -5.05 (2.011) | -5.18 (2.044)
  Week 52: HAQ-DI score: number analyzed (Participants) | 227 | 232 | 226
  Week 52: HAQ-DI score | -0.3899 (0.58250) | -0.4801 (0.56246) | -0.5111 (0.58347)
  Week 68: HAQ-DI score: number analyzed (Participants) | 222 | 230 | 222
  Week 68: HAQ-DI score | -0.4668 (0.59226) | -0.5120 (0.54928) | -0.5631 (0.54528)
  Week 76: HAQ-DI score: number analyzed (Participants) | 221 | 225 | 223
  Week 76: HAQ-DI score | -0.4740 (0.57852) | -0.5694 (0.56421) | -0.5448 (0.54739)
  Week 84: HAQ-DI score: number analyzed (Participants) | 216 | 222 | 219
  Week 84: HAQ-DI score | -0.5041 (0.59716) | -0.5653 (0.59488) | -0.5656 (0.57921)
  Week 100: HAQ-DI score: number analyzed (Participants) | 214 | 224 | 220
  Week 100: HAQ-DI score | -0.5356 (0.56707) | -0.5859 (0.58199) | -0.6000 (0.56858)
  Week 52: CRP: number analyzed (Participants) | 225 | 232 | 226
  Week 52: CRP | -1.262 (2.8315) | -1.021 (2.2301) | -0.959 (2.4188)
  Week 68: CRP: number analyzed (Participants) | 218 | 228 | 220
  Week 68: CRP | -1.212 (2.3061) | -1.081 (2.1585) | -1.060 (2.3334)
  Week 76: CRP: number analyzed (Participants) | 220 | 224 | 223
  Week 76: CRP | -1.283 (2.8163) | -1.098 (2.3654) | -1.017 (2.2801)
  Week 84: CRP: number analyzed (Participants) | 217 | 222 | 217
  Week 84: CRP | -1.230 (2.4262) | -1.101 (2.1216) | -0.940 (2.3781)
  Week 100: CRP: number analyzed (Participants) | 211 | 223 | 220
  Week 100: CRP | -1.244 (2.5828) | -1.129 (2.2261) | -1.042 (2.0600)

144. Secondary Outcome: Percent Change From Baseline in ACR Components at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 72
Time Frame: Baseline, Weeks 52, 68, 76, 84 and 100
Population: as for outcome 142
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percent change
  Week 52: Swollen Joint Count: number analyzed (Participants) | 228 | 232 | 226
  Week 52: Swollen Joint Count | -82.64 (30.161) | -83.03 (30.210) | -84.27 (23.698)
  Week 68: Swollen Joint Count: number analyzed (Participants) | 223 | 229 | 220
  Week 68: Swollen Joint Count | -87.41 (24.049) | -86.08 (29.764) | -86.41 (22.642)
  Week 76: Swollen Joint Count: number analyzed (Participants) | 222 | 225 | 223
  Week 76: Swollen Joint Count | -87.98 (20.617) | -86.05 (21.096) | -85.82 (22.291)
  Week 84: Swollen Joint Count: number analyzed (Participants) | 215 | 220 | 216
  Week 84: Swollen Joint Count | -87.72 (22.243) | -87.68 (23.304) | -87.16 (24.888)
  Week 100: Swollen Joint Count: number analyzed (Participants) | 213 | 224 | 220
  Week 100: Swollen Joint Count | -87.61 (21.214) | -86.19 (40.865) | -86.31 (24.106)
  Week 52: Tender Joint Count: number analyzed (Participants) | 228 | 232 | 226
  Week 52: Tender Joint Count | -67.29 (35.725) | -70.18 (32.062) | -70.54 (31.311)
  Week 68: Tender Joint Count: number analyzed (Participants) | 223 | 229 | 220
  Week 68: Tender Joint Count | -74.28 (29.764) | -75.63 (29.437) | -74.40 (29.760)
  Week 76: Tender Joint Count: number analyzed (Participants) | 222 | 225 | 223
  Week 76: Tender Joint Count | -75.71 (27.653) | -74.71 (29.728) | -75.11 (28.559)
  Week 84: Tender Joint Count: number analyzed (Participants) | 215 | 220 | 216
  Week 84: Tender Joint Count | -77.21 (27.045) | -78.01 (26.112) | -75.45 (32.489)
  Week 100: Tender Joint Count: number analyzed (Participants) | 213 | 224 | 220
  Week 100: Tender Joint Count | -77.04 (27.510) | -75.96 (32.600) | -76.21 (27.345)
  Week 52: Patient's Assessment of Pain: number analyzed (Participants) | 228 | 232 | 226
  Week 52: Patient's Assessment of Pain | -39.52 (44.939) | -48.81 (39.191) | -43.86 (45.891)
  Week 68: Patient's Assessment of Pain: number analyzed (Participants) | 223 | 230 | 222
  Week 68: Patient's Assessment of Pain | -44.91 (44.371) | -55.77 (38.780) | -52.43 (41.186)
  Week 76: Patient's Assessment of Pain: number analyzed (Participants) | 222 | 225 | 223
  Week 76: Patient's Assessment of Pain | -46.02 (44.989) | -54.38 (39.135) | -51.34 (41.903)
  Week 84: Patient's Assessment of Pain: number analyzed (Participants) | 217 | 222 | 219
  Week 84: Patient's Assessment of Pain | -49.64 (40.991) | -55.28 (40.388) | -52.59 (43.131)
  Week 100: Patient's Assessment of Pain: number analyzed (Participants) | 215 | 224 | 220
  Week 100: Patient's Assessment of Pain | -50.82 (42.970) | -56.36 (41.310) | -54.27 (40.819)
  Week 52: PtGA of Disease Activity: number analyzed (Participants) | 228 | 232 | 226
  Week 52: PtGA of Disease Activity | -39.70 (44.981) | -48.48 (38.982) | -46.07 (40.614)
  Week 68: PtGA of Disease Activity: number analyzed (Participants) | 223 | 230 | 222
  Week 68: PtGA of Disease Activity | -42.93 (44.220) | -53.84 (35.096) | -52.47 (38.155)
  Week 76: PtGA of Disease Activity: number analyzed (Participants) | 222 | 225 | 223
  Week 76: PtGA of Disease Activity | -46.42 (45.106) | -54.41 (35.276) | -50.66 (40.992)
  Week 84: PtGA of Disease Activity: number analyzed (Participants) | 217 | 222 | 219
  Week 84: PtGA of Disease Activity | -49.38 (42.315) | -54.17 (37.132) | -51.86 (44.532)
  Week 100: PtGA of Disease Activity: number analyzed (Participants) | 215 | 224 | 220
  Week 100: PtGA of Disease Activity | -48.17 (44.804) | -55.08 (37.052) | -57.09 (34.970)
  Week 52: PGA of Disease Activity: number analyzed (Participants) | 226 | 232 | 226
  Week 52: PGA of Disease Activity | -71.24 (24.771) | -72.95 (24.168) | -72.58 (24.579)
  Week 68: PGA of Disease Activity: number analyzed (Participants) | 223 | 227 | 217
  Week 68: PGA of Disease Activity | -74.76 (23.290) | -76.00 (22.550) | -74.48 (26.280)
  Week 76: PGA of Disease Activity: number analyzed (Participants) | 221 | 223 | 223
  Week 76: PGA of Disease Activity | -77.68 (23.015) | -74.42 (25.014) | -75.56 (23.613)
  Week 84: PGA of Disease Activity: number analyzed (Participants) | 213 | 220 | 216
  Week 84: PGA of Disease Activity | -75.77 (23.674) | -76.77 (24.433) | -76.49 (24.355)
  Week 100: PGA of Disease Activity: number analyzed (Participants) | 212 | 224 | 220
  Week 100: PGA of Disease Activity | -78.11 (24.049) | -77.15 (23.217) | -77.82 (22.733)
  Week 52: HAQ-DI score: number analyzed (Participants) | 224 | 223 | 223
  Week 52: HAQ-DI score | -27.27 (54.587) | -33.28 (64.067) | -35.17 (66.105)
  Week 68: HAQ-DI score: number analyzed (Participants) | 220 | 221 | 219
  Week 68: HAQ-DI score | -33.34 (49.027) | -37.47 (57.370) | -44.33 (44.064)
  Week 76: HAQ-DI score: number analyzed (Participants) | 219 | 216 | 220
  Week 76: HAQ-DI score | -34.38 (47.311) | -40.08 (58.932) | -41.84 (47.877)
  Week 84: HAQ-DI score: number analyzed (Participants) | 214 | 214 | 216
  Week 84: HAQ-DI score | -36.73 (47.541) | -40.10 (58.703) | -43.18 (52.116)
  Week 100: HAQ-DI score: number analyzed (Participants) | 212 | 215 | 217
  Week 100: HAQ-DI score | -40.36 (44.407) | -42.84 (54.187) | -47.54 (47.265)
  Week 52: CRP: number analyzed (Participants) | 225 | 232 | 226
  Week 52: CRP | -2.67 (205.761) | -23.41 (104.622) | -1.34 (194.673)
  Week 68: CRP: number analyzed (Participants) | 218 | 228 | 220
  Week 68: CRP | -1.68 (330.574) | -28.38 (138.159) | -13.91 (174.522)
  Week 76: CRP: number analyzed (Participants) | 220 | 224 | 223
  Week 76: CRP | -10.76 (226.332) | 7.85 (502.170) | -24.22 (110.486)
  Week 84: CRP: number analyzed (Participants) | 217 | 222 | 217
  Week 84: CRP | -0.72 (387.986) | -26.87 (114.471) | -19.89 (131.695)
  Week 100: CRP: number analyzed (Participants) | 211 | 223 | 220
  Week 100: CRP | -4.33 (196.246) | -23.99 (150.816) | -14.35 (171.666)

145. Secondary Outcome: Percentage of Participants Who Maintained an ACR 20 Response at Week 100 Among Participants Who Achieved an ACR 20 Response at Week 52
Description: as for outcome 69
Time Frame: Week 100
Population: FAS3 among participants who achieved ACR20 response at Week 52.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 147 | 178 | 171
percentage of participants | 94.6 | 90.4 | 93.0

146. Secondary Outcome: Percentage of Participants Who Maintained an ACR 50 Response at Week 100 Among Participants Who Achieved an ACR 50 Response at Week 52
Description: as for outcome 70
Time Frame: Week 100
Population: FAS3 among participants who achieved ACR50 response at Week 52.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 96 | 116 | 111
percentage of participants | 81.3 | 81.9 | 83.8

147. Secondary Outcome: Percentage of Participants Who Maintained an ACR 70 Response at Week 100 Among Participants Who Achieved an ACR 70 Response at Week 52
Description: as for outcome 77
Time Frame: Week 100
Population: FAS3 among participants who achieved ACR70 response at Week 52.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 43 | 68 | 64
percentage of participants | 65.1 | 80.9 | 71.9

148. Secondary Outcome: Change From Baseline in HAQ-DI Score at Weeks 52, 68, 76, 84 and 100
Description: HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3, where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning. Negative change from baseline indicates improvement of physical function.
Time Frame: Baseline, Weeks 52, 68, 76, 84 and 100
Population: as for outcome 140
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | -0.3899 (0.58250) | -0.4801 (0.56246) | -0.5111 (0.58347)
  Week 68: number analyzed (Participants) | 222 | 230 | 222
  Week 68 | -0.4668 (0.59226) | -0.5120 (0.54928) | -0.5631 (0.54528)
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | -0.4740 (0.57852) | -0.5694 (0.56421) | -0.5448 (0.54739)
  Week 84: number analyzed (Participants) | 216 | 222 | 219
  Week 84 | -0.5041 (0.59716) | -0.5653 (0.59488) | -0.5656 (0.57921)
  Week 100: number analyzed (Participants) | 214 | 224 | 220
  Week 100 | -0.5356 (0.56707) | -0.5859 (0.58199) | -0.6000 (0.56858)

149. Secondary Outcome: Percentage of Participants Who Achieved a Clinically Meaningful Improvement (>=0.35 Improvement From Baseline) in HAQ-DI Score at Weeks 52, 68, 76, 84 and 100 Among Participants With HAQ-DI Score >=0.35 at Baseline
Description: HAQ-DI score assess functional status of participant. It is 20 question instrument that assess degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area were scored from 0=indicating no difficulty, to 3=indicating inability to perform a task in that area. Total HAQ score is average of the computed categories scores ranging from 0-3, where 0=least difficulty and 3=extreme difficulty. Lower scores are indicative of better functioning and a decrease of 0.35 from baseline in HAQ-DI score indicates a meaningful improvement.
Time Frame: Weeks 52, 68, 76, 84 and 100
Population: Analysis population is FAS3 among participants with HAQ-DI score >=0.35 at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 219 | 213 | 211
percentage of participants
  Week 52: number analyzed (Participants) | 219 | 213 | 210
  Week 52 | 51.1 | 60.6 | 63.3
  Week 68: number analyzed (Participants) | 215 | 211 | 206
  Week 68 | 57.2 | 64.9 | 69.4
  Week 76: number analyzed (Participants) | 214 | 206 | 207
  Week 76 | 59.3 | 68.4 | 64.7
  Week 84: number analyzed (Participants) | 209 | 205 | 203
  Week 84 | 58.9 | 66.8 | 65.5
  Week 100: number analyzed (Participants) | 207 | 205 | 204
  Week 100 | 63.3 | 70.7 | 70.1

150. Secondary Outcome: Percentage of Participants Who Maintained a HAQ-DI Response (>=0.35 Improvement From Baseline in HAQ-DI Score) at Week 100 Among Participants Who Achieved a HAQ-DI Response at Week 52
Description: as for outcome 149
Time Frame: Week 100
Population: Analysis population is FAS3 among participants with HAQ-DI Score >=0.35 at Baseline and who achieved a HAQ-DI response at Week 52. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 107 | 125 | 131
percentage of participants | 91.6 | 90.4 | 88.5

151. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 (CRP) Response at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 81
Time Frame: Weeks 52, 68, 76, 84 and 100
Population: as for outcome 140
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 225 | 232 | 225
  Week 52 | 89.3 | 89.7 | 90.2
  Week 68: number analyzed (Participants) | 218 | 227 | 218
  Week 68 | 92.7 | 92.5 | 92.7
  Week 76: number analyzed (Participants) | 220 | 224 | 223
  Week 76 | 94.1 | 90.2 | 93.3
  Week 84: number analyzed (Participants) | 213 | 218 | 212
  Week 84 | 94.8 | 92.7 | 92.5
  Week 100: number analyzed (Participants) | 210 | 223 | 219
  Week 100 | 94.3 | 90.6 | 92.7

152. Secondary Outcome: Percentage of Participants Who Achieved a DAS28 (CRP) Remission at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 82
Time Frame: Weeks 52, 68, 76, 84 and 100
Population: as for outcome 140
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 225 | 232 | 225
  Week 52 | 34.7 | 39.7 | 40.4
  Week 68: number analyzed (Participants) | 218 | 227 | 218
  Week 68 | 39.0 | 44.9 | 49.1
  Week 76: number analyzed (Participants) | 220 | 224 | 223
  Week 76 | 43.2 | 44.2 | 43.5
  Week 84: number analyzed (Participants) | 213 | 218 | 212
  Week 84 | 41.8 | 50.9 | 48.1
  Week 100: number analyzed (Participants) | 210 | 223 | 219
  Week 100 | 42.4 | 47.5 | 51.6

153. Secondary Outcome: Change From Baseline in DAS28 (CRP) Score at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 24
Time Frame: Baseline, Weeks 52, 68, 76, 84 and 100
Population: as for outcome 140
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 225 | 232 | 225
  Week 52 | -2.14 (1.142) | -2.08 (1.124) | -2.14 (1.118)
  Week 68: number analyzed (Participants) | 218 | 227 | 218
  Week 68 | -2.29 (1.132) | -2.25 (1.170) | -2.30 (1.143)
  Week 76: number analyzed (Participants) | 220 | 224 | 223
  Week 76 | -2.35 (1.110) | -2.24 (1.147) | -2.24 (1.087)
  Week 84: number analyzed (Participants) | 213 | 218 | 212
  Week 84 | -2.40 (1.087) | -2.35 (1.181) | -2.31 (1.156)
  Week 100: number analyzed (Participants) | 210 | 223 | 219
  Week 100 | -2.42 (1.144) | -2.37 (1.215) | -2.36 (1.120)

154. Secondary Outcome: Percentage of Participants Who Achieved a Response Based on Modified Psoriatic Arthritis Responder Criteria (PsARC) at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 25
Time Frame: Weeks 52, 68, 76, 84 and 100
Population: as for outcome 140
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 226 | 232 | 226
  Week 52 | 81.4 | 86.2 | 83.6
  Week 68: number analyzed (Participants) | 223 | 227 | 218
  Week 68 | 84.3 | 89.9 | 87.6
  Week 76: number analyzed (Participants) | 221 | 223 | 223
  Week 76 | 84.6 | 88.8 | 90.6
  Week 84: number analyzed (Participants) | 214 | 220 | 217
  Week 84 | 87.4 | 87.7 | 87.6
  Week 100: number analyzed (Participants) | 212 | 224 | 220
  Week 100 | 86.3 | 89.3 | 88.6

155. Secondary Outcome: Percentage of Participants With Resolution of Enthesitis (LEI) at Weeks 52, 76 and 100 Among the Participants With Enthesitis (LEI) at Baseline
Description: as for outcome 26
Time Frame: Weeks 52, 76, and 100
Population: Analysis population is FAS3 among the participants with enthesitis (LEI) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 165 | 147 | 160
percentage of participants
  Week 52: number analyzed (Participants) | 165 | 147 | 159
  Week 52 | 67.3 | 66.0 | 61.0
  Week 76: number analyzed (Participants) | 159 | 142 | 157
  Week 76 | 72.3 | 71.8 | 67.5
  Week 100: number analyzed (Participants) | 153 | 142 | 155
  Week 100 | 75.2 | 77.5 | 67.7

156. Secondary Outcome: Change From Baseline in Enthesitis Score (Based on LEI) at Weeks 52, 76 and 100 Among the Participants With Enthesitis at Baseline
Description: as for outcome 28
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 155
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 165 | 147 | 160
units on a scale
  Week 52: number analyzed (Participants) | 163 | 146 | 155
  Week 52 | -2.1 (1.59) | -1.9 (1.66) | -2.1 (1.72)
  Week 76: number analyzed (Participants) | 157 | 141 | 154
  Week 76 | -2.3 (1.52) | -2.1 (1.66) | -2.2 (1.69)
  Week 100: number analyzed (Participants) | 151 | 141 | 152
  Week 100 | -2.4 (1.70) | -2.1 (1.65) | -2.2 (1.80)

157. Secondary Outcome: Percentage of Participants With Resolution of Dactylitis at Weeks 52, 76 and 100 Among Participants With Dactylitis at Baseline
Description: as for outcome 27
Time Frame: Weeks 52, 76 and 100
Population: Analysis population is FAS3 among participants with dactylitis at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 92 | 104 | 110
percentage of participants
  Week 52: number analyzed (Participants) | 92 | 104 | 109
  Week 52 | 78.3 | 81.7 | 80.7
  Week 76: number analyzed (Participants) | 91 | 100 | 108
  Week 76 | 80.2 | 84.0 | 82.4
  Week 100: number analyzed (Participants) | 86 | 101 | 105
  Week 100 | 83.7 | 91.1 | 82.9

158. Secondary Outcome: Change From Baseline in Dactylitis Scores at Weeks 52, 76 and 100 Among the Participants With Dactylitis at Baseline
Description: as for outcome 29
Time Frame: Baseline, Weeks 52, 76 and 100
Population: Analysis population is FAS3 among the participants with dactylitis at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 92 | 104 | 110
units on a scale
  Week 52: number analyzed (Participants) | 92 | 104 | 109
  Week 52 | -7.4 (9.22) | -7.3 (9.78) | -7.4 (8.66)
  Week 76: number analyzed (Participants) | 91 | 100 | 108
  Week 76 | -8.0 (9.55) | -7.8 (10.24) | -7.6 (8.93)
  Week 100: number analyzed (Participants) | 86 | 101 | 105
  Week 100 | -8.1 (9.63) | -7.9 (10.12) | -7.9 (9.14)

159. Secondary Outcome: Change From Baseline in PASDAS Score at Weeks 52, 76 and 100
Description: as for outcome 30
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 140
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 220 | 230 | 221
  Week 52 | -3.054 (1.4954) | -3.189 (1.5216) | -3.184 (1.4576)
  Week 76: number analyzed (Participants) | 215 | 220 | 220
  Week 76 | -3.503 (1.4708) | -3.418 (1.5646) | -3.436 (1.4428)
  Week 100: number analyzed (Participants) | 204 | 221 | 215
  Week 100 | -3.574 (1.4785) | -3.586 (1.5425) | -3.549 (1.4635)

160. Secondary Outcome: Percentage of Participants With Low or Very Low Disease Activity Based on PASDAS at Weeks 52, 76 and 100
Description: PASDAS (score range of 0 to 10, where higher score indicated more severe disease) is a composite score of overall disease activity combining PtGA of Disease Activity (arthritis and psoriasis, using VAS [0-100 mm, 0=excellent and 100= poor), PGA of Disease Activity (using VAS [0-100 mm, 0=no arthritis activity and 100=extremely active arthritis]), swollen joint count (0-66 joints), tender joint count (0-68 joints), CRP (mg/L), enthesitis based on LEI (0= 0 sites with tenderness to 6= worst possible score; 6 sites with tenderness), tender dactylitis count (scoring each digit from 0-3 [where 0= no tenderness and 3= extreme tenderness] and recoding to 0-1, where any score > 0 equaled 1), and the PCS score with score range 0-100 (higher score-better quality of life) of the SF-36 health survey. The cutoffs for disease activity were 3.2 (low) to 5.4 (high). Negative changes from baseline indicate improvement of overall disease activity. Low: PASDAS <= 3.2; Very low: PASDAS <= 1.9.
Time Frame: Weeks 52, 76 and 100
Population: Analysis population is FAS3. Here, n (number analyzed) signifies the number of participants analyzed for specified categories at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: Low: number analyzed (Participants) | 223 | 232 | 225
  Week 52: Low | 39.0 | 44.8 | 46.7
  Week 52: Very Low: number analyzed (Participants) | 223 | 232 | 225
  Week 52: Very Low | 13.0 | 22.0 | 16.0
  Week 76: Low: number analyzed (Participants) | 219 | 222 | 223
  Week 76: Low | 52.1 | 50.0 | 49.8
  Week 76: Very Low: number analyzed (Participants) | 219 | 222 | 223
  Week 76: Very Low | 18.3 | 23.4 | 22.0
  Week 100: Low: number analyzed (Participants) | 206 | 223 | 218
  Week 100: Low | 55.3 | 54.7 | 57.8
  Week 100: Very Low: number analyzed (Participants) | 206 | 223 | 218
  Week 100: Very Low | 19.9 | 26.0 | 23.4

161. Secondary Outcome: Change From Baseline in GRAPPA Composite Score (GRACE) at Weeks 52, 76 and 100
Description: as for outcome 31
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 140
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 225 | 232 | 226
  Week 52 | -3.105 (1.6208) | -3.266 (1.6443) | -3.298 (1.5457)
  Week 76: number analyzed (Participants) | 220 | 223 | 223
  Week 76 | -3.499 (1.6303) | -3.528 (1.5778) | -3.541 (1.5048)
  Week 100: number analyzed (Participants) | 211 | 223 | 220
  Week 100 | -3.561 (1.6389) | -3.656 (1.6071) | -3.664 (1.5205)

162. Secondary Outcome: Percentage of Participants With Low Disease Activity Based on Group of Research and Assessment of Psoriasis and Psoriatic Arthritis Composite (GRACE) Score Index at Weeks 52, 76 and 100
Description: as for outcome 92
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 140
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 226 | 232 | 226
  Week 52 | 35.4 | 42.7 | 43.8
  Week 76: number analyzed (Participants) | 221 | 223 | 223
  Week 76 | 45.7 | 48.9 | 49.8
  Week 100: number analyzed (Participants) | 212 | 223 | 220
  Week 100 | 48.1 | 51.1 | 54.5

163. Secondary Outcome: Change From Baseline in DAPSA at Weeks 52, 68, 76, 84 and 100
Description: as for outcome 37
Time Frame: Baseline, Weeks 52, 68, 76, 84 and 100
Population: as for outcome 140
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 225 | 232 | 225
  Week 52 | -31.274 (18.8900) | -30.604 (17.5366) | -32.563 (16.4765)
  Week 68: number analyzed (Participants) | 218 | 227 | 218
  Week 68 | -33.918 (18.0463) | -33.146 (18.1727) | -34.900 (17.5749)
  Week 76: number analyzed (Participants) | 220 | 224 | 223
  Week 76 | -34.391 (17.4074) | -33.062 (17.5186) | -34.590 (16.5401)
  Week 84: number analyzed (Participants) | 213 | 218 | 212
  Week 84 | -35.240 (17.7891) | -33.622 (18.0612) | -34.570 (18.2685)
  Week 100: number analyzed (Participants) | 210 | 223 | 219
  Week 100 | -34.819 (17.9807) | -34.019 (19.2678) | -35.549 (16.5533)

164. Secondary Outcome: Percentage of Participants With Low Disease Activity or Remission Based on DAPSA at Weeks 52, 68, 76, 84 and 100
Description: DAPSA assessed the joint domain of PsA and was derived from the sum of the following components: tender joint count (0-68), swollen joint count (0-66), CRP level (mg/dL), patient assessment of pain (0-10 cm VAS, 0=no pain, 10=worst possible pain), and patient's global assessment of disease activity on arthritis (0 to 10 cm VAS, 0=excellent and 10=poor). A higher score indicates more active disease activity. The assessment does not have a score range with an upper or lower bound. Low: DAPSA<=14; Remission: DAPSA<=4.
Time Frame: Weeks 52, 68, 76, 84 and 100
Population: as for outcome 142
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: Low Disease Activity: number analyzed (Participants) | 225 | 232 | 225
  Week 52: Low Disease Activity | 50.7 | 55.2 | 55.6
  Week 52: Remission: number analyzed (Participants) | 225 | 232 | 225
  Week 52: Remission | 10.2 | 19.4 | 17.3
  Week 68: Low Disease Activity: number analyzed (Participants) | 218 | 227 | 218
  Week 68: Low Disease Activity | 54.1 | 64.3 | 63.3
  Week 68: Remission: number analyzed (Participants) | 218 | 227 | 218
  Week 68: Remission | 15.6 | 23.8 | 23.9
  Week 76: Low Disease Activity: number analyzed (Participants) | 220 | 224 | 223
  Week 76: Low Disease Activity | 58.2 | 61.2 | 61.4
  Week 76: Remission: number analyzed (Participants) | 220 | 224 | 223
  Week 76: Remission | 16.4 | 26.8 | 19.7
  Week 84: Low Disease Activity: number analyzed (Participants) | 213 | 218 | 212
  Week 84: Low Disease Activity | 60.6 | 66.5 | 64.6
  Week 84: Remission: number analyzed (Participants) | 213 | 218 | 212
  Week 84: Remission | 17.8 | 28.0 | 23.6
  Week 100: Low Disease Activity: number analyzed (Participants) | 210 | 223 | 219
  Week 100: Low Disease Activity | 61.9 | 65.9 | 68.9
  Week 100: Remission: number analyzed (Participants) | 210 | 223 | 219
  Week 100: Remission | 18.6 | 26.9 | 23.7

165. Secondary Outcome: Change From Baseline in mCPDAI Score at Weeks 52, 76 and 100
Description: as for outcome 36
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 140
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 223 | 230 | 222
  Week 52 | -3.78 (2.392) | -3.83 (2.458) | -4.14 (2.358)
  Week 76: number analyzed (Participants) | 217 | 221 | 220
  Week 76 | -4.39 (2.425) | -4.16 (2.539) | -4.47 (2.347)
  Week 100: number analyzed (Participants) | 207 | 221 | 216
  Week 100 | -4.44 (2.484) | -4.38 (2.433) | -4.52 (2.519)

166. Secondary Outcome: Percentage of Participants With Low Disease Activity Based on mCPDAI at Weeks 52, 76 and 100
Description: as for outcome 95
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 140
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 226 | 232 | 226
  Week 52 | 56.6 | 61.2 | 60.6
  Week 76: number analyzed (Participants) | 221 | 223 | 223
  Week 76 | 64.3 | 63.7 | 68.6
  Week 100: number analyzed (Participants) | 209 | 223 | 219
  Week 100 | 67.5 | 71.7 | 68.0

167. Secondary Outcome: Percentage of Participants Who Achieved Minimal Disease Activity (MDA) at Weeks 52, 76 and 100
Description: as for outcome 38
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 140
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 228 | 232 | 226
  Week 52 | 32.0 | 32.8 | 37.2
  Week 76: number analyzed (Participants) | 222 | 225 | 223
  Week 76 | 34.7 | 40.0 | 39.0
  Week 100: number analyzed (Participants) | 212 | 224 | 220
  Week 100 | 42.5 | 44.6 | 42.7

168. Secondary Outcome: Percentage of Participants With VLDA at Weeks 52, 76 and 100
Description: as for outcome 97
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 140
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 228 | 232 | 226
  Week 52 | 7.0 | 16.8 | 12.4
  Week 76: number analyzed (Participants) | 222 | 225 | 223
  Week 76 | 12.2 | 19.6 | 14.8
  Week 100: number analyzed (Participants) | 213 | 224 | 220
  Week 100 | 14.6 | 18.8 | 15.0

169. Secondary Outcome: Change From Baseline in BASDAI Score at Weeks 52, 76 and 100 Among Participants With Spondylitis and Peripheral Arthritis and BASDAI Score>0 at Baseline
Description: as for outcome 39
Time Frame: Baseline, Weeks 52, 76 and 100
Population: Analysis population is FAS3 among participants with spondylitis and peripheral arthritis and BASDAI Score>0 at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 88 | 63 | 79
units on a scale
  Week 52 | -2.986 (2.4945) | -2.923 (2.5194) | -3.084 (2.1843)
  Week 76: number analyzed (Participants) | 85 | 61 | 77
  Week 76 | -3.311 (2.6106) | -3.377 (2.5969) | -3.129 (2.1122)
  Week 100: number analyzed (Participants) | 82 | 61 | 76
  Week 100 | -3.718 (2.3960) | -3.472 (2.5233) | -3.330 (2.1598)

170. Secondary Outcome: Percentage of Participants Who Achieved >= 20%, >=50%, >=70%, and >=90% Improvement From Baseline in BASDAI Score at Weeks 52, 76 and 100 Among the Participants With Spondylitis and Peripheral Arthritis and BASDAI Score >0 at Baseline
Description: as for outcome 39
Time Frame: Weeks 52, 76 and 100
Population: Analysis population is FAS3 among participants with spondylitis and peripheral arthritis and BASDAI score >0 at Baseline. Here, n (number analyzed) signifies the number of participants analyzed for specified categories at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 88 | 63 | 79
percentage of participants
  Week 52: Participants with >=20% Improvement | 71.6 | 69.8 | 79.7
  Week 76: Participants with >=20% Improvement: number analyzed (Participants) | 85 | 61 | 77
  Week 76: Participants with >=20% Improvement | 74.1 | 82.0 | 81.8
  Week 100: Participants with >=20% Improvement: number analyzed (Participants) | 82 | 61 | 76
  Week 100: Participants with >=20% Improvement | 87.8 | 77.0 | 82.9
  Week 52: Participants with >=50% Improvement | 50.0 | 42.9 | 50.6
  Week 76: Participants with >=50% Improvement: number analyzed (Participants) | 85 | 61 | 77
  Week 76: Participants with >=50% Improvement | 52.9 | 52.5 | 50.6
  Week 100: Participants with >=50% Improvement: number analyzed (Participants) | 82 | 61 | 76
  Week 100: Participants with >=50% Improvement | 59.8 | 57.4 | 55.3
  Week 52: Participants with >=70% Improvement | 23.9 | 27.0 | 30.4
  Week 76: Participants with >=70% Improvement: number analyzed (Participants) | 85 | 61 | 77
  Week 76: Participants with >=70% Improvement | 31.8 | 31.1 | 26.0
  Week 100: Participants with >=70% Improvement: number analyzed (Participants) | 82 | 61 | 76
  Week 100: Participants with >=70% Improvement | 32.9 | 39.3 | 32.9
  Week 52: Participants with >=90% Improvement | 6.8 | 11.1 | 8.9
  Week 76: Participants with >=90% Improvement: number analyzed (Participants) | 85 | 61 | 77
  Week 76: Participants with >=90% Improvement | 11.8 | 13.1 | 7.8
  Week 100: Participants with >=90% Improvement: number analyzed (Participants) | 82 | 61 | 76
  Week 100: Participants with >=90% Improvement | 18.3 | 11.5 | 9.2

171. Secondary Outcome: Change From Baseline in PASI Score at Weeks 52, 76 and 100 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 44
Time Frame: Baseline, Weeks 52, 76 and 100
Population: Analysis population is FAS3 among participants with >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (mild) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 169 | 174
units on a scale
  Week 52: number analyzed (Participants) | 171 | 169 | 173
  Week 52 | -11.030 (10.0077) | -11.991 (12.1194) | -12.875 (11.2905)
  Week 76: number analyzed (Participants) | 166 | 165 | 172
  Week 76 | -11.313 (10.0631) | -11.991 (12.2656) | -13.242 (11.8845)
  Week 100: number analyzed (Participants) | 160 | 164 | 170
  Week 100 | -11.089 (10.0239) | -12.101 (12.1322) | -13.274 (11.9673)

172. Secondary Outcome: Percentage of Participants Who Achieved PASI 50 Response at Weeks 52, 76 and 100 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 101
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 171
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 169 | 174
percentage of participants
  Week 52: number analyzed (Participants) | 171 | 169 | 173
  Week 52 | 95.9 | 97.0 | 98.3
  Week 76: number analyzed (Participants) | 166 | 165 | 172
  Week 76 | 97.6 | 96.4 | 97.1
  Week 100: number analyzed (Participants) | 160 | 164 | 170
  Week 100 | 95.6 | 97.0 | 98.2

173. Secondary Outcome: Percentage of Participants Who Achieved PASI 75 Response at Weeks 52, 76 and 100 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 102
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 171
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 169 | 174
percentage of participants
  Week 52: number analyzed (Participants) | 171 | 169 | 173
  Week 52 | 88.3 | 88.8 | 91.9
  Week 76: number analyzed (Participants) | 166 | 165 | 172
  Week 76 | 92.8 | 87.9 | 93.0
  Week 100: number analyzed (Participants) | 160 | 164 | 170
  Week 100 | 91.9 | 87.8 | 89.4

174. Secondary Outcome: Percentage of Participants Who Achieved PASI 90 Response at Weeks 52, 76 and 100 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 103
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 171
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 169 | 174
percentage of participants
  Week 52: number analyzed (Participants) | 171 | 169 | 173
  Week 52 | 76.6 | 76.9 | 81.5
  Week 76: number analyzed (Participants) | 166 | 165 | 172
  Week 76 | 85.5 | 75.8 | 80.2
  Week 100: number analyzed (Participants) | 160 | 164 | 170
  Week 100 | 87.5 | 75.0 | 80.0

175. Secondary Outcome: Percentage of Participants Who Achieved PASI 100 Response at Weeks 52, 76 and 100 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 104
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 171
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 169 | 174
percentage of participants
  Week 52: number analyzed (Participants) | 171 | 169 | 173
  Week 52 | 55.0 | 54.4 | 60.7
  Week 76: number analyzed (Participants) | 166 | 165 | 172
  Week 76 | 65.1 | 59.4 | 68.0
  Week 100: number analyzed (Participants) | 160 | 164 | 170
  Week 100 | 69.4 | 57.3 | 64.1

176. Secondary Outcome: Percentage of Participants Who Achieved Both PASI 75 and ACR 20 Responses at Weeks 52, 76 and 100 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 48
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 171
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 169 | 174
percentage of participants
  Week 52: number analyzed (Participants) | 170 | 169 | 173
  Week 52 | 59.4 | 73.4 | 70.5
  Week 76: number analyzed (Participants) | 166 | 165 | 172
  Week 76 | 71.1 | 75.8 | 76.7
  Week 100: number analyzed (Participants) | 159 | 163 | 169
  Week 100 | 73.0 | 76.1 | 77.5

177. Secondary Outcome: Percentage of Participants Who Achieved Both PASI 75 and Modified PsARC Response at Weeks 52, 76, and 100 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 49
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 171
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 169 | 174
percentage of participants
  Week 52: number analyzed (Participants) | 171 | 169 | 173
  Week 52 | 70.8 | 79.3 | 76.9
  Week 76: number analyzed (Participants) | 166 | 165 | 172
  Week 76 | 78.3 | 79.4 | 82.6
  Week 100: number analyzed (Participants) | 160 | 164 | 170
  Week 100 | 78.8 | 81.1 | 78.8

178. Secondary Outcome: Percentage of Participants With an IGA Response at Weeks 52, 76 and 100 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: A psoriasis IGA response was defined as an IGA score of 0 (cleared) or 1 (minimal) and >= 2 grade reduction from baseline in the IGA psoriasis score. The IGA documents the investigator's assessment of the patient's psoriasis and lesions are graded for induration, erythema and scaling, each using a 5 point scale: 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe). The IGA score of psoriasis was based upon the average of induration, erythema and scaling scores. The participant's psoriasis was assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4). IGA Response is defined as achieving IGA score of 0 or 1, and >=2 grade reduction from baseline.
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 171
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 169 | 174
percentage of participants
  Week 52: number analyzed (Participants) | 171 | 169 | 173
  Week 52 | 84.2 | 76.9 | 84.4
  Week 76: number analyzed (Participants) | 166 | 165 | 172
  Week 76 | 85.5 | 77.6 | 86.0
  Week 100: number analyzed (Participants) | 160 | 165 | 170
  Week 100 | 88.1 | 76.4 | 82.4

179. Secondary Outcome: Percentage of Participants With an IGA Score of 0 (Cleared) at Weeks 52, 76 and 100 Among Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 107
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 171
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 169 | 174
percentage of participants
  Week 52: number analyzed (Participants) | 171 | 169 | 173
  Week 52 | 66.7 | 59.8 | 65.9
  Week 76: number analyzed (Participants) | 166 | 165 | 172
  Week 76 | 72.9 | 64.2 | 72.1
  Week 100: number analyzed (Participants) | 160 | 165 | 170
  Week 100 | 76.9 | 58.8 | 67.1

180. Secondary Outcome: Percentage of Participants Who Achieved a DLQI Score of 0 or 1 at Weeks 52, 76 and 100 Among the Participants With DLQI Score >1, With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 45
Time Frame: Weeks 52, 76 and 100
Population: Analysis population is FAS3 among the participants with DLQI Score >1, with >=3% BSA psoriatic involvement and an IGA score of >=2 (mild) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 161 | 152 | 163
percentage of participants
  Week 52: number analyzed (Participants) | 161 | 152 | 162
  Week 52 | 56.5 | 68.4 | 68.5
  Week 76: number analyzed (Participants) | 157 | 150 | 161
  Week 76 | 66.9 | 66.7 | 68.9
  Week 100: number analyzed (Participants) | 154 | 148 | 159
  Week 100 | 74.7 | 69.6 | 64.8

181. Secondary Outcome: Percentage of Participants Who Achieved >=5-point Improvement From Baseline in DLQI Score at Weeks 52, 76 and 100 Among the Participants With DLQI Score >=5, >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 46
Time Frame: Weeks 52, 76 and 100
Population: Analysis population is FAS3 among the participants with DLQI score >=5, >=3% BSA psoriatic involvement and an IGA score of >=2 (mild) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 138 | 129 | 143
percentage of participants
  Week 52: number analyzed (Participants) | 138 | 129 | 142
  Week 52 | 84.8 | 92.2 | 89.4
  Week 76: number analyzed (Participants) | 135 | 127 | 141
  Week 76 | 91.9 | 89.0 | 90.1
  Week 100: number analyzed (Participants) | 132 | 125 | 139
  Week 100 | 91.7 | 94.4 | 88.5

182. Secondary Outcome: Change From Baseline in DLQI Score at Weeks 52, 76 and 100 Among the Participants With >=3% BSA Psoriatic Involvement and an IGA Score of >=2 (Mild) at Baseline
Description: as for outcome 47
Time Frame: Baseline, Weeks 52, 76 and 100
Population: Analysis population is FAS3 among the participants with >=3% BSA psoriatic involvement and an IGA Score of >=2 (mild) at baseline. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 172 | 169 | 174
units on a scale
  Week 52: number analyzed (Participants) | 172 | 169 | 173
  Week 52 | -8.855 (7.2738) | -9.272 (7.3903) | -9.873 (6.8832)
  Week 76: number analyzed (Participants) | 167 | 167 | 172
  Week 76 | -10.090 (7.0888) | -9.180 (7.2977) | -9.610 (7.0383)
  Week 100: number analyzed (Participants) | 162 | 165 | 170
  Week 100 | -10.130 (7.2798) | -9.291 (7.2851) | -9.635 (7.0884)

183. Secondary Outcome: Change in Modified vdH-S Score From Baseline to Week 100
Description: as for outcome 6
Time Frame: Baseline to Week 100
Population: FAS3 for structural damage (FAS3-SD) included all randomized participants who were continuing study treatment at Week 52. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 204 | 216 | 211
units on a scale | 1.49 (6.859) | 1.50 (4.393) | 1.68 (7.018)

184. Secondary Outcome: Change in Total Modified vdH-S Score From Week 52 to Week 100
Description: as for outcome 113
Time Frame: From Week 52 to Week 100
Population: as for outcome 183
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 202 | 216 | 211
units on a scale | 0.13 (3.742) | 0.46 (2.419) | 0.75 (4.021)

185. Secondary Outcome: Change in Modified vdH-s Erosion Score From Baseline to Week 100
Description: as for outcome 6
Time Frame: Baseline to Week 100
Population: as for outcome 183
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 204 | 216 | 211
units on a scale | 1.01 (4.034) | 1.01 (3.355) | 1.02 (4.676)

186. Secondary Outcome: Change in Modified vdH-s Erosion Score From Week 52 to Week 100
Description: as for outcome 6
Time Frame: From Week 52 to Week 100
Population: as for outcome 183
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 202 | 216 | 211
units on a scale | 0.09 (1.978) | 0.26 (1.751) | 0.45 (2.900)

187. Secondary Outcome: Change in Modified vdH-s JSN Score From Baseline to Week 100
Description: as for outcome 6
Time Frame: Baseline to Week 100
Population: as for outcome 183
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 204 | 216 | 211
units on a scale | 0.49 (2.984) | 0.50 (1.387) | 0.66 (2.722)

188. Secondary Outcome: Change in Modified vdH-s JSN Score From Week 52 to Week 100
Description: as for outcome 6
Time Frame: From Week 52 to Week 100
Population: as for outcome 183
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 202 | 216 | 211
units on a scale | 0.04 (1.904) | 0.20 (0.917) | 0.30 (1.319)

189. Secondary Outcome: Change From Baseline to Week 100 in Modified vdH-S Score by Region and Type of Damage (ie, Hand Erosion, Hand JSN, Foot Erosion, Foot JSN Subscores)
Description: as for outcome 52
Time Frame: Baseline to Week 100
Population: FAS3 for structural damage (FAS3-SD) included all randomized participants who were continuing study treatment at Week 52. Here, n (number analyzed) signifies the number of participants analyzed at specified category.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Hand Erosion Score: number analyzed (Participants) | 204 | 216 | 211
  Hand Erosion Score | 0.67 (2.917) | 0.67 (2.807) | 0.49 (3.007)
  Hand JSN Score: number analyzed (Participants) | 204 | 216 | 211
  Hand JSN Score | 0.35 (2.443) | 0.34 (1.247) | 0.32 (1.845)
  Hand Score: number analyzed (Participants) | 204 | 216 | 211
  Hand Score | 1.02 (5.244) | 1.02 (3.815) | 0.81 (4.532)
  Foot Erosion Score: number analyzed (Participants) | 204 | 216 | 211
  Foot Erosion Score | 0.34 (1.596) | 0.33 (1.362) | 0.53 (2.436)
  Foot JSN Score: number analyzed (Participants) | 204 | 216 | 211
  Foot JSN Score | 0.13 (0.912) | 0.15 (0.652) | 0.34 (1.608)
  Foot Score: number analyzed (Participants) | 204 | 216 | 211
  Foot Score | 0.48 (2.373) | 0.48 (1.652) | 0.87 (3.761)

190. Secondary Outcome: Percentage of Participants With a Change of <=0 or <=0.5 From Baseline to Week 100 in Modified vdH-S Score
Description: as for outcome 6
Time Frame: Baseline to Week 100
Population: as for outcome 189
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Change of <=0 from Baseline: number analyzed (Participants) | 204 | 216 | 211
  Change of <=0 from Baseline | 60.8 | 55.6 | 62.6
  Change of <=0.5 from Baseline: number analyzed (Participants) | 204 | 216 | 211
  Change of <=0.5 from Baseline | 72.1 | 63.9 | 72.5

191. Secondary Outcome: Percentage of Participants With a Change of <=0 or <=0.5 From Baseline to Week 100 in Modified vdH-S Erosion Score
Description: as for outcome 6
Time Frame: Baseline to Week 100
Population: as for outcome 189
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Change of <=0 from Baseline: number analyzed (Participants) | 204 | 216 | 211
  Change of <=0 from Baseline | 64.2 | 61.1 | 65.4
  Change of <=0.5 from Baseline: number analyzed (Participants) | 204 | 216 | 211
  Change of <=0.5 from Baseline | 75.0 | 73.1 | 75.4

192. Secondary Outcome: Percentage of Participants With a Change of <=0 or <=0.5 From Baseline to Week 100 in Modified vdH-S JSN Score
Description: as for outcome 6
Time Frame: Baseline to Week 100
Population: as for outcome 189
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Change of <=0 from Baseline: number analyzed (Participants) | 204 | 216 | 211
  Change of <=0 from Baseline | 77.5 | 68.5 | 73.9
  Change of <=0.5 from Baseline: number analyzed (Participants) | 204 | 216 | 211
  Change of <=0.5 from Baseline | 84.3 | 79.6 | 81.0

193. Secondary Outcome: Percentage of Participants Without Radiographic Modified vdH-S Progression Based on (SDC) From Baseline to Week 100
Description: Modified vdH-S score is the sum of the erosion score (hand, feet) and JSN score (hand, feet). Joint erosion score is the summary of erosion severity in 40 joints of hand scored according to the surface area, from 0 (no erosion) to 5 (complete collapse of bone) and 12 joints of 2 feet (each side of foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum erosion score of 320. JSN score is the total JSN score in same 52 joints as above, each joint scored according to the subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum JSN score of 208. Total score ranges from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score indicates more joint damage. SDC was defined as the cut-off above which the changes can be detected beyond measurement error. Without radiographic progression was defined as change from baseline in the modified vdH-S score <=SDC of 3.46.
Time Frame: Baseline to Week 100
Population: as for outcome 183
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 204 | 216 | 211
percentage of participants | 86.8 | 84.7 | 87.2

194. Secondary Outcome: Percentage of Participants Without Radiographic Erosion Progression (Based on SDC) From Baseline to Week 100
Description: Modified vdH-S score is sum of the erosion score (hand, feet) and JSN score (hand, feet). Joint erosion score is summary of erosion severity in 40 joints of hand scored according to surface area, from 0 (no erosion) to 5 (complete collapse of bone) and 12 joints of 2 feet (each side of foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum erosion score of 320. JSN score is the total JSN score in same 52 joints as above, each joint scored according to subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum JSN score of 208. Total score ranges from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score indicates more joint damage. SDC was defined as the cut-off above which the changes can be detected beyond measurement error. Without radiographic erosion progression was defined as change from baseline in the modified vdH-S erosion score <=SDC of 2.66.
Time Frame: Baseline to Week 100
Population: as for outcome 183
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 204 | 216 | 211
percentage of participants | 86.8 | 87.0 | 88.6

195. Secondary Outcome: Percentage of Participants Without Radiographic JSN Progression (Based on SDC) From Baseline to Week 100
Description: Modified vdH-S score is sum of erosion score (hand, feet) and JSN score (hand, feet). Joint erosion score is summary of erosion severity in 40 joints of hand scored according to surface area, from 0 (no erosion) to 5 (complete collapse of bone) and 12 joints of 2 feet (each side of foot joint is graded on same 0-5 scale, thus maximum erosion score for a foot joint is 10), for a maximum erosion score of 320. JSN score is the total JSN score in same 52 joints as above, each joint scored according to the subluxation from 0 (normal) to 4 (bony ankylosis or complete luxation), for a maximum JSN score of 208. Total score ranges from 0 (best) to 528 (worst = worst possible erosion score of 320 + worst possible JSN score of 208). Higher score indicates more joint damage. SDC was defined as the cut-off above which the changes can be detected beyond measurement error. Without radiographic JSN progression was defined as change from baseline in the modified vdH-S JSN score <=SDC of 1.66.
Time Frame: Baseline to Week 100
Population: as for outcome 183
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 204 | 216 | 211
percentage of participants | 90.7 | 89.4 | 88.2

196. Secondary Outcome: Percentage of Participants With Pencil in Cup or Gross Osteolysis Deformities at Baseline, Weeks 24, 52, and 100
Description: Pencil in Cup or Gross Osteolytis Deformities are radiographic features specific for psoriatic arthritis.
Time Frame: Baseline, Weeks 24, 52, and 100
Population: FAS3 for structural damage (FAS3-SD) included all randomized participants who were continuing study treatment at Week 52. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Baseline: number analyzed (Participants) | 215 | 228 | 221
  Baseline | 3.7 | 3.9 | 3.6
  Week 24: number analyzed (Participants) | 215 | 228 | 221
  Week 24 | 3.7 | 3.9 | 4.1
  Week 52: number analyzed (Participants) | 213 | 228 | 221
  Week 52 | 4.2 | 4.4 | 3.6
  Week 100: number analyzed (Participants) | 204 | 216 | 211
  Week 100 | 4.9 | 4.6 | 3.8

197. Secondary Outcome: Change From Baseline in SF-36 PCS Score at Weeks 52, 76 and 100
Description: as for outcome 11
Time Frame: Baseline, Weeks 52, 76 and 100
Population: Analysis population is FAS3. Here, n (number analyzed) signifies the number of participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | 8.170 (8.2195) | 9.438 (8.2854) | 9.023 (8.6263)
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | 9.762 (8.5908) | 10.814 (9.0290) | 9.707 (8.5010)
  Week 100: number analyzed (Participants) | 214 | 224 | 220
  Week 100 | 10.508 (8.6819) | 11.282 (9.2753) | 10.559 (8.7449)

198. Secondary Outcome: Change From Baseline in SF-36 MCS Score at Weeks 52, 76 and 100
Description: as for outcome 13
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 197
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | 4.383 (10.9402) | 4.540 (9.7848) | 4.127 (9.1368)
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | 4.838 (11.0526) | 5.034 (10.0334) | 5.194 (9.4899)
  Week 100: number analyzed (Participants) | 214 | 224 | 220
  Week 100 | 4.610 (11.2527) | 4.718 (9.9014) | 4.936 (9.5935)

199. Secondary Outcome: Change From Baseline in Norm Based Scores of SF-36 Scales at Weeks 52, 76 and 100
Description: as for outcome 62
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 160
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: Physical Function Score: number analyzed (Participants) | 227 | 232 | 226
  Week 52: Physical Function Score | 7.757 (8.9727) | 8.406 (8.8407) | 8.493 (8.7691)
  Week 76: Physical Function Score: number analyzed (Participants) | 221 | 225 | 223
  Week 76: Physical Function Score | 8.824 (9.6648) | 9.807 (9.5044) | 9.294 (8.2020)
  Week 100: Physical Function Score: number analyzed (Participants) | 214 | 224 | 220
  Week 100: Physical Function Score | 9.738 (9.8405) | 10.953 (9.7761) | 10.126 (8.9271)
  Week 52: Role-physical Score: number analyzed (Participants) | 227 | 232 | 226
  Week 52: Role-physical Score | 6.538 (8.5151) | 7.665 (8.2925) | 7.372 (7.7581)
  Week 76: Role-physical Score: number analyzed (Participants) | 221 | 225 | 223
  Week 76: Role-physical Score | 8.372 (8.7202) | 9.171 (8.5844) | 8.579 (7.6709)
  Week 100: Role-physical Score: number analyzed (Participants) | 214 | 224 | 220
  Week 100: Role-physical Score | 9.181 (8.6596) | 9.342 (9.1746) | 8.921 (8.1775)
  Week 52: Bodily Pain Score: number analyzed (Participants) | 227 | 232 | 226
  Week 52: Bodily Pain Score | 8.536 (8.4602) | 10.201 (8.7312) | 9.525 (9.8357)
  Week 76: Bodily Pain Score: number analyzed (Participants) | 221 | 225 | 223
  Week 76: Bodily Pain Score | 10.368 (9.1058) | 11.552 (9.8591) | 10.300 (9.0504)
  Week 100: Bodily Pain Score: number analyzed (Participants) | 214 | 224 | 220
  Week 100: Bodily Pain Score | 10.696 (9.3854) | 11.585 (10.3527) | 10.998 (8.9230)
  Week 52: General Health Score: number analyzed (Participants) | 227 | 232 | 226
  Week 52: General Health Score | 6.533 (8.5245) | 7.097 (7.2500) | 6.450 (8.4316)
  Week 76: General Health Score: number analyzed (Participants) | 221 | 225 | 223
  Week 76: General Health Score | 7.203 (8.3372) | 7.470 (7.6119) | 6.761 (7.9631)
  Week 100: General Health Score: number analyzed (Participants) | 214 | 224 | 220
  Week 100: General Health Score | 6.710 (8.7265) | 7.066 (7.5829) | 7.132 (8.4887)
  Week 52: Vitality Score: number analyzed (Participants) | 227 | 232 | 226
  Week 52: Vitality Score | 7.997 (9.3878) | 8.695 (9.5033) | 7.637 (9.4393)
  Week 76: Vitality Score: number analyzed (Participants) | 221 | 225 | 223
  Week 76: Vitality Score | 8.859 (9.4372) | 9.388 (9.8618) | 8.659 (9.6026)
  Week 100: Vitality Score: number analyzed (Participants) | 214 | 224 | 220
  Week 100: Vitality Score | 9.648 (9.4778) | 9.827 (9.9348) | 9.155 (9.3569)
  Week 52: Social Function Score: number analyzed (Participants) | 227 | 232 | 226
  Week 52: Social Function Score | 6.361 (10.9927) | 7.304 (10.1003) | 6.810 (9.5118)
  Week 76: Social Function Score: number analyzed (Participants) | 221 | 225 | 223
  Week 76: Social Function Score | 7.509 (10.4249) | 8.623 (9.5176) | 7.914 (9.5191)
  Week 100: Social Function Score: number analyzed (Participants) | 214 | 224 | 220
  Week 100: Social Function Score | 7.825 (10.8558) | 8.080 (9.5383) | 8.113 (9.4847)
  Week 52: Role-emotional Score: number analyzed (Participants) | 227 | 232 | 226
  Week 52: Role-emotional Score | 4.111 (10.9413) | 4.998 (10.1964) | 4.699 (8.7759)
  Week 76: Role-emotional Score: number analyzed (Participants) | 221 | 225 | 223
  Week 76: Role-emotional Score | 5.199 (11.1875) | 5.757 (10.0737) | 5.433 (9.2389)
  Week 100: Role-emotional Score: number analyzed (Participants) | 214 | 224 | 220
  Week 100: Role-emotional Score | 4.784 (11.9482) | 5.720 (10.1991) | 5.128 (9.7998)
  Week 52: Mental Health Score: number analyzed (Participants) | 227 | 232 | 226
  Week 52: Mental Health Score | 5.209 (10.0958) | 4.826 (9.4038) | 4.839 (9.4029)
  Week 76: Mental Health Score: number analyzed (Participants) | 221 | 225 | 223
  Week 76: Mental Health Score | 5.481 (10.5927) | 5.430 (10.0802) | 6.124 (8.7930)
  Week 100: Mental Health Score: number analyzed (Participants) | 214 | 224 | 220
  Week 100: Mental Health Score | 5.514 (10.6204) | 5.477 (10.1202) | 6.148 (8.8743)

200. Secondary Outcome: Percentage of Participants Who Achieved >=5-point Improvement From Baseline in SF-36 PCS Score at Weeks 52, 76 and 100
Description: as for outcome 64
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 197
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | 63.4 | 66.8 | 65.9
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | 70.6 | 73.8 | 65.5
  Week 100: number analyzed (Participants) | 214 | 224 | 220
  Week 100 | 72.4 | 70.1 | 68.6

201. Secondary Outcome: Percentage of Participants Who Achieved >=5-point Improvement From Baseline in SF-36 MCS Score at Weeks 52, 76 and 100
Description: as for outcome 63
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 197
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | 42.3 | 45.3 | 38.9
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | 43.9 | 44.4 | 43.5
  Week 100: number analyzed (Participants) | 214 | 224 | 220
  Week 100 | 42.1 | 46.4 | 43.6

202. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Weeks 52, 76 and 100
Description: as for outcome 65
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 197
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | 7.692 (9.3071) | 8.935 (9.5033) | 7.699 (9.1417)
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | 9.167 (9.0455) | 9.596 (10.4788) | 8.632 (8.8429)
  Week 100: number analyzed (Participants) | 214 | 224 | 220
  Week 100 | 9.435 (9.4513) | 10.107 (10.2076) | 9.127 (8.9948)

203. Secondary Outcome: Percentage of Participants Who Achieved >=4-point Improvement From Baseline in FACIT-Fatigue Score at Weeks 52, 76 and 100
Description: as for outcome 66
Time Frame: Weeks 52, 76 and 100
Population: as for outcome 197
Measure: Number; unit: percentage of participants
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
percentage of participants
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | 68.7 | 69.4 | 68.1
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | 70.6 | 69.3 | 74.4
  Week 100: number analyzed (Participants) | 214 | 224 | 220
  Week 100 | 72.0 | 72.8 | 74.1

204. Secondary Outcome: Change From Baseline in EQ-5D-5L at Weeks 52, 76 and 100: EQ-VAS
Description: as for outcome 67
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 197
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | 21.608 (25.5992) | 23.392 (23.6990) | 20.190 (24.8348)
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | 24.176 (27.7205) | 25.053 (26.0372) | 22.251 (24.6934)
  Week 100: number analyzed (Participants) | 213 | 224 | 219
  Week 100 | 25.901 (28.4028) | 27.152 (26.5221) | 25.909 (26.0995)

205. Secondary Outcome: Change From Baseline in EQ-5D-5L at Weeks 52, 76 and 100: EQ-5D Index
Description: as for outcome 68
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 197
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | 0.138 (0.1608) | 0.150 (0.1445) | 0.138 (0.1458)
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | 0.154 (0.1744) | 0.169 (0.1564) | 0.147 (0.1471)
  Week 100: number analyzed (Participants) | 213 | 224 | 219
  Week 100 | 0.164 (0.1605) | 0.164 (0.1596) | 0.156 (0.1543)

206. Secondary Outcome: Change From Baseline in WPAI Scores (Percent Work Time Missed) at Weeks 52, 76 and 100
Description: as for outcome 32
Time Frame: Baseline, Weeks 52, 76 and 100
Population: Analysis population is FAS3. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, n (number analyzed) signifies the number of participants analyzed for specified categories at specified timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 136 | 130 | 130
units on a scale
  Week 52 | -5.45 (25.544) | -4.50 (20.530) | -1.83 (17.191)
  Week 76: number analyzed (Participants) | 134 | 126 | 125
  Week 76 | -5.92 (26.032) | -6.22 (23.133) | -2.39 (19.277)
  Week 100: number analyzed (Participants) | 125 | 120 | 115
  Week 100 | -8.81 (24.313) | -5.81 (21.606) | -1.56 (16.956)

207. Secondary Outcome: Change From Baseline in WPAI Scores (Percent Impairment While Working) at Weeks 52, 76 and 100
Description: as for outcome 32
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 206
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 116 | 121 | 122
units on a scale
  Week 52 | -21.81 (31.391) | -27.93 (25.263) | -22.62 (26.058)
  Week 76: number analyzed (Participants) | 116 | 113 | 111
  Week 76 | -26.90 (28.965) | -29.91 (24.549) | -26.13 (25.412)
  Week 100: number analyzed (Participants) | 109 | 108 | 103
  Week 100 | -30.73 (30.933) | -30.65 (24.771) | -27.77 (26.119)

208. Secondary Outcome: Change From Baseline in WPAI Scores (Percent Overall Work Impairment) at Weeks 52, 76 and 100
Description: as for outcome 32
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 206
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 116 | 121 | 122
units on a scale
  Week 52 | -22.61 (31.979) | -28.19 (25.536) | -22.79 (26.793)
  Week 76: number analyzed (Participants) | 116 | 113 | 111
  Week 76 | -27.98 (29.709) | -30.27 (26.058) | -26.21 (28.115)
  Week 100: number analyzed (Participants) | 109 | 108 | 103
  Week 100 | -31.87 (31.013) | -31.75 (25.615) | -25.21 (26.317)

209. Secondary Outcome: Change From Baseline in WPAI Scores (Percent Activity Impairment Outside of Work) Weeks 52, 76 and 100
Description: as for outcome 32
Time Frame: Baseline, Weeks 52, 76 and 100
Population: as for outcome 197
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo to Guselkumab 100 mg q4w | Guselkumab 100 mg q8w | Guselkumab 100 mg q4w
Number analyzed (Participants) | 228 | 232 | 227
units on a scale
  Week 52: number analyzed (Participants) | 227 | 232 | 226
  Week 52 | -24.67 (27.106) | -27.16 (25.662) | -26.24 (25.113)
  Week 76: number analyzed (Participants) | 221 | 225 | 223
  Week 76 | -28.05 (26.411) | -31.38 (25.449) | -28.70 (24.635)
  Week 100: number analyzed (Participants) | 213 | 224 | 219
  Week 100 | -30.70 (28.632) | -30.98 (26.650) | -30.68 (25.305)

ADVERSE EVENTS:
Time Frame: From baseline after the first administration of study drug through End of Study (up to Week 112)
Description: Safety population included participants randomized at Week 0 who received at least 1 (partial or complete) dose of study agent and were analyzed according to the actual treatment received after randomization. Data for Guselkumab 100 mg q8w and q4w arms was planned to be reported separately for Week 0 to 24 and Week 0 to 52.
Groups:
- Placebo (CP): Participants received placebo matched to guselkumab subcutaneous injections every 4 weeks through Week 20 in the placebo controlled period (CP). Data prior to the first administration of guselkumab, or through the last follow-up visit if the participant did not receive any guselkumab, were included.
- Guselkumab 100 mg q8w (CP): Participants received guselkumab 100 milligram (mg) subcutaneous injections at Weeks 0 and 4 then every 8 weeks and placebo matched to guselkumab injections at other visits through Week 20 in the placebo controlled period (CP). Data through Week 24, or through the last follow-up visit if the participant did not receive any study drug at or after Week 24, were included.
- Guselkumab 100 mg q4w (CP): Participants received guselkumab 100 milligram (mg) subcutaneous injections every 4 weeks from Week 0 through Week 20 in the placebo controlled period (CP). Data through Week 24, or through the last follow-up visit if the participant did not receive any study drug at or after Week 24, were included.
- Placebo to Guselkumab 100 mg q4w (After CP Through Week 112): Participants who received placebo matched to guselkumab subcutaneous injections every 4 weeks through Week 20 in the placebo controlled period (CP) received guselkumab 100 milligram (mg) subcutaneous injections every 4 weeks from Week 24 through Week 100. Data from the first administration of guselkumab through Week 112 (End of Study) were included.
- Guselkumab 100 mg q8w (Through Week 112): Participants received guselkumab 100 milligram (mg) subcutaneous injections at Weeks 0 and 4 then every 8 weeks and placebo matched to guselkumab injections at other visits through Week 100. Data from Week 0 through Week 112 (End of Study) were included.
- Guselkumab 100 mg q4w (Through Week 112): Participants received guselkumab 100 milligram (mg) subcutaneous injections every 4 weeks from Week 0 through Week 100. Data from Week 0 through Week 112 (End of Study) were included.
Arm/Group | Placebo (CP) | Guselkumab 100 mg q8w (CP) | Guselkumab 100 mg q4w (CP) | Placebo to Guselkumab 100 mg q4w (After CP Through Week 112) | Guselkumab 100 mg q8w (Through Week 112) | Guselkumab 100 mg q4w (Through Week 112)
All-Cause Mortality (participants affected / at risk) | 0/246 | 0/248 | 0/245 | 1/238 | 0/248 | 0/245
Serious Adverse Events (participants affected / at risk) | 7/246 | 3/248 | 8/245 | 16/238 | 22/248 | 22/245
Other Adverse Events (participants affected / at risk) | 30/246 | 42/248 | 52/245 | 48/238 | 88/248 | 79/245
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=246) | Guselkumab 100 mg q8w (CP) (N=248) | Guselkumab 100 mg q4w (CP) (N=245) | Placebo to Guselkumab 100 mg q4w (After CP Through Week 112) (N=238) | Guselkumab 100 mg q8w (Through Week 112) (N=248) | Guselkumab 100 mg q4w (Through Week 112) (N=245)
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Angina Unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 2 | 0 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diverticular Perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Inflammatory Bowel Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pancreatitis Chronic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Umbilical Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Post Cholecystectomy Syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute Hepatitis B (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Acute Hepatitis C (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Complicated Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Dacryocystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Dengue Fever (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Herpes Zoster Disseminated (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Infective Periostitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Medical Device Site Joint Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Meningitis Listeria (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Oophoritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 2 | 1
Pneumonia Influenzal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia Necrotising (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Vaginitis Gardnerella (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Vulvovaginitis Trichomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 3 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Metal Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Muscle Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Post Procedural Fistula (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 2
Psoriatic Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Clear Cell Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Extrapyramidal Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tubulointerstitial Nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cervical Polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Sinus Perforation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blue Toe Syndrome (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic Venous Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (CP) (N=246) | Guselkumab 100 mg q8w (CP) (N=248) | Guselkumab 100 mg q4w (CP) (N=245) | Placebo to Guselkumab 100 mg q4w (After CP Through Week 112) (N=238) | Guselkumab 100 mg q8w (Through Week 112) (N=248) | Guselkumab 100 mg q4w (Through Week 112) (N=245)
Bronchitis (Infections and infestations) | 3 | 1 | 10 | 7 | 10 | 15
Nasopharyngitis (Infections and infestations) | 9 | 10 | 12 | 9 | 25 | 21
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 7 | 13 | 18 | 24 | 20
Alanine Aminotransferase Increased (Investigations) | 11 | 15 | 22 | 11 | 29 | 31
Aspartate Aminotransferase Increased (Investigations) | 6 | 14 | 11 | 10 | 23 | 23
Headache (Nervous system disorders) | 2 | 6 | 3 | 7 | 16 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT03158285/Prot_002.pdf
  • Statistical Analysis Plan (2019-03-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03158285/SAP_001.pdf